Bempedoic Acid (ETC-1002) Clinical Study Report: 1002-050

### 16.1.9 **Documentation of Statistical Methods**

| Original Statistical Analysis Plan (SAP) Version 1.0 | 14 February 2017 |
|---------------------------------------------------------|------------------|
| SAP Version 1.1 | 19 October 2018 |
| SAP Version 1.2 | 05 December 2018 |
| SAP Addendum for Day 120 Safety Update Interim Analysis | 23 May 2019 |
| SAP Version 1.3 | 04 December 2019 |

#### Statistical Analysis Plan

Title: A MULTICENTER OPEN-LABEL EXTENSION (OLE) STUDY

TO ASSESS THE LONG-TERM SAFETY AND EFFICACY OF

BEMPEDOIC ACID (ETC-1002) 180 MG

**Protocol:** ETC-1002-050

**Clinical Phase:** 3

ETC-1002 **Product:** 

Statistical Analysis Plan – Version 1.0 Version (Date):

**Status:** 

Final This document was signed in February 2020 because a signed version from 2017 could not be located.

# Prepared by: 05 Feb 2020 13:50:010+0000 REASON: I approve this document as author. a05dfa7f-b536-4636-ad10-1bb0fd2ce580 Date 04 Feb 2020 20:56:021+0000 REASON: I approve this document 17064876-dedd-4660-9752-8d3bc4287a9e Date signed on behalf of 04 Feb 2020 21:02:016+0000 REASON: I approve this document 71728b78-53ad-43bd-94f5-4416d0d23979 Date **Esperion Therapeutics** signed on behalf of 12 Feb 2020 13:22:010+0000 REASON: I approve this document 4901ad6b-ef32-4d59-80a4-a17c1403b3b6 Date

**Esperion Therapeutics** 


### **Table of Contents**

| 1 | List | of Abbreviations | 4 |
|---|---------|-------------------------------------------------|------|
| 2 | Intr | oduction | 7 |
| 3 | Stu | dy Objectives and Endpoints | 7 |
| | 3.1 | Objectives | 7 |
| | 3.2 | Primary Endpoint | |
| | 3.3 | Secondary Endpoints | |
| | 3.3. | • 1 | |
| | | 2 Clinical Safety Laboratories | |
| | 3.3. | · | |
| | 3.4 | Lipids | |
| | 3.5 | Pharmacokinetic (PK) and Other Biomarkers | |
| 4 | | | |
| 4 | 4.1 | dy Design | |
| | | Study Design | |
| | 4.2 | Study Treatments and Assessments | |
| | 4.3 | Randomization and Blinding | |
| | 4.4 | Sample Size Justification | |
| | 4.5 | Interim Analyses, Final Analyses and Unblinding | |
| | 4.6 | Change from Planned Analyses | |
| 5 | | tistical and Analytical Plans | |
| | 5.1 | General Statistical Considerations | |
| | 5.2 | Statistical Analysis Plans | 2 |
| | 5.2. | 1 Analysis Sets | 2 |
| | 5 | .2.1.1 Safety Population (SP) | 2 |
| | 5 | .2.1.2 Full Analysis Set (FAS) | 2 |
| | 5.2. | 2 Protocol Violations and Deviations | 2 |
| | 5.2. | 3 Subject Disposition | 3 |
| | 5.2. | 4 Demographic and Baseline Characteristics | 3 |
| | 5.2. | | |
| | 5.2. | · | |
| | 5.2. | | |
| | 5.3 | Efficacy Endpoints and Analyses | |
| | 5.4 | Safety Data Endpoints and Analyses | |
| | | 1 Adverse Events (AEs) | |
| | 5.4. | | |
| | 5.4. | | |
| | 5.4. | • | |
| | 5.4. | | |
| | | .4.5.1 Hepatic Safety | |
| | | 1 | |
| | | <b>→</b> | |
| | | .4.5.3 Diabetes and Glycemia | |
| | | .4.5.4 Renal Safety 2 | |
| | 5.4. | • | |
| | 5.4. | $oldsymbol{o}$ | |
| | 5.4. | | 1 |
| C | onfider | ntial Page 2 of | f 24 |

| Esperion | Therapeutics, Inc. |
|-----------|--------------------|
| Protocol: | ETC-1002-050 |

## Version 1.0, Feb 14, 2017 Statistical Analysis Plan

| 6 | DMC Analyses | . 21 |
|---|--------------|------|
| 7 | Reference | . 21 |
| | Appendices | |

## 1 List of Abbreviations

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|-----------------------------------------|
| ACL | Adenosine triphosphate-citrate lyase |
| ACS | Acyl-CoA synthetase |
| ADR | Adverse drug reaction |
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ALB | Albumin |
| ALK-P | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| ApoB | Apolipoprotein B |
| ASCVD | Atherosclerotic cardiovascular diseases |
| AST | Aspartate aminotransferase |
| ATP | Adenosine triphosphate |
| AUC | Area under the concentration-time curve |
| AUC <sub>0-24</sub> | Area under the curve during 24 hours |
| BMI | Body mass index |
| BP | Blood pressure |
| BUN | Blood urea nitrogen |
| Ca | Calcium |
| CEC | Clinical Event Committee |
| CFR | Code of Federal Regulations |
| CHD | Coronary heart disease |
| CI | Confidence interval |
| CK | Creatine kinase |
| Cl | Chloride |
| CNS | Central nervous system |
| CoA | Acetyl-coenzyme A |
| $CO_2$ | Carbon dioxide |
| CV | Cardiovascular |
| CYP | Cytochrome P450 |
| DBP | Diastolic blood pressure |
| DMC | Data Monitoring Committee |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| eGFR | Estimated glomerular filtration rate |
| EMA | European Medicines Agency |


| Abbreviation or Specialist Term | Explanation |
|---|---|
| EOS | End of Study |
| ETC-1002 | Bempedoic acid |
| EU | European Union |
| FAS | Full analysis set |
| FDA | Food and Drug Administration |
| FPFV | First patient first visit |
| FSH | Follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GI | Gastrointestinal |
| HbA <sub>1C</sub> | Glycosylated hemoglobin, Type A <sub>1C</sub> |
| HBsAg | Hepatitis B surface antigen |
| Het | Hematocrit |
| HCV | Hepatitis C virus |
| HDL-C | High-density lipoprotein cholesterol |
| HeFH | Heterozygous familial hypercholesterolemia |
| Hgb | Hemoglobin |
| HMG-CoA | 3-hydroxy-3-methylglutaryl-coenzyme A |
| hs-CRP | High-sensitivity C-reactive protein |
| IB | Investigator's Brochure |
| ICD | Informed Consent Document |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IMP | Investigational medicinal product |
| IND | Investigational New Drug Application |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| ITT | Intention-to-treat |
| IUD | Intrauterine device |
| IWRS | Interactive web response system |
| K | Potassium |
| LDH | Lactate dehydrogenase |
| LDL-C | Low-density lipoprotein cholesterol |
| LDLR | LDL receptor |
| LFT | Liver function test |
| LPLV | Last patient last visit |
| LS | Least square |
| MACE | Major adverse cardiac event |
| МСН | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean corpuscular volume |


| Abbreviation or Specialist Term | Explanation |
|---|---|
| MDRD | Modification of diet in renal disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Myocardial infarction |
| MRI | Magnetic resonance imaging |
| Na | Sodium |
| NA | Not applicable |
| NLA | National Lipid Association |
| NOAEL | No-observed-adverse-effect level |
| non-HDL-C | Non-high-density lipoprotein cholesterol |
| OLE | Open-label extension (study) |
| Parent study | Study 1002-040 |
| PCSK9 | Proprotein convertase subtilisin/kexin type 9 |
| PE | Physical exam |
| PK | Pharmacokinetic(s) |
| PT | Prothrombin time |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SOC | System organ class |
| SP | Safety population |
| SUSARS | Suspected and unexpected serious adverse reactions |
| T2DM | Type 2 diabetes mellitus |
| TB | Total bilirubin |
| TC | Total cholesterol |
| TEAE | Treatment-emergent adverse event |
| TG | Triglycerides |
| TQT | Thorough QT/QTc |
| ULN | Upper limit of normal |
| US | United States |
| WBC | White blood cell |
| WHO | World Health Organization |


DocUUID: 48cc0ac5-92b1-46d4-8169-561a83ab7e61

### 2 Introduction

The purpose of this document is to describe the statistical methods, data derivations and data summaries to be employed in ETC-1002-050. The preparation of this statistical analysis plan (SAP) has been based on International Conference on Harmonisation (ICH) E3 and E9 Guidelines and in reference to Protocol ETC-1002-050 (Protocol V1.0, November 01, 2016).

The SAP will supersede the protocol in the event of any differences between the two documents in the plans for data analysis, and the protocol will be amended if appropriate. The SAP will be included as an appendix in the clinical study report for this protocol.

## 3 Study Objectives and Endpoints

## 3.1 Objectives

- The primary objective for this study is to characterize the safety and tolerability of long-term administration of bempedoic acid (ETC-1002) 180 mg
- The secondary objective is to characterize the efficacy of long-term administration of bempedoic acid 180 mg/day as assessed by changes in low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-high-density lipoprotein cholesterol (non-HDL-C), apolipoprotein B (ApoB), total cholesterol (TC), triglycerides TG and high-sensitivity C-reactive protein (hs-CRP) in patients with hyperlipidemia

## 3.2 Primary Endpoint

• The primary endpoint for this study is patient incidence of AEs

## 3.3 Secondary Endpoints

- Percent change from baseline in LDL-C at Weeks 52 and 78
- Change from baseline in LDL-C at Weeks 52 and 78
- Percent change from baseline in non-HDL-C at Weeks 52 and 78
- Percent change from baseline in TC at Weeks 52 and 78
- Percent change from baseline in ApoB at Weeks 52 and 78
- Percent change from baseline in hs-CRP at Weeks 52 and 78
- Percent change from baseline in TG at Weeks 52 and 78


• Percent change from baseline in HDL-C at Weeks 52 and 78

#### 3.3.1 Adverse Events

The evaluation of AEs will include only incidence of treatment-emergent AEs (TEAEs), defined as AEs that begin or worsen after the first dose of study drug administration in OLE period and until 30 days after last dose of study drug. Clinical endpoints (details see section 4.2) will be collected and adjudicated by an independent Clinical Events Committee (CEC). Clinical endpoints will also be reported as SAEs. Adverse events of special interest (AESI) will further be examined (See Section 5.4.2 for more information).

#### 3.3.2 Clinical Safety Laboratories

The evaluation of clinical safety laboratories, including blood hematology, chemistry, coagulation, and urinalysis, will be based on the observed values. Observed values and changes from baseline will be summarized for all post-baseline study visits.

#### 3.3.3 ECG, Vital Signs and PE

The evaluation of ECG and vital signs (including heart rate, systolic blood pressure, diastolic blood pressure, height, and weight will be based on the observed values. For ECGs, shifts from baseline to end-of-study will be summarized. For vital signs, observed values and changes from baseline will be summarized for all post-baseline study visits. Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant.'

## 3.4 Lipids

After enrollment, patients will return to clinic at Months 12, 52, and 78. Clinical laboratory samples will be collected and analyzed for calculated LDL-C and lipid and cardiometabolic biomarkers including non-HDL-C, HDL-C, TC, ApoB, and TG at baseline and all clinic visits for evaluation of bempedoic acid effects on lipids and cardiometabolic parameters.

## 3.5 Pharmacokinetic (PK) and Other Biomarkers

NA.

## 4 Study Design

### 4.1 Study Design

This is a multicenter OLE study designed to assess the long-term safety and efficacy of bempedoic acid (ETC-1002) 180 mg. All patients will receive open-label bempedoic acid 180 mg for up to 1.5 years after rolling over from the parent study (Study 1002-040), where they receive either bempedoic acid or placebo treatment. Investigators, site staff, patients,


and the study team will be masked to study lipid levels until the Week 12 study visit, after which time lipid values will be made available.

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other ongoing studies of bempedoic acid. A blinded independent expert Clinical Events Committee (CEC) will adjudicate designated clinical endpoints across the program, including all major adverse cardiac events (MACE) and non-MACE endpoints defined as: cardiovascular (CV) death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction [MI] (MACE), nonfatal stroke (MACE), hospitalization for unstable angina (MACE), coronary revascularization (MACE), noncoronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE) using standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs as well as a clinical endpoint.

The study will be conducted at approximately 125 clinical sites in the United States, Canada, Germany, Netherlands, Poland, and United Kingdom. The study will end when the last randomized patient completes their last study visit (last patient last visit [LPLV] for last randomized patient). The estimated overall duration of the study (first patient first visit [FPFV] to LPLV) is approximately 2.5 years.

1.5 Years

ETC-1002
Protocol 1002-040

ETC-1002 + Standard of Care

Figure 1. Study 1002-040 Study Design

### 4.2 Study Treatments and Assessments

Day 1 for this study should occur on the same day as the end of study visit for the parent study (1002-040). Patients who provide informed consent and sign the ICD will be eligible to enroll in the study.

The schedule of study events is provided in Appendix 1. However, a patient can be seen at any time for reasons of safety.

The investigational products were listed in Table 1 below:


**Table 1: Investigational Medicinal Products** 

| | Investigational Medicinal Product |
|---|---|
| Product Name: | Bempedoic acid |
| Dosage Form: | Film-coated tablets |
| Unit Dose: | 180 mg |
| Container/Closure <sup>a</sup> | 100-count bottle with screw on, child proof cap |
| Route of Administration: | Oral, daily with or without food |
| Physical Description: | |
| Manufacturer<br>(Fill/Finish): | |

Study drug should be taken once a day (once every 24 hours) at approximately the same time every day and may be taken with or without food. Patients will fast (no food or drink, other than water) for a minimum of 10 hours prior to collection of all laboratory samples.

Please see Pharmacy Manual for detailed storage requirements and instructions.

Patients who withdraw from investigational medicinal product (IMP) treatment will be asked to continue to be followed for safety using the protocol-specified visit schedule and procedures. For details of study assessments, see Appendix 1: Schedule of Events (Subject Visit Schedule).

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other any ongoing studies of ETC-1002. All clinical endpoints, including all major cardiac events (MACE) and non-MACE endpoints defined as: CV death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction (MI) (MACE), nonfatal stroke (MACE), hospitalization for unstable (MACE), coronary revascularization (MACE), angina non-coronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE), will be adjudicated by an independent blinded expert Clinical Events Committee (CEC), using standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs.


DocUUID: 48cc0ac5-92b1-46d4-8169-561a83ab7e61

### 4.3 Randomization and Blinding

- Randomization is not applicable for this OLE study.
- Laboratory results for lipid panel and hs-CRP will be masked to investigators, patients, and the study team until the Week 12 visit is completed. All site staff involved with this trial should refrain from obtaining lipid panels between date of last study medication (bempedoic acid or placebo) dose at end of parent study Week 52 (Visit T7) and Week 12 in this OLE trial.

### **4.4** Sample Size Justification

The number of patients entering this study will depend on the number of patients completing Study 1002-040 and their willingness to enroll.

### 4.5 Interim Analyses, Final Analyses and Unblinding

No formal interim analysis is planned for this study.

An interim data cut-off may occur in order to provide safety assessment to support NDA submission; the actual date will be determined by Esperion team.

The final analysis will be performed after the database is locked, and the database released.

## 4.6 Change from Planned Analyses

There is no change from planned analyses for this study.

## 5 Statistical and Analytical Plans

#### 5.1 General Statistical Considerations

The ETC-1002 treatment group will be displayed in the tables, listings and figures (TLFs) as "bempedoic acid 180 mg."

In general, all safety and efficacy data will be reported as observed. No imputation will be performed for missing data. Descriptive statistics (n, mean, standard deviation [SD] or Standard Error [SE], median, minimum, and maximum) will be calculated for continuous data. Minimum and maximum will be presented same number of decimal places as reported/collected, one additional decimal place for mean and median, and two additional decimal places for SD.

Categorical data will be summarized using n and percentage based on number of nonmissing values. Percentage will be presented with one decimal place. The number of missing values will be presented as a separate category with no percentage, but only if 1 or more patients are missing data for the summary. Otherwise, all categories will be


presented (even if no patients are counted in the category). Counts of zero in any category will be presented without percentage. Ninety-five percent (95%) confidence intervals (CIs) will be calculated for select continuous and categorical endpoint estimates. All patients will be summarized together as well as by their prior treatment group in the parent study.

Data will be presented on listings in order of patient/subject, assessment date and assessment (in order collected on CRF, unless specified otherwise). Dates will be presented in format DDMMMYYYY.

Relative day calculations will be [date of interest – relative date + 1? (date of interest >= relative date)]. This calculation will result in dates prior to the relative date being presented as negative days, and those occurring on or after the relative date as Day 1 or later, i.e., there will be no Day 0.

For efficacy endpoint analysis, baseline is defined as the same baseline as parent study. For safety analysis, baseline is defined as the last value/result where assessment date is less than or equal to the date of first study treatment, unless otherwise specified. If last dose of study treatment is missing, then the date of last visit at which study assessments were obtained on CRF will be used in its place.

The visit schedules and window are shown below.

| Visit | Day 1/Week 0 | Week<br>12 | Week 24 | Week 36 | Week 52 | Week 64 | Week<br>78/EOS |
|---|---|---|---|---|---|---|---|
| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOS |
| Slotted Study Week | EOS Parent | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 |
| Target Study Day | 1 | 84 | 168 | 252 | 364 | 448 | 546 |
| Analysis Window | 1 | [2,126] | [127,210] | [211,308] | [309,406] | [407,497] | [498,∞] |
| Protocol defined visit<br>Windows | [30 Days, Pre<br>M0] | 84±7 | 168±7 | 252±7 | 364±7 | 448±7 | 546±7 |

### 5.2 Statistical Analysis Plans

#### 5.2.1 Analysis Sets

#### **5.2.1.1 Safety Population (SP)**

The Safety Population (SP) is defined as all enrolled patients who received at least 1 dose of study medication and will be used for demographics and baseline characteristics, treatment exposure, concomitant medications, and all safety summaries.

#### 5.2.1.2 Full Analysis Set (FAS)

The Full Analysis Set (FAS) is defined as all enrolled patients and is also known as the intention-to-treat (ITT) set of patients. FAS will be used for all of the efficacy summaries and analyses.

#### 5.2.2 Protocol Violations and Deviations

A full list of protocol violations and deviations will be compiled and reviewed by the clinical team to identify major versus minor violations/deviations before final database Confidential


lock. For violations at study entry, patients will be assessed against the inclusion and exclusion criteria of the protocol. For on-study deviations, compliance with the protocol will be examined with regard to prohibited therapies, and timing and availability of planned assessments.

#### 5.2.3 Subject Disposition

The number of patients enrolled, and included in each analysis population, along with study completion status, will be summarized by the treatment group in parent ETC-1002-040 study and overall. In addition, the number of patients who withdraw from the study and withdraw from study drug will be summarized by discontinuation reason.

#### **5.2.4** Demographic and Baseline Characteristics

Demographic and baseline characteristics collected from the parent study will be used for this study. The following demographic and baseline characteristics will be summarized by previous treatment group in parent study, as well as overall, for safety population and for FAS population: age (years), gender, race, ethnicity, region, height (cm), weight (kg), body mass index (kg/m²), waist circumference (cm), systolic and diastolic blood pressure (mmHg), fasting lipid parameters (TC [mg/dL], calculated LDL-C [mg/dL], HDL-C [mg/dL], non-HDL-C [mg/dL] and TG [mg/dL]), apoB (mg/dL), hs-CRP (mg/dL), ASCVD only/HeFH, baseline statin intensity (low, moderate, high), eGFR category, tobacco history, alcohol history, and weekly average number of alcoholic drinks, history of diabetics, history of hypertension. Data will be summarized using descriptive statistics for continuous variables and using counts and percentages for categorical variables by treatment group and overall. Age will be summarized as a continuous variable and by age group (18-40, 41-64, 65-74, and >=75).

The baseline estimated glomerular filtration rate (eGFR) categories are: normal: ≥90 mL/min/1.73m<sup>2</sup>; mild Renal Impairment: 60-89 mL/min/1.73m<sup>2</sup>; moderate Renal Impairment: 30-59 mL/min/1.73m<sup>2</sup>, and severe Renal Impairment (15-29 mL/min/1.73m<sup>2</sup>).

The reasons for patients who are not on a highest dose of a high intensity statin will be summarized and presented in a by-patient listing.

#### 5.2.5 Medical History

General medical history, cardiovascular history/risk factors, previous statin use and statin tolerance history will be summarized by previous treatment group in parent study, as well as overall in OLE study, for safety population and FAS population and presented in a bypatient listing. Where appropriate, terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 18.1 or later.

If a patient is entering the study beyond the 30 day rollover window, changes to medical history that occur during that period will be collected. The changes will be summarized for safety population and presented in a by-patient listing.


#### 5.2.6 Prior and Concomitant Medications

Prior medications are defined as medications that ended prior to the initiation of study drug in this OLE study. Concomitant medications are defined as medications that were ongoing at the time of study drug initiation in this OLE study or new medications that started post study drug initiation and within 30 days following the date of the last dose of study drug.

Medications, including prior statin medications, will be coded using WHO Drug (March, 2015, or later if appropriate). The frequency of use of prior medications and use of concomitant medications will be summarized by previous treatment group in parent study, as well as overall in OLE study, for the safety population according to Anatomical Therapeutic Chemical (ATC) class and preferred term. If there is no enough prior medication data, prior medications will be presented in a by-patient listing only. Prior and concomitant medications will be listed for each patient. Prior and concomitant statin medications will be summarized and listed similarly.

#### 5.2.7 Study Drug Exposure and Compliance

The length of exposure to study drug will be calculated as the number of days from the first dose of study drug to the last dose of study drug, regardless if the patient missed one or more doses of study drug. Length of exposure will be summarized by previous treatment group in parent study and overall in OLE study using descriptive statistics for the safety population.

The number and percentage of patients who were compliant with taking study drug will be summarized by previous treatment group in parent study and overall in OLE study and post-baseline time point for the safety population for the following categories 0 - <50%; >= 50 - <80%; >= 80%. Compliance at each Visit (x)will be assessed by site staff by counting the number of tablets that are returned as unused study drug and querying the patient regarding daily intake and calculated using the formula: 100\* (Number Dispensed at Visit x-1 – Number Returned at Visit x) / (Duration in days between Visit x and Visit x-1). Overall compliance during the study will be similarly calculated.

The study drug administration and compliance data, including reasons for poor compliance, will be listed for each patient.

### 5.3 Efficacy Endpoints and Analyses

For all efficacy endpoints and analyses, the FAS will be used. For summary by previous treatment group in parent study, patient will be summarized in their randomized group in parent study, regardless of the treatment they actually received.

For change from baseline in efficacy endpoints, baseline will be same baseline as parent study. For summaries of efficacy endpoints, only observed case data will be used (no imputation for missing data).

LDL-C, HDL-C, TG, TC, non-HDL-C, apoB and hs-CRP values at week 0, Weeks 52, and 78 will be summarized based on the FAS. For each parameter at each time point, the value


of the parameter and the percent change from baseline in the parameter will be summarized by previous treatment group in parent study and overall in OLE study. Ninety-five percent (95%) CI will be provided for the estimates at week 0, Week 52 and 78 for the change values. Lipid and cardiometabolic data from all visits will be listed.

#### **5.4** Safety Data Endpoints and Analyses

No statistical analyses will be performed on any of the safety data in this study.

The safety and tolerability of ETC-1002 will be assessed by examination of TEAEs (including muscle related events and other AESI), physical exams, vital signs, electrocardiograms (ECGs), clinical laboratory values (serum chemistry, hematology, coagulation and urinalysis), and weight. All patients included in the SP will be evaluated in the safety analyses.

Unless otherwise stated, descriptive summaries will be displayed by previous treatment group actually received in parent study and overall and based on the SP.

#### 5.4.1 Adverse Events (AEs)

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 18.1 or later and will be categorized by system organ class (SOC) and preferred term (PT). Patients with AEs that are ongoing at study completion or study withdrawal must be followed until resolution or for 30 days after the last study visit, whichever comes first. Summary tables will focus on TEAEs; however, listings will include all AEs (with non-TEAEs flagged). An additional listing will be provided for AEs occurred during rollover period for patients who entered the study beyond the 30-day rollover window, if data available.

In summary tables, TEAEs will be counted as "Not Related" if relationship to study drug was recorded as 'Not Related' or "Unlikely". Events will be counted as "Related" if relationship to study drug was recorded as 'Possible', 'Probable', 'Definite' or if relationship to study drug is missing.

The severity of the AE will be characterized as mild, moderate, or severe, to the following definitions:

- Mild: Events are usually transient and do not interfere with the patient's daily activities
- Moderate: Events introduce a low level of inconvenience or concern to the patient and may interfere with daily activities
- Severe: Events interrupt the patient's usual daily activity, are incapacitating with inability to do usual activities, or significantly affect clinical status and warrant intervention and/or close follow-up

Overviews of TEAEs will be presented by previous treatment group in parent study and overall containing the following counts and percentages for:


- patients with TEAEs
- Patients with TEAEs occurred during the rollover period for patients entered the study beyond the 30 day rollover window (if available)
- patients with TEAEs by SOC and PT
- patients with TEAEs by maximum severity
- patients with treatment-related TEAEs
- patients with treatment-emergent serious adverse events (TE SAEs)
- patients with TE SAEs (TE SAEs) by SOC and PT
- patients with TE SAEs by maximum severity
- patients with treatment-related TE SAEs
- withdrawal from study drug due to TEAEs

In addition, summary tables will be provided, by prior treatment group and overall, for the number and percent of patients experiencing:

- investigator reported major adverse cardiovascular events and mortality (MACE) by event type
- adjudicated major adverse cardiovascular events and mortality (MACE) by event type
- non-CV deaths (non-MACE),
- nonfatal myocardial infarction [MI] (MACE),
- nonfatal stroke (MACE),
- hospitalization for unstable angina (MACE),
- coronary revascularization (MACE),
- noncoronary arterial revascularization (non-MACE),
- hospitalization for heart failure (non-MACE) using standardized definitions.

Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs as well as a clinical endpoint.

The AE overview summaries will count a patient at most once in each AE category (at the "highest/most extreme" designation of each category regardless of preferred term) and percentages will be based on the total number of patients in the safety population.

In addition to a comprehensive listing of all AEs (with non-TEAEs flagged), separate listings will be generated for SAEs, AEs resulting in withdrawal of study drug, and AEs with a fatal outcome, investigator reported major adverse cardiovascular events and mortality, and adjudicated major adverse cardiovascular events and mortality.

#### **5.4.2** Adverse Events of Special Interest

Across clinical studies to date, the most frequently reported TEAEs associated with the experiences with ETC-1002 included musculoskeletal and connective tissue disorders (back pain, pain in extremity, myalgia, arthralgia, and muscle spasms), nervous system disorders (headache), GI disorders (nausea and diarrhea), and infections and infestations.


Adverse events of special interest (AESI) include hepatic, muscular (AE and CK evaluation), new onset diabetes/glycemia, renal, cardiovascular, metabolic acidosis and hypoglycemia and neurocognitive/neurologic events. These events will be pulled out of the AE databases with help of clinical team by SOC and PT, and will be identified as safety monitoring endpoint.

- Hepatic safety will be assessed via liver-associated enzymes and TB.
- Musculoskeletal safety will be assessed via AEs involving muscle related symptoms, CPK laboratories will also be summarized.
- New onset diabetes/glycemia will be assessed via AEs and monitoring of glucose and HbA1c.
- Renal safety will be assessed via eGFR, CK and muscle-related AEs.
- Cardiovascular safety will be assessed via AEs (note that the AESI of cardiovascular safety is broader than the MACE assessment).
- Neurocognitive events will be assessed by routine monitoring of PE findings and AEs.
- Hypoglycemia will be assessed by routine clinical laboratories and summarized based on AE evaluations
- Metabolic acidosis occurrences will be monitored by routine laboratories and summarized based on AE evaluations.

AESI will be presented in a listing and summarized by SOC, PT and previous treatment group in parent study and overall in OLE study. Muscle-related TEAEs will be summarized by SOC, PT and baseline eGFR category.

#### 5.4.3 Clinical Cardiovascular Endpoints

Clinical cardiovascular endpoints will be monitored and adjudicated by an independent blinded expert CEC for this study and other ongoing studies the ETC-1002 program. Adjudicated clinical endpoints will be summarized by event type and previous treatment group in parent study and overall in OLE study. Additional details regarding clinical endpoints and clinical endpoint definitions will be included in CEC charter.

#### **5.4.4** Neurocognitive Events

Neurocognitive events will be identified and evaluated by routine safety monitoring of PE findings and AEs. Summarization of neurocognitive events will occur using pre-specified MedDRA terms and will be performed by SOC, severity, and relationship to study drug by previous treatment group in parent study and overall in OLE study.


#### **5.4.5** Laboratory Evaluations

Continuous laboratory parameters (serum chemistry, hematology, coagulation (only in patients receiving anticoagulant therapy that in the investigator's judgment require monitoring at Month 0 and 3 to 5 days post-Month 0), urinalysis, urinalysis [microscopic]) listed in Table 2; glucose, and HbA1c will be summarized using descriptive statistics for the observed value and the change from baseline. Missing values for any of the laboratory evaluations will not be imputed; that is, only observed case data will be used. Baseline is defined as the last value prior to the first dose of study medication in OLE study. Categorical urinalysis data will be listed, but will not be summarized.


**Table 2:** Clinical Laboratory Parameters (Safety)

| Clinical Laboratory Test | Clinical Laboratory Test |
|---|---|
| Hematology | Blood Chemistry (serum, fasting) |
| Hematocrit (Hct) | Albumin (Alb) |
| Hemoglobin (Hgb) | Alkaline phosphatase (ALK-P) |
| Mean corpuscular hemoglobin (MCH) | • Alanine aminotransferase (ALT; SGPT) |
| Mean corpuscular hemoglobin | <ul> <li>Aspartate aminotransferase (AST;</li> </ul> |
| concentration (MCHC) | SGOT) |
| Mean corpuscular volume (MCV) | Blood urea nitrogen (BUN) |
| Platelet count | • Calcium (Ca) |
| Red blood (RBC) cell count | • Carbon dioxide (CO2) |
| White blood (WBC) cell count with | • Chloride (Cl) |
| differential (absolute and %) | • Creatinine |
| <u>Urinalysis (Dipstick)</u> | • Creatine kinase (CK) |
| Clarity | Glucose |
| Bilirubin | Lactate dehydrogenase (LDH) |
| • Color | <ul> <li>Phosphorus</li> </ul> |
| • Glucose | Potassium (K) |
| • Ketones | Sodium (Na) |
| Leukocyte esterase | Total and direct bilirubin (TB)a |
| • Nitrate | Total protein |
| Occult blood | Uric acid |
| • pH | Coagulation—only in patients receiving |
| • Protein | anticoagulant therapy that in the investigator's |
| Specific gravity | judgment require monitoring at Month 0 and |
| Urobilinogen | 3 to 5 days post-Month 0 |
| | • Prothrombin time (PT) |
| | International normalized ration (INR) |
| Urinalysis (Microscopic)-only if urine dipstick | Other Labs: |
| <u>abnormal</u> | Urine pregnancy test |
| Bacteria | • Hemoglobin A <sub>1C</sub> (HbA <sub>1C</sub> ) |
| • Casts | |
| • Crystals | |
| Epithelial cells | |
| • RBC | |
| • WBC | |

<sup>&</sup>lt;sup>a</sup> If TB ≥1.2 × ULN, a reflex indirect (unconjugated) bilirubin will be obtained.

The number and percentage of patients with laboratory abnormalities (i.e., laboratory values outside the stated laboratory normal range) will be summarized at each time point Confidential


(i.e., including baseline and post-baseline time points) for each laboratory parameter. The determination of laboratory abnormalities will take into account any unscheduled laboratory assessments. Additional lab-related summaries will be provided as follows for hepatic safety, musculoskeletal safety, diabetes and glycemia, and renal safety.

#### **5.4.5.1** Hepatic Safety

For liver-associated enzymes and total bilirubin (TB), the number and percent of patients with abnormal values for ALT (>=  $3 \times ULN$ , >=  $5 \times ULN$ ), AST (>=  $3 \times ULN$ , >=  $5 \times ULN$ ), and TB (>=  $2 \times ULN$ ) will be summarized by overall, normal baseline ALT/AST/TB and abnormal baseline ALT/AST/TB.

Hy's law criteria ( $\geq 3 \times \text{upper limit of normal [ULN]}$  for either ALT or AST, with accompanying TB > 2 × ULN, with no other known cause) will also be applied to the data; any potential Hy's law cases will be listed separately. In the case of patients with Gilbert's disease, TB will be fractionated and the determination of 2 × ULN will be based upon direct (conjugated) bilirubin.

#### **5.4.5.2** Musculoskeletal Safety

CK levels will be summarized by the value and change from baseline in the value, by treatment group and visit as well as baseline eGFR category. In addition, the number and percent of patients with abnormal CK values ( $\geq 5$  X ULN,  $\geq 10$  × ULN) will be summarized. These summaries of patients with abnormal CK will be performed overall, normal baseline CK, and abnormal baseline CK.

#### 5.4.5.3 Diabetes and Glycemia

For fasting glucose and HbA1C (%), a shift table from baseline with the number and percent of patients will be categorized as below:

```
Fasting glucose: >= 126 mg/dL; 100-125 mg/dL, and < 100 mg/dL; HbA1C (%): >=6.5%; >5.5 to <=6.4% and <=5.5%.
```

#### 5.4.5.4 Renal Safety

Shift tables of eGFR category from baseline over the study, will be provided by treatment group. If needed, post-baseline eGFR categories will be modified to include the possibility of patients with eGFR values <45 mL/min/1.73m<sup>2</sup> (e.g., including <30 mL/min/1.73m<sup>2</sup> and updating to include moderate renal impairment to 30-59 mL/min/1.73m<sup>2</sup>).

In addition, renal function will be categorized as: (1) A creatinine change from baseline of > 1 mg/dL or occurrences of eGFR  $< 30 \text{mg/dL/m}^2$ ; (2) A Creatinine change <= 1 mg/dL from baseline ULN or eGFR  $>= 30 \text{ mg/dL/m}^2$ . A shift table from baseline with the number and percent of patients using the two categories will be presented.

Shift tables of urine protein (negative/positive) from baseline over the study, will be provided by treatment group. Values of CK over the study will be summarized by treatment group and by baseline eGFR category. Finally, muscle-related AEs will be summarized by treatment group and by baseline eGFR category.


#### 5.4.6 Physical Examinations (PEs)

Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant.' Baseline is defined as the last value prior to the first dose of study medication. Only changes from baseline physical examination findings that meet the definition of an AE will be recorded on the AE page of the eCRF and will be summarized with other AE outcomes.

#### 5.4.7 Vital Signs

Actual values and changes from baseline in vital signs (heart rate, systolic blood pressure, diastolic blood pressure, weight, height [baseline only], and BMI) will be summarized using descriptive statistics by treatment group and post-baseline time point. Baseline is defined as the last value prior to the first dose of study medication.

Vital signs data will be listed for each patient, with increases from baseline of >15 mmHg in systolic or diastolic blood pressure flagged.

#### 5.4.8 Electrocardiogram (ECG)

Shift tables for ECG data from baseline to end-of-study will be provided by treatment group. The data will be categorized as 'Normal'; 'Abnormal, not clinically significant'; and 'Abnormal, clinically significant.' Baseline is defined as the last value prior to the first dose of study medication. Listings of ECG data will include only those records where the baseline ECG was either 'Normal' or 'Abnormal, not clinically significant', but the end-of-study ECG was marked as 'Abnormal, clinically significant'.

## 6 DMC Analyses

Refer to DMC charter.

### 7 Reference

- 1. Sharrett AR, Ballantyne CM, Coady SA, Heiss G, Sorlie PD, Catellier D, et al. Atherosclerosis Risk in Communities Study Group. Coronary Heart Disease Prediction from Lipoprotein Cholesterol Levels, Triglycerides, Lipoprotein(A), Apolipoproteins A-I and B, and HDL Density Subfractions. The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2001;104:1108-13.
- 2. World Health Organization (WHO) Fact Sheet No 317 Updated January 2015.
- 3. Robinson JG. Management of Familial Hypercholesterolemia: A Review of the recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Managed Care Pharm. 2013;19(2):139-49.


- 4. Pharmacokinetics in Patients with Impaired Renal Function Study Design, Data Analysis, and Impact on Dosing and Labeling. FDA Draft Guidance. March 2010
- 5. Haase A, Goldberg AC. Identification of people with heterozygous familial hypercholesterolemia. Curr Opin Lipidol. 2012;23:282-9.
- 6. Glynn RJ, Laird NM, and Rubin DB. (1986). Selection modelling versus mixture modelling with nonignorable nonresponse. In H. Wainer (ed.), Drawing Inferences from Self-Selected Samples, pp. 115–142. New York: Springer.


## 8 Appendices

**Appendix 1: Schedule of Events (Subject Visit Schedule)** 

| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOS <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| Week | EOS | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 |
| | Parent | | | | | | |
| Visit Window | 30 Days<br>pre-M0 | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days |
| In-clinic Visit | X | X | | | X | | X |
| <b>Phone Visit</b> | | | X | X | | X | |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Enrollment Criteria | X | | | | | | |
| Medical History | X | | | | | | |
| Concomitant<br>Medications | X | X | X | X | X | X | X |
| Adverse Event<br>Recording | X | X | X | X | X | X | X |
| Physical Exam | X | | | | X | | X |
| Weight <sup>2</sup> | X | X | | | X | | X |
| Vital Signs <sup>3</sup> | X | X | | | X | | X |
| Urine Pregnancy Test | X | | | | | | |
| Clinical Safety Labs <sup>4</sup> | X | X | | | X | | X |
| Basic Fasting Lipids <sup>5</sup> | X | X | | | X | | X |
| Coagulation <sup>6</sup> | X | | | | | | |
| ApoB and hsCRP | X | X | | | X | | X |
| HbA <sub>1C</sub> | X | | | | X | | X |
| IWRS Contact <sup>7</sup> | X | X | | _ | X | | X |
| Drug Dispensing | X | X | | | X | | |
| Drug<br>Return/Compliance | | X | | | X | | X |

NOTE: For patients who withdraw from study drug treatment, but consent to be followed for safety assessments and return to clinic for these visit, the visits will occur according to the protocol schedule. Safety assessments should include clinical safety and basic lipid laboratories, adverse events (AEs), physical examination (PE), vital signs, and electrocardiograms (ECGs). For patients who withdraw from study drug treatment, but consent to be followed for safety assessments by phone, the telephone contacts will occur according the protocol schedule with information regarding current health status and to collect information on AEs (eg, recent procedures, hospitalizations, and if the patient has died, the cause of death). If a patient does not provide consent to be followed for safety assessments per the protocol (either by returning to clinic or by phone), Visit week 78 will be considered the End of Study (EOS)/Early Withdrawal from study and no further visits will be scheduled.

- 1 All procedures will be completed for all patients at either EOS if completing the study or early withdrawal.
- 2 Body weight will be measured in the morning while fasting, using consistent scales, after voiding, and without shoes and outerwear (eg, coats).
- 3 Vital signs will include diastolic blood pressure (DBP), systolic blood pressure (SBP), heart rate (HR) and will be collected prior to any blood sample collection. Patient will rest for 5 minutes prior to assessments
- 4 Clinical safety labs include hematology, blood chemistry, and urinalysis at all visits. Please refer to laboratory manual for detailed schedule of tests.
- 5 Basic fasting lipids include total cholesterol (TC), calculated low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-HDL-C,), and triglycerides (TG).


6 Only in patients receiving anticoagulant therapy that in the investigator's judgment require monitoring at Month 0 and 3 to 5 days post-Month 0

7 Interactive web response system (IWRS) contact at either an early withdrawal or an EOS visit to register study discontinuation visit date

#### Statistical Analysis Plan

Title: A MULTICENTER OPEN-LABEL EXTENSION (OLE) STUDY

TO ASSESS THE LONG-TERM SAFETY AND EFFICACY OF

BEMPEDOIC ACID (ETC-1002) 180 MG

**Protocol:** ETC-1002-050

Clinical Phase: 3

**Product:** ETC-1002

**Version (Date):** Statistical Analysis Plan – Version 1.1

**Status:** Final





REASON: I approve this document as author.

5e9eb6ba-ac95-46d1-aa92-422b0263855d





REASON: I approve this document e2f1bc36-0729-4d08-8328-dde7950d0dd1

Esperion Therapeutics

REASON: I approve this document fdfe4eec-c142-42c7-bf98-459047a30340

Date

**Esperion Therapeutics** 


22 Oct 2018 19:07:045+0000

### **Table of Contents**

| 1 | List of A | Abbreviations | . 4 |
|---|---|---|---|
| 2 | Introduc | tion | . 7 |
| 3 | | bjectives and Endpoints | |
| | 3.1 Obje | ectives | . 7 |
| | | nary Endpoint | |
| | | ondary Endpoints | |
| | 3.3.1 | Adverse Events | |
| | 3.3.2 | Clinical Safety Laboratories | . 8 |
| | 3.3.3 | Vital Signs | |
| | | PE (Physical Exam) | |
| | 3.4 Lipi | ds | . 8 |
| | 3.5 Phan | rmacokinetic (PK) and Other Biomarkers | . 8 |
| 4 | | esign | |
| | 4.1 Stud | ly Design | . 9 |
| | 4.2 Stud | ly Treatments and Assessments | . 9 |
| | 4.3 Ran | domization and Blinding | 11 |
| | 4.4 Sam | ple Size Justification | 11 |
| | 4.5 Inter | rim Analyses, Final Analyses and Unblinding | 11 |
| | | nge from Planned Analyses | |
| 5 | Statistica | al and Analytical Plans | 11 |
| | 5.1 Gen | eral Statistical Considerations | 11 |
| | 5.2 Stati | istical Analysis Plans | 13 |
| | 5.2.1 | Analysis Sets | 13 |
| | 5.2.1. | Safety Population (SP) | 13 |
| | 5.2.1. | 2 Completer Analysis Set (CAS) | 13 |
| | 5.2.2 | Protocol Violations and Deviations | |
| | 5.2.3 | Subject Disposition | 13 |
| | 5.2.4 | Demographic and Baseline Characteristics | 13 |
| | 5.2.5 | Subgroup Variables | 14 |
| | 5.2.6 | Medical History | 14 |
| | 5.2.7 | Concomitant Medications | 15 |
| | 5.2.8 | Study Drug Exposure and Compliance | 15 |
| | 5.3 Efficient | cacy Endpoints and Analyses | 15 |
| | 5.4 Safe | ety Data Endpoints and Analyses | 16 |
| | 5.4.1 | Adverse Events (AEs) | 16 |
| | 5.4.2 | Adverse Events of Special Interest | |
| | 5.4.3 | Clinical Cardiovascular Endpoints | 18 |
| | 5.4.4 | Neurocognitive Events | 18 |
| | 5.4.5 | Laboratory Evaluations | 18 |
| | 5.4.5. | 1 Hepatic Safety | 21 |
| | 5.4.5. | 2 Musculoskeletal Safety | 21 |
| | 5.4.5. | 3 Diabetes and Glycemia | 21 |
| | | the control of the co | |


## Version 1.1, Oct 19, 2018 Statistical Analysis Plan

| | 5.4. | 5.4 Renal Safety | 21 |
|---|---|---|---|
| | | Physical Examinations (PEs) | |
| | | Vital Signs | |
| 6 | | Analyses | |
| 7 Reference | | | |
| | | dices | |
| | 11 | opendix 1: Schedule of Events (Subject Visit Schedule) | |
| | - | opendix 2: Adverse Event of Special Interest (AESI) | |
| | | 1 / | |


## 1 List of Abbreviations

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|-----------------------------------------|
| ACL | Adenosine triphosphate-citrate lyase |
| ACS | Acyl-CoA synthetase |
| ADR | Adverse drug reaction |
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ALB | Albumin |
| ALK-P | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| ApoB | Apolipoprotein B |
| ASCVD | Atherosclerotic cardiovascular diseases |
| AST | Aspartate aminotransferase |
| ATP | Adenosine triphosphate |
| AUC | Area under the concentration-time curve |
| AUC <sub>0-24</sub> | Area under the curve during 24 hours |
| BMI | Body mass index |
| BP | Blood pressure |
| BUN | Blood urea nitrogen |
| Ca | Calcium |
| CAS | Completer Analysis Set |
| CEC | Clinical Event Committee |
| CFR | Code of Federal Regulations |
| CHD | Coronary heart disease |
| CI | Confidence interval |
| CK | Creatine kinase |
| Cl | Chloride |
| CNS | Central nervous system |
| CoA | Acetyl-coenzyme A |
| CO <sub>2</sub> | Carbon dioxide |
| CV | Cardiovascular |
| CYP | Cytochrome P450 |
| DBP | Diastolic blood pressure |
| DMC | Data Monitoring Committee |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| eGFR | Estimated glomerular filtration rate |
| EMA | European Medicines Agency |
| EOS | End of Study |


| Abbreviation or Specialist Term | Explanation |
|---|---|
| ETC-1002 | Bempedoic acid |
| EU | European Union |
| FDA | Food and Drug Administration |
| FPFV | First patient first visit |
| FSH | Follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GI | Gastrointestinal |
| HbA <sub>1C</sub> | Glycosylated hemoglobin, Type A <sub>1C</sub> |
| HBsAg | Hepatitis B surface antigen |
| Hct | Hematocrit |
| HCV | Hepatitis C virus |
| HDL-C | High-density lipoprotein cholesterol |
| HeFH | Heterozygous familial hypercholesterolemia |
| Hgb | Hemoglobin |
| HMG-CoA | 3-hydroxy-3-methylglutaryl-coenzyme A |
| hs-CRP | High-sensitivity C-reactive protein |
| IB | Investigator's Brochure |
| ICD | Informed Consent Document |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IMP | Investigational medicinal product |
| IND | Investigational New Drug Application |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| ITT | Intention-to-treat |
| IUD | Intrauterine device |
| IWRS | Interactive web response system |
| K | Potassium |
| LDH | Lactate dehydrogenase |
| LDL-C | Low-density lipoprotein cholesterol |
| LDLR | LDL receptor |
| LFT | Liver function test |
| LPLV | Last patient last visit |
| LS | Least square |
| MACE | Major adverse cardiac event |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean corpuscular volume |


DocUUID : 56c02f8e-9400-4951-9733-c0dc2889592d

| Abbreviation or Specialist Term | Explanation |
|---|---|
| MDRD | Modification of diet in renal disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Myocardial infarction |
| MRI | Magnetic resonance imaging |
| Na | Sodium |
| NA | Not applicable |
| NLA | National Lipid Association |
| NOAEL | No-observed-adverse-effect level |
| non-HDL-C | Non-high-density lipoprotein cholesterol |
| OLE | Open-label extension (study) |
| Parent study | Study 1002-040 |
| PCSK9 | Proprotein convertase subtilisin/kexin type 9 |
| PE | Physical exam |
| PK | Pharmacokinetic(s) |
| PT | Prothrombin time |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SOC | System organ class |
| SP | Safety population |
| SUSARS | Suspected and unexpected serious adverse reactions |
| T2DM | Type 2 diabetes mellitus |
| TB | Total bilirubin |
| TC | Total cholesterol |
| TEAE | Treatment-emergent adverse event |
| TG | Triglycerides |
| TQT | Thorough QT/QTc |
| ULN | Upper limit of normal |
| US | United States |
| WBC | White blood cell |
| WHO | World Health Organization |


DocUUID : 56c02f8e-9400-4951-9733-c0dc2889592d

#### 2 Introduction

The purpose of this document is to describe the statistical methods, data derivations and data summaries to be employed in ETC-1002-050. The preparation of this statistical analysis plan (SAP) has been based on International Conference on Harmonisation (ICH) E3 and E9 Guidelines and in reference to Protocol ETC-1002-050 (Protocol Amendment 2, 10 May 2017).

The SAP will supersede the protocol in the event of any differences between the two documents in the plans for data analysis, and the protocol will be amended if appropriate. The SAP will be included as an appendix in the clinical study report for this protocol.

## 3 Study Objectives and Endpoints

### 3.1 Objectives

- The primary objective for this study is to characterize the safety and tolerability of long-term administration of bempedoic acid (ETC-1002) 180 mg
- The secondary objective is to characterize the efficacy of long-term administration of bempedoic acid 180 mg/day as assessed by changes in low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-high-density lipoprotein cholesterol (non-HDL-C), apolipoprotein B (ApoB), total cholesterol (TC), triglycerides TG and high-sensitivity C-reactive protein (hs-CRP) in patients with hyperlipidemia

## 3.2 Primary Endpoint

• The primary endpoint for this study is patient incidence of AEs

## 3.3 Secondary Endpoints

- Percent change from baseline in LDL-C at Weeks 52 and 78
- Change from baseline in LDL-C at Weeks 52 and 78
- Percent change from baseline in non-HDL-C at Weeks 52 and 78
- Percent change from baseline in TC at Weeks 52 and 78
- Percent change from baseline in ApoB at Weeks 52 and 78
- Percent change from baseline in hs-CRP at Weeks 52 and 78
- Percent change from baseline in TG at Weeks 52 and 78
- Percent change from baseline in HDL-C at Weeks 52 and 78


#### 3.3.1 Adverse Events

The evaluation of AEs will include only incidence of treatment-emergent AEs (TEAEs), defined as AEs that begin or worsen on or after the date of first dose of study drug administration in OLE period and until 30 days after last dose of study drug. Clinical endpoints (details see section 4.2) will be collected and adjudicated by an independent Clinical Events Committee (CEC). Clinical endpoints will also be reported as SAEs. Adverse events of special interest (AESI) will further be examined (See Section 5.4.2 for more information).

#### 3.3.2 Clinical Safety Laboratories

The evaluation of clinical safety laboratories, including blood hematology, chemistry, coagulation, and urinalysis, will be based on the observed values. Observed values, changes and percent change from baseline of both the parent study and OLE study will be summarized for all post-baseline study visits.

#### 3.3.3 Vital Signs

The evaluation of vital signs (including heart rate, systolic blood pressure, diastolic blood pressure, height, and weight will be based on the observed values. For vital signs, observed values, and changes from baseline of both the parent study and OLE study will be summarized for all post-baseline study visits.

#### 3.3.4 PE (Physical Exam)

Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant.'

### 3.4 Lipids

After enrollment, patients will return to clinic at week 12, 52, 78/EOT and 82/EOS. Clinical laboratory samples will be collected and analyzed for calculated LDL-C and lipid and cardiometabolic biomarkers including non-HDL-C, HDL-C, TC, ApoB, and TG at baseline and all clinic visits for evaluation of bempedoic acid effects on lipids and cardiometabolic parameters.

## 3.5 Pharmacokinetic (PK) and Other Biomarkers

NA.

## 4 Study Design

#### 4.1 Study Design

This is a multicenter OLE study designed to assess the long-term safety and efficacy of bempedoic acid (ETC-1002) 180 mg. All patients will receive open-label bempedoic acid 180 mg for up to 1.5 years after rolling over from the parent study (Study 1002-040) followed by a follow-up period off study drug for 4 weeks. Investigators, site staff, patients, and the study team will be masked to study lipid levels until the Week 12 study visit, after which time lipid values will be made available.

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other ongoing studies of bempedoic acid. A blinded independent expert Clinical Events Committee (CEC) will adjudicate designated clinical endpoints across the program, including all major adverse cardiac events (MACE) and non-MACE endpoints defined as: cardiovascular (CV) death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction [MI] (MACE), nonfatal stroke (MACE), hospitalization for unstable angina (MACE), coronary revascularization (MACE), noncoronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE) using standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs as well as a clinical endpoint.

The study will be conducted at approximately 125 clinical sites in the United States, Canada, Germany, Netherlands, Poland, and United Kingdom. The study will end when the last randomized patient completes their last study visit (last patient last visit [LPLV] for last randomized patient). The estimated overall duration of the study (first patient first visit [FPFV] to LPLV) is approximately 2.5 years.

Parent Study
Patients on ETC-1002
or Placebo and
Background Therapy

1.5 Years

4 weeks
Washout

Figure 1. Study 1002-040 Study Design

### 4.2 Study Treatments and Assessments

Day 1 for this study should occur on the same day as the end of study visit for the parent study (1002-040). Patients who provide informed consent and sign the ICD will be eligible to enroll in the study.

The schedule of study events is provided in Appendix 1. However, a patient can be seen at any time for reasons of safety.


The investigational products were listed in Table 1 below:

**Table 1: Investigational Medicinal Products** 

| | Investigational Medicinal Product |
|---|---|
| <b>Product Name:</b> | Bempedoic acid |
| Dosage Form: | Film-coated tablets |
| Unit Dose: | 180 mg |
| Container/Closure <sup>a</sup> | 100-count bottle with screw on, child proof cap |
| Route of Administration: | Oral, daily with or without food |
| Physical Description: | |
| Manufacturer<br>(Fill/Finish): | |

Study drug should be taken once a day (once every 24 hours) at approximately the same time every day and may be taken with or without food. Patients will fast (no food or drink, other than water) for a minimum of 10 hours prior to collection of all laboratory samples.

Please see Pharmacy Manual for detailed storage requirements and instructions.

Patients who withdraw from investigational medicinal product (IMP) treatment will be asked to continue to be followed for safety using the protocol-specified visit schedule and procedures. For details of study assessments, see Appendix 1: Schedule of Events (Subject Visit Schedule).

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other any ongoing studies of ETC-1002. All clinical endpoints, including all major cardiac events (MACE) and non-MACE endpoints defined as: CV death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction (MI) (MACE), nonfatal stroke (MACE), hospitalization for unstable angina (MACE), coronary revascularization (MACE), non-coronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE), will be adjudicated by an independent blinded expert Clinical Events Committee (CEC), using


standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs.

### 4.3 Randomization and Blinding

- Randomization is not applicable for this OLE study.
- Laboratory results for lipid panel and hs-CRP will be masked to investigators, patients, and the study team until the Week 12 visit is completed. All site staff involved with this trial should refrain from obtaining lipid panels between date of last study medication (bempedoic acid or placebo) dose at end of parent study Week 52 (Visit T7) and Week 12 in this OLE trial.

### 4.4 Sample Size Justification

The number of patients entering this study will depend on the number of patients completing Study 1002-040 and their willingness to enroll.

### 4.5 Interim Analyses, Final Analyses and Unblinding

An interim analysis will be conducted in 2H, 2018 in order to provide safety assessment to support NDA submission. Another interim analysis for Day120 safety update will be approximately 120 days after the NDA cutoff. The endpoints and analyses are the same as the defined in final analysis if applicable.

The final analysis will be performed after the database is locked, and the database released.

## 4.6 Change from Planned Analyses

There is no change from planned analyses for this study.

## 5 Statistical and Analytical Plans

#### 5.1 General Statistical Considerations

The treatment groups will be displayed as previous treatment in parent study as well as overall treatment group in OLE study.

In general, all safety and efficacy data will be reported as observed. No imputation will be performed for missing data. Descriptive statistics (n, mean, standard deviation [SD] or Standard Error [SE], median, Q1, Q3, minimum, and maximum) will be calculated for continuous data. Minimum and maximum will be presented same number of decimal places as reported/collected, one additional decimal place for mean and median, and two additional decimal places for SD.


Categorical data will be summarized using n and percentage based on number of non-missing values. Percentage will be presented with one decimal place. The number of missing values will be presented as a separate category with no percentage, but only if 1 or more patients are missing data for the summary. Otherwise, all categories will be presented (even if no patients are counted in the category). Counts of zero in any category will be presented without percentage. Ninety-five percent (95%) confidence intervals (CIs) will be calculated for select continuous and categorical endpoint estimates. All patients will be summarized together as well as by their prior treatment group in the parent study.

Data will be presented on listings in order of patient/subject, assessment date and assessment (in order collected on CRF, unless specified otherwise). Dates will be presented in format DDMMMYYYY.

Relative day calculations will be [date of interest – relative date + (date of interest >= relative date)]. This calculation will result in dates prior to the relative date being presented as negative days, and those occurring on or after the relative date as Day 1 or later, i.e., there will be no Day 0.

Two sets of baseline are defined for any laboratory parameters and vital signs: baseline in parent study (1002-040) and baseline in OLE study (1002-050). The parent baseline values will be directly extracted from parent study database and baseline for the OLE study is defined as the last non-missing value on or prior to the date of first dose in the OLE. If last dose of study treatment is missing, then the date of last visit at which study assessments were obtained on CRF will be used in its place.

The visit schedules and window are shown below.

| Visit | Day 1/Week 0 | Week<br>12 | Week 24 | Week 36 | Week 52 | Week 64 | Week<br>78/EOT | Week<br>82/EOS |
|---|---|---|---|---|---|---|---|---|
| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOT | 19/EOS |
| Slotted Study<br>Week | EOS Parent | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 | Wk 82 |
| Target Study<br>Day | 1 | 84 | 168 | 252 | 364 | 448 | 546 | 574 |
| Analysis<br>Window | 1 | [2,126] | [127,210 | [211,308 | [309,406 | [407,497<br>] | [498,562<br>] | [563,∞] |
| Protocol<br>defined visit<br>Windows | [30 Days, Pre<br>M0] | 84±7 | 168±7 | 252±7 | 364±7 | 448±7 | 546±7 | 574±14 |

### 5.2 Statistical Analysis Plans

#### 5.2.1 Analysis Sets

#### 5.2.1.1 Safety Population (SP)

The Safety Population (SP) is defined as all enrolled patients who received at least 1 dose of bempedoic acid during the OLE period and will be used for demographics and baseline characteristics, treatment exposure, concomitant medications, and all safety summaries.

#### 5.2.1.2 Completer Analysis Set (CAS)

The completer analysis set is defined as patients who completed the full 78 weeks treatment as per end of treatment CRF page.

#### 5.2.2 Protocol Violations and Deviations

A full list of protocol violations and deviations will be compiled and reviewed by the clinical team to identify key versus non-key violations/deviations before final database lock. For violations at study entry, patients will be assessed against the inclusion and exclusion criteria of the protocol. For on-study deviations, compliance with the protocol will be examined with regard to prohibited therapies, and timing and availability of planned assessments. The final list of protocol deviation will be approved by the study team prior to interim analysis cutoff or database lock and will be used to generate the PD deviation summary and listing.

### 5.2.3 Subject Disposition

The number of patients enrolled, and included in each analysis population, along with IMP and study completion status, will be summarized by the treatment group in parent ETC-1002-040 study and overall. In addition, the number of patients who withdraw from the study and withdraw from study drug will be summarized by discontinuation reason.

#### 5.2.4 Demographic and Baseline Characteristics

Demographic collected from the parent study will be used for this study. Two sets of baseline values will be defined: baseline of parent study and OLE study. The parent study baseline will be taken directly from the parent study, and the OLE baseline is defined as last non-missing value prior to the first dose of IMP in the OLE study. The following demographic and two sets of baseline characteristics will be summarized by previous treatment group in parent study, as well as overall, for safety population:

age group (18-40, 41-64, 65-74, and >=75), gender, race, ethnicity, region (North America, and EU), height (cm), weight (kg), body mass index (kg/m<sup>2</sup>) ( $< 25, 25 - < 30, \ge 30 \text{ kg/m}^2$ ), waist circumference, systolic and diastolic blood pressure, fasting lipid parameters (TC, LDL-C, HDL-C, non-HDL-C and TG), apoB, hs-CRP).


Cardiovascular risk factors from the parent study: ASCVD (Yes/No), HeFH (Yes/No), baseline statin intensity (derived) (low or moderate, high), eGFR category, tobacco history, alcohol history, history of diabetics, history of hypertension.

Data will be summarized using descriptive statistics for continuous variables and using counts and percentages for categorical variables.

The estimated glomerular filtration rate (eGFR) categories are: normal: ≥90 mL/min/1.73m<sup>2</sup>; mild Renal Impairment: 60-89 mL/min/1.73m<sup>2</sup>; moderate Renal Impairment: 30-59 mL/min/1.73m<sup>2</sup>, and severe Renal Impairment (15-29 mL/min/1.73m<sup>2</sup>).

### **5.2.5** Subgroup Variables

Subgroups defined by below variables will be evaluated for safety and the LDL-C efficacy endpoint.

- 1) Gender (male vs. female)
- 2) Age (< 65 yrs. vs.  $\ge 65$  yrs. and < 75 yrs. vs.  $\ge 75$  yrs.)
- 3) Baseline CVD risk category (HeFH (with/without ASCVD) vs. ASCVD only)
- 4) Baseline statin intensity (low vs. moderate vs. high)
- 5) Race (White vs. other)
- 6) Baseline LDL category (< 100 mg/dL vs. ≥100 mg/dL) (efficacy only)
- 7) History of diabetes (yes vs. no)
- 8) Body Mass Index (BMI) ( $< 25, 25 < 30, \ge 30 \text{ kg/m}^2$ )
- 9) Region (North America, EU)

In case the number of patients within a subgroup is too small, e.g. less than 5% of the overall population, the analyses may not be performed or the subgroup levels may be combined.

#### 5.2.6 Medical History

General medical history, cardiovascular history/risk factors, previous statin use and statin tolerance history will be summarized by previous treatment group in parent study, as well as overall in OLE study for safety population and presented in a by-patient listing. Where appropriate, terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 or later.

If a patient is entering the study beyond the 30 day rollover window, new medical history that occur between more than 30 days after the end of the parent study and treatment start in OLE study (exclusive) that period will be collected and presented in a by-patient listing.

#### **5.2.7** Concomitant Medications

Concomitant medications are defined as medications that were ongoing at the time of study drug initiation in this OLE study or new medications that started post study drug initiation and within 30 days following the date of the last dose of study drug.

Medications, including lipid modifying therapy (LMT) medications, will be coded using WHO Drug (March, 2017, or later if appropriate). The frequency of use of concomitant medications will be summarized by previous treatment group in parent study, as well as overall in OLE study, for the safety population according to Anatomical Therapeutic Chemical (ATC) class and preferred term. Concomitant medications will be listed for each patient. Concomitant LMT medications will be summarized by ATC class and medication name and listed separately in a similar fashion.

#### 5.2.8 Study Drug Exposure and Compliance

The length of exposure to study drug will be calculated as the number of days from the first dose of study drug to the last dose of study drug, regardless if the patient missed one or more doses of study drug. Length of exposure in OLE study will be summarized by previous treatment group in parent study and overall in OLE study using descriptive statistics for the safety population.

The number and percentage of patients who were compliant with taking study drug will be summarized by previous treatment group in parent study and overall in OLE study for the safety population using the following categories 0 - <80%; >= 80%. Overall compliance will be calculated as: 100\* (Total Number of Tablets Dispensed – Total Number of Tablets Returned) / (Treatment Duration in Days).

The study drug administration and compliance data, including reasons for poor compliance, will be listed for each patient.

## 5.3 Efficacy Endpoints and Analyses

Given the primary objective of the study being long term safety, efficacy analyses will be using the safety population (SP). The efficacy data will be summarized by previous treatment group in parent study as well as an overall group.

For each efficacy parameter, descriptive summary statistics at each visit will be provided for the actual value, change from baseline and percent change from baseline for both conventional and International System of Units (SI). Two sets of summaries will be provided using the baseline from the parent study and from the OLE study. The visits to be included in the overtime summary are baseline of parent study (1002-040), baseline of OLE study, week 12, week 52, week 78, and Week 82. There will be no imputation for missing data, all summaries will use observed data. Ninety-five percent (95%) CI will be provided for the estimates at post-baseline visits.


In addition, efficacy parameters will also be summarized using the Completer Analysis Set (CAS).

For LDL-C, Same descriptive summary statistics at each visit will be provided within subgroups for the actual value, change from baseline and percent change from baseline.

Efficacy data (actual value, change and percent change from baseline) from all visits will be presented using descriptive statistics using both conventional and standard units.

Figures (mean+/-se or median/IQR) supporting the summary tables will be provided for each efficacy parameter. Efficacy data from all visits will be provided in listings as well.

## 5.4 Safety Data Endpoints and Analyses

The safety and tolerability of ETC-1002 will be assessed by examination of TEAEs, physical exams, vital signs, clinical laboratory values (serum chemistry, hematology, coagulation and urinalysis), and weight. SP will be used for all safety analyses.

Unless otherwise stated, descriptive summaries will be displayed by previous treatment group actually received in parent study and overall group.

#### 5.4.1 Adverse Events (AEs)

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 or later and will be categorized by system organ class (SOC) and preferred term (PT). Summary tables will focus on TEAEs; however, listings will include all AEs (with non-TEAEs flagged). An additional AE listing will be provided for AEs occurred during rollover period (i.e. after completion of the parent Study, ETC1002-040 but < 30 days prior to providing consent for Study 1002-050.

In summary tables, TEAEs will be counted as "Not Related" if relationship to study drug was recorded as 'Not Related' or "Unlikely". Events will be counted as "Related" if relationship to study drug was recorded as 'Possible', 'Probable', 'Definite' or if relationship to study drug is missing.

The severity of the AE will be characterized as mild, moderate, or severe, to the following definitions:

- Mild: Events are usually transient and do not interfere with the patient's daily activities
- Moderate: Events introduce a low level of inconvenience or concern to the patient and may interfere with daily activities
- Severe: Events interrupt the patient's usual daily activity, are incapacitating with inability to do usual activities, or significantly affect clinical status and warrant intervention and/or close follow-up


Overviews of TEAEs will include total number of TEAEs and patient incidence of TEAE, TE SAE, related TEAE, related TE SAE, withdrew due to TEAE, AE with fatal outcome. Individual TEAE summary will be presented by previous treatment group in parent study and overall containing the following counts and percentages for:

- patients with TEAEs
- patients with TEAE by PT
- patients with TEAEs by SOC, PT and maximum severity
- patients with treatment-related TEAEs
- patients with treatment-related TEAEs by PT
- patients with treatment-related TEAEs by SOC and PT
- patients with treatment-emergent serious adverse events (TE SAEs)
- patients with TE SAEs by PT
- patients with TE SAEs by SOC, PT and maximum severity
- patients with treatment-related TE SAEs
- patients with treatment-related TE SAEs by SOC and PT
- TEAEs leading to discontinuation of IMP
- Fatal AEs by SOC and PT

In addition, summary tables will be provided, by prior treatment group and overall, for the number and percent of patients experiencing:

- adjudicated major adverse cardiovascular events and mortality (MACE) by event type
- non-CV deaths (non-MACE),
- nonfatal myocardial infarction [MI] (MACE),
- nonfatal stroke (MACE),
- hospitalization for unstable angina (MACE),
- coronary revascularization (MACE),
- noncoronary arterial revascularization (non-MACE),
- hospitalization for heart failure (non-MACE) using standardized definitions.

The TEAE, related TEAE, TE SAE, and AESI summaries by SOC, PT and maximum severity will be provided for relevant subgroups described in 5.2.5 with the exception of baseline LDL category.

The AE overview summaries will count a patient at most once in each AE category (at the "highest/most extreme" designation of each category regardless of preferred term) and percentages will be based on the total number of patients in the safety population.

In addition to a comprehensive listing of all AEs (with non-TEAEs flagged), separate listings will be generated for SAEs, AEs resulting in withdrawal of study drug, and AEs with a fatal


outcome, investigator reported major adverse cardiovascular events and mortality, and adjudicated major adverse cardiovascular events and mortality.

#### **5.4.2** Adverse Events of Special Interest

Adverse events of special interest (AESI) will be identified based a pre-defined list of preferred terms provided by the sponsor (Appendix 2).

AESI will be presented in a listing and summarized by SOC, PT and previous treatment group in parent study and overall in OLE study.

In addition to adverse events, AESI is also being evaluated based on safety lab parameters. The details are provided in 5.4.5.

### 5.4.3 Clinical Cardiovascular Endpoints

Clinical cardiovascular endpoints will be monitored and adjudicated by an independent blinded expert CEC for this study and other ongoing studies the ETC-1002 program. Positively adjudicated clinical endpoints that are treatment-emergent will be summarized by event type and previous treatment group in parent study and overall in OLE study. All events that were adjudicated will be provided in a listing. Additional details regarding clinical endpoints and clinical endpoint definitions will be included in CEC charter.

#### **5.4.4** Neurocognitive Events

Neurocognitive events will be identified and evaluated by routine safety monitoring of PE findings and AEs. Summarization of neurocognitive events will occur using pre-specified MedDRA terms and will be performed by SOC, severity, and relationship to study drug by previous treatment group in parent study and overall in OLE study.

#### 5.4.5 Laboratory Evaluations

Two sets of baseline for safety parameters are defined, similar to that for the efficacy parameters, baseline from the parent study and the baseline from the OLE study.

Continuous laboratory parameters (serum chemistry, hematology, coagulation (only for those patients receiving anti-coagulation), urinalysis, urinalysis [microscopic]) listed in Table 4 will be summarized using descriptive statistics at each scheduled visit starting from the baseline of the parent study. The similar on-treatment and completer analysis set approach for efficacy analysis described in section 5.3 will be used for safety laboratory analysis. All analysis will use conventional unit and SI unit will be provided for selected parameters.

Fasting serum glucose and HbA1c will be summarized using descriptive statistics for the observed value and the change, percent change from baseline by history of diabetics. Missing


values for any of the laboratory evaluations will not be imputed; that is, only observed case data will be used.

Categorical urinalysis data will be listed, but will not be summarized.

As part of the AESI evaluation, below safety lab abnormality will be summarized by treatment group. All post-baseline lab values during the on-treatment period are being considered. Further details are provided in Section 5.4.6.1 through 5.4.6.4.

- ALT or AST (> 3x ULN and >5xULN)
- TB (> 2x ULN)
- Potential Hy's Law case: (ALT and/or AST > 3xULN with concurrent TB > 2xULN)
- CK (> 5x ULN) and (>10x ULN)
- Fasting Serum Glucose (mg/dL) ( $\leq$ 50, and  $\geq$ 126) by history of diabetics
- HbA1C ( $\geq$ 6.5%) by history of diabetics
- Creatinine (change from baseline for >1 mg/dL)
- eGFR (< 15 mL/min/1.73m2, 15 -< 30 mL/min/1.73m2)
- Hgb (g/dL) (decrease from baseline for  $\geq 2$  g/dL)
- Hgb (<8 g/dL)


**Table 2:** Clinical Laboratory Parameters (Safety)

| Clinical Laboratory Test | Clinical Laboratory Test |
|---|---|
| <ul> <li>Clinical Laboratory Test</li> <li>Hematology</li> <li>Hematocrit (Hct)</li> <li>Hemoglobin (Hgb)</li> <li>Mean corpuscular hemoglobin (MCH)</li> <li>Mean corpuscular hemoglobin concentration (MCHC)</li> <li>Mean corpuscular volume (MCV)</li> <li>Platelet count</li> <li>Red blood (RBC) cell count</li> <li>White blood (WBC) cell count with differential (absolute and %)</li> <li>Urinalysis (Dipstick)</li> <li>Clarity</li> <li>Bilirubin</li> </ul> | Clinical Laboratory Test Blood Chemistry (serum, fasting) Albumin (Alb) Alkaline phosphatase (ALK-P) Alanine aminotransferase (ALT; SGPT) Aspartate aminotransferase (AST; SGOT) Blood urea nitrogen (BUN) Calcium (Ca) Carbon dioxide (CO2) Chloride (Cl) Creatinine Creatine kinase (CK) Glucose |
| <ul> <li>Color</li> <li>Glucose</li> <li>Ketones</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Occult blood</li> <li>pH</li> <li>Protein</li> <li>Specific gravity</li> <li>Urobilinogen</li> </ul> | <ul> <li>Lactate dehydrogenase (LDH)</li> <li>Phosphorus</li> <li>Potassium (K)</li> <li>Sodium (Na)</li> <li>Total and direct bilirubin (TB)a</li> <li>Total protein</li> <li>Uric acid</li> <li>Coagulation—only in patients receiving anticoagulant therapy that in the investigator's judgment require monitoring at Month 0 and 3 to 5 days post-Month 0</li> <li>Prothrombin time (PT)</li> <li>International normalized ration (INR)</li> </ul> |
| Urinalysis (Microscopic)-only if urine dipstick abnormal Bacteria Casts Crystals Epithelial cells RBC WBC | Other Labs: Urine pregnancy test Hemoglobin A <sub>1C</sub> (HbA <sub>1C</sub> ) |

<sup>&</sup>lt;sup>a</sup> If TB ≥1.2 × ULN, a reflex indirect (unconjugated) bilirubin will be obtained.


DocUUID : 56c02f8e-9400-4951-9733-c0dc2889592d

The number and percentage of patients with laboratory abnormalities (i.e., laboratory values outside the stated laboratory normal range) will be summarized at each time point (i.e., including baseline and post-baseline time points) for each laboratory parameter. The determination of laboratory abnormalities will take into account any unscheduled laboratory assessments. Additional lab-related summaries will be provided as follows for hepatic safety, musculoskeletal safety, diabetes and glycemia, and renal safety.

#### 5.4.5.1 Hepatic Safety

For liver-associated enzymes and total bilirubin (TB), the number and percent of patients with abnormal values for ALT (>3 × ULN, > 5 × ULN), AST (> 3 × ULN, > 5 × ULN), and TB (> 2×ULN) will be summarized by overall, normal baseline ALT/AST/TB and abnormal baseline ALT/AST/TB.

Hy's law criteria (>3 × upper limit of normal [ULN] for either ALT or AST, with accompanying TB > 2 × ULN) will also be applied to the data; any potential Hy's law cases will be listed separately. In the case of patients with Gilbert's disease, TB will be fractionated and the determination of  $2 \times ULN$  will be based upon direct (conjugated) bilirubin.

A separate listing for direct TB will be provided for those who have Gilbert's syndrome.

#### 5.4.5.2 Musculoskeletal Safety

CK levels will be summarized by the value and change from baseline in the value, by treatment group and visit as well as baseline eGFR category. In addition, the number and percent of patients with abnormal CK values (>5 X ULN, >10 × ULN) will be summarized. These summaries of patients with abnormal CK will be performed overall, normal baseline CK, and abnormal baseline CK.

#### 5.4.5.3 Diabetes and Glycemia

For fasting glucose and HbA1C (%), a shift table from baseline of both parent study and OLE study with the number and percent of patients will be categorized as below:

```
Fasting glucose: >= 126 mg/dL; 100-125 mg/dL, and < 100 mg/dL; HbA1C (%): >=6.5%; >5.5 to <=6.4% and <=5.5%.
```

These tables will be summarized by history of Diabetes.

Descriptive summary for fasting serum glucose and HbA1C will be provided by history of diabetics, previous treatment group in parent study and overall at each scheduled visit.

#### 5.4.5.4 Renal Safety

Shift tables of eGFR category from baseline of both parent study and OLE study over the study, will be provided by previous treatment group in parent study and overall.


In addition, renal function abnormality will be identified as: (1) A creatinine change from baseline of > 1 mg/dL (2) eGFR value <30 mL/min/1.73m2. A shift table from baseline of both parent study and OLE study with the number and percent of patients using the two categories will be presented.

#### 5.4.6 Physical Examinations (PEs)

Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant'. Baseline is defined as the last value prior to the first dose of study medication in OLE study. Only changes from baseline physical examination findings that meet the definition of an AE will be recorded on the AE page of the eCRF and will be summarized with other AE outcomes.

### 5.4.7 Vital Signs

Actual values and changes from baseline of both parent study and OLE study in vital signs (heart rate, systolic blood pressure, diastolic blood pressure, weight, height [baseline only], and BMI) will be summarized using descriptive statistics by previous treatment group in parent study, overall and post-baseline time point.

Vital signs data will be listed for each patient, with increases from baseline of >15 mmHg in systolic or diastolic blood pressure flagged.

## 6 DMC Analyses

Refer to DMC charter.

#### 7 Reference

- 1. Sharrett AR, Ballantyne CM, Coady SA, Heiss G, Sorlie PD, Catellier D, et al. Atherosclerosis Risk in Communities Study Group. Coronary Heart Disease Prediction from Lipoprotein Cholesterol Levels, Triglycerides, Lipoprotein(A), Apolipoproteins A-I and B, and HDL Density Subfractions. The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2001;104:1108-13.
- 2. World Health Organization (WHO) Fact Sheet No 317 Updated January 2015.
- 3. Robinson JG. Management of Familial Hypercholesterolemia: A Review of the recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Managed Care Pharm. 2013;19(2):139-49.


- 4. Pharmacokinetics in Patients with Impaired Renal Function Study Design, Data Analysis, and Impact on Dosing and Labeling. FDA Draft Guidance. March 2010
- 5. Haase A, Goldberg AC. Identification of people with heterozygous familial hypercholesterolemia. Curr Opin Lipidol. 2012;23:282-9.
- 6. Glynn RJ, Laird NM, and Rubin DB. (1986). Selection modelling versus mixture modelling with nonignorable nonresponse. In H. Wainer (ed.), Drawing Inferences from Self-Selected Samples, pp. 115–142. New York: Springer.


## 8 Appendices

## 8.1 Appendix 1: Schedule of Events (Subject Visit Schedule)

| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOT1 | 19/EOS <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|
| Week | EOS | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 | Wk 82 |
| | Parent | | | | | | | |
| Visit Window | 30 Days | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days | +14 days |
| | pre-M0 | | | | | | | |
| In-clinic Visit | X | X | | | X | | X | X |
| Phone Visit | | | X | X | | X | | |
| Procedure | | | | | | | | |
| Informed Consent | X | | | | | | | |
| Enrollment Criteria | X | | | | | | | |
| Medical History | X | | | | | | | |
| Concomitant | X | X | X | X | X | X | X | X |
| Medications | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X |
| Recording | | | | | | | | |
| Physical Exam | X | | | | X | | X | |
| Weight <sup>3</sup> | X | X | | | X | | X | X |
| Vital Signs <sup>4</sup> | X | X | | | X | | X | X |
| Urine Pregnancy | X | | | | | | | |
| Test <sup>5</sup> | | | | | | | | |
| Clinical Safety Labs <sup>6</sup> | X | X | | | X | | X | X |
| Basic Fasting Lipids <sup>7</sup> | X | X | | | X | | X | X |
| Coagulation <sup>8</sup> | X | | | | | | | |
| ApoB and hsCRP | X | X | | | X | | X | X |
| HbA <sub>1C</sub> | X | | | | X | | X | X |
| IWRS Contact <sup>9</sup> | X | X | | | X | | X | |
| Drug Dispensing | X | X | | | X | | | |
| Drug Return/ | | X | | | X | | X | |
| Compliance | | | | | | | 1.6 6.4 | |

NOTE: For patients who withdraw from study drug treatment, but consent to be followed for safety assessments and return to clinic for these visit, the visits will occur according to the protocol schedule. Safety assessments should include clinical safety and basic lipid laboratories, adverse events (AEs), physical examination (PE), and vital signs. For patients who withdraw from study drug treatment, but consent to be followed for safety assessments by phone, the telephone contacts will occur according the protocol schedule with information regarding current health status and to collect information on AEs (eg, recent procedures, hospitalizations, and if the patient has died, the cause of death). If a patient does not provide consent to be followed for safety assessments per the protocol (either by returning to clinic or by phone), Visit Week 78/End of Treatment (EOT) will be scheduled as soon as possible and the patient will be asked to come back 4 weeks after last investigational medicinal product (IMP) dose for Visit Week 82/End of Study (EOS). No further visits will be scheduled.


<sup>&</sup>lt;sup>1</sup> All procedures will be completed for all patients at either EOT or early withdrawal.

<sup>&</sup>lt;sup>2</sup> All procedures will be completed for all patients 4 weeks after last IMP dose if completing the study or early withdrawal.

<sup>&</sup>lt;sup>3</sup> Body weight will be measured in the morning while fasting, using consistent scales, after voiding, and without shoes and outerwear (eg, coats).

- <sup>4</sup> Vital signs will include diastolic blood pressure (DBP), systolic blood pressure (SBP), heart rate (HR) and will be collected prior to any blood sample collection. Patient will rest for 5 minutes prior to assessments
- <sup>5</sup> Urine pregnancy test in women of childbearing potential only
- <sup>6</sup> Clinical safety labs include hematology, blood chemistry, and urinalysis at all visits. Please refer to laboratory manual for detailed schedule of tests.
- <sup>7</sup> Basic fasting lipids include total cholesterol (TC), calculated low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-HDL-C,), and triglycerides (TG).
- <sup>8</sup> Only in patients receiving anticoagulant therapy that in the investigator's judgment require monitoring at Month 0 and 3 to 5 days post-Month 0
- <sup>9</sup> Interactive web response system (IWRS) contact at either an early withdrawal or an EOS visit to register study discontinuation visit date

# 8.2 Appendix 2: Adverse Event of Special Interest (AESI)

| Adverse Event Terms per Protocol | Associated MedDRA Preferred Terms |
|---|---|
| Creatine kinase elevations | Blood creatine phosphokinase abnormal |
| Creatine kinase elevations | Blood creatine phosphokinase increased |
| Creatine kinase elevations | Blood creatine phosphokinase MM abnormal |
| Creatine kinase elevations | Blood creatine phosphokinase MM increased |
| New onset or worsening diabetes mellitus | Blood glucose abnormal |
| New onset or worsening diabetes mellitus | Blood glucose increased |
| New onset or worsening diabetes mellitus | Diabetes mellitus |
| New onset or worsening diabetes mellitus | Diabetes mellitus inadequate control |
| New onset or worsening diabetes mellitus | Diabetic ketoacidosis |
| New onset or worsening diabetes mellitus | Glucose tolerance impaired |
| New onset or worsening diabetes mellitus | Glucose urine present |
| New onset or worsening diabetes mellitus | Glycosuria |
| New onset or worsening diabetes mellitus | Glycosylated haemoglobin increased |
| New onset or worsening diabetes mellitus | Hyperglycaemia |
| New onset or worsening diabetes mellitus | Impaired fasting glucose |
| New onset or worsening diabetes mellitus | Ketoacidosis |
| New onset or worsening diabetes mellitus | Ketosuria |
| New onset or worsening diabetes mellitus | Ketosis |
| New onset or worsening diabetes mellitus | Type 2 diabetes mellitus |
| New onset or worsening diabetes mellitus | Urine ketone body present |
| Hepatic disorders | Alanine aminotransferase abnormal |
| Hepatic disorders | Alanine aminotransferase increased |
| Hepatic disorders | Aspartate aminotransferase abnormal |
| Hepatic disorders | Aspartate aminotransferase increased |
| Hepatic disorders | Blood bilirubin abnormal |
| Hepatic disorders | Blood bilirubin increased |
| Hepatic disorders | Hepatic enzyme abnormal |
| Hepatic disorders | Hepatic enzyme increased |
| Hepatic disorders | Hypertransaminaseaemia |
| Hepatic disorders | Liver function test abnormal |
| Hepatic disorders | Liver function test increased |
| Hepatic disorders | Transaminases abnormal |
| Hepatic disorders | Transaminases increased |
| Hypoglycemia | Blood glucose abnormal |
| Hypoglycemia | Blood glucose decreased |
| Hypoglycemia | Hypoglycaemia |
| Hypoglycemia | Hypoglycaemic coma |
| Hypoglycemia | Hypoglycaemic encephalopathy |
| Hypoglycemia | Hypoglycaemic seizure |
| Hypoglycemia | Shock hypoglycaemic |
| Metabolic acidosis | Metabolic acidosis |
| Muscular disorders | Muscular weakness |
| Muscular disorders | Muscle necrosis |


| Muscular disorders | Muscle spasms |
|---|---|
| Muscular disorders | Myalgia |
| Muscular disorders | Myoglobin blood increased |
| Muscular disorders | Myoglobin blood present |
| Muscular disorders | Myoglobin urine present |
| Muscular disorders | Myoglobinaemia |
| Muscular disorders | Myoglininuria |
| Muscular disorders | Myopathy |
| Muscular disorders | Myopathy toxic |
| Muscular disorders | Necrotizing myositis |
| Muscular disorders | Pain in extremity |
| Muscular disorders | Rhabdomyolysis |
| Neurocognitive/Neurologic disorders | Amnesia |
| Neurocognitive/Neurologic disorders | Cognitive disorder |
| Neurocognitive/Neurologic disorders | Confusional state |
| Neurocognitive/Neurologic disorders | Disorientation |
| Neurocognitive/Neurologic disorders | Memory impairment |
| Neurocognitive/Neurologic disorders | Mental status changes |
| Renal disorders | Acute kidney injury |
| Renal disorders | Acute prerenal failure |
| Renal disorders | Blood creatinine abnormal |
| Renal disorders | Blood creatinine increased |
| Renal disorders | Blood urea abnormal |
| Renal disorders | Blood urea increased |
| Renal disorders | Blood urea nitrogen/Creatinine ratio increased |
| Renal disorders | Creatinine renal clearance abnormal |
| Renal disorders | Creatinine renal clearance decreased |
| Renal disorders | Glomerular filtration rate abnormal |
| Renal disorders | Glomerular filtration rate decreased |
| Renal disorders | Gout |
| Renal disorders | Oliguria |
| Renal disorders | Prerenal failure |
| Renal disorders | Renal failure |
| Renal disorders | Renal function test abnormal |
| Renal disorders | Renal impairment |


DocUUID : 56c02f8e-9400-4951-9733-c0dc2889592d

### Statistical Analysis Plan

Title: A MULTICENTER OPEN-LABEL EXTENSION (OLE) STUDY

TO ASSESS THE LONG-TERM SAFETY AND EFFICACY OF

BEMPEDOIC ACID (ETC-1002) 180 MG

**Protocol:** ETC-1002-050

Clinical Phase: 3

**Product:** ETC-1002

**Version (Date):** Statistical Analysis Plan – Version 1.2

**Status:** Final

Prepared by:

06 Dec 2018 01:14:051+0000

REASON: I approve this document f1330a26-8e65-4f1e-b28b-172f4186890d



17064876-dedd-4660-9752-8d3bc4287a9e



REASON: I approve this document 086860ea-c4a5-4e1a-a755-f8a0a04d5e64

Esperion Therapeutics

07 Dec 2018 15:53:016+0000

REASON: I approve this document fdfe4eec-c142-42c7-bf98-459047a30340

**Esperion Therapeutics** 


Date

## **Table of Contents**

| 1 | List of Abb | oreviations | . 4 |
|---|--------------|-------------------------------------------|-----|
| 2 | Introduction | on | . 7 |
| 3 | | ectives and Endpoints | |
| | | ives | |
| | | y Endpoint | |
| | | dary Endpoints | |
| | | dverse Events | |
| | | linical Safety Laboratories | |
| | | ital Signs. | |
| | | E | |
| | _ | acokinetic (PK) and Other Biomarkers | |
| 4 | | ign | |
| | • | Design | |
| | | Treatments and Assessments | |
| | | mization and Blinding | |
| | | e Size Justification | |
| | - | n Analyses, Final Analyses and Unblinding | |
| | | e from Planned Analyses | |
| 5 | | and Analytical Plans | |
| | | al Statistical Considerations | |
| | | ical Analysis Plans | |
| | | nalysis Sets | |
| | 5.2.1.1 | | |
| | 5.2.1.2 | | |
| | 5.2.2 Pr | otocol Violations and Deviations | |
| | 5.2.3 Su | abject Disposition | 13 |
| | | emographic and Baseline Characteristics | |
| | | ıbgroup Variables | |
| | | ledical History | |
| | 5.2.7 Co | oncomitant Medications | 15 |
| | 5.2.8 St | udy Drug Exposure and Compliance | 15 |
| | 5.3 Efficac | cy Endpoints and Analyses. | 15 |
| | 5.4 Safety | Data Endpoints and Analyses | 16 |
| | | dverse Events (AEs) | |
| | | dverse Events of Special Interest | |
| | | linical Cardiovascular Endpoints | |
| | | eurocognitive Events | |
| | | aboratory Evaluations | |
| | 5.4.5.1 | Hepatic Safety | |
| | 5.4.5.2 | Musculoskeletal Safety | |
| | 5.4.5.3 | Diabetes and Glycemia | |

Confidential

| | 5.4 | .5.4 Renal Safety | 22 |
|---|-----|---------------------------------------------------------|----|
| | | Physical Examinations (PEs) | |
| | | Vital Signs | |
| 6 | | Analyses | |
| | | ence | |
| | | ndices | |
| | | appendix 1: Schedule of Events (Subject Visit Schedule) | |
| | | ppendix 2: Adverse Event of Special Interest (AESI) | |

# 1 List of Abbreviations

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|-----------------------------------------|
| ACL | Adenosine triphosphate-citrate lyase |
| ACS | Acyl-CoA synthetase |
| ADR | Adverse drug reaction |
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ALB | Albumin |
| ALK-P | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| ApoB | Apolipoprotein B |
| ASCVD | Atherosclerotic cardiovascular diseases |
| AST | Aspartate aminotransferase |
| ATP | Adenosine triphosphate |
| AUC | Area under the concentration-time curve |
| AUC <sub>0-24</sub> | Area under the curve during 24 hours |
| BMI | Body mass index |
| BP | Blood pressure |
| BUN | Blood urea nitrogen |
| Ca | Calcium |
| CAS | Completer Analysis Set |
| CEC | Clinical Event Committee |
| CFR | Code of Federal Regulations |
| CHD | Coronary heart disease |
| CI | Confidence interval |
| CK | Creatine kinase |
| Cl | Chloride |
| CNS | Central nervous system |
| CoA | Acetyl-coenzyme A |
| CO <sub>2</sub> | Carbon dioxide |
| CV | Cardiovascular |
| CYP | Cytochrome P450 |
| DBP | Diastolic blood pressure |
| DMC | Data Monitoring Committee |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| eGFR | Estimated glomerular filtration rate |


| Abbreviation or Specialist Term | Explanation |
|---|---|
| EMA | European Medicines Agency |
| EOS | End of Study |
| ETC-1002 | Bempedoic acid |
| EU | European Union |
| FDA | Food and Drug Administration |
| FPFV | First patient first visit |
| FSH | Follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GI | Gastrointestinal |
| HbA <sub>1C</sub> | Glycosylated hemoglobin, Type A <sub>1C</sub> |
| HBsAg | Hepatitis B surface antigen |
| Hct | Hematocrit |
| HCV | Hepatitis C virus |
| HDL-C | High-density lipoprotein cholesterol |
| HeFH | Heterozygous familial hypercholesterolemia |
| Hgb | Hemoglobin |
| HMG-CoA | 3-hydroxy-3-methylglutaryl-coenzyme A |
| hs-CRP | High-sensitivity C-reactive protein |
| IB | Investigator's Brochure |
| ICD | Informed Consent Document |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IMP | Investigational medicinal product |
| IND | Investigational New Drug Application |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| ITT | Intention-to-treat |
| IUD | Intrauterine device |
| IWRS | Interactive web response system |
| K | Potassium |
| LDH | Lactate dehydrogenase |
| LDL-C | Low-density lipoprotein cholesterol |
| LDLR | LDL receptor |
| LFT | Liver function test |
| LPLV | Last patient last visit |
| LS | Least square |
| MACE | Major adverse cardiac event |
| MCH | Mean corpuscular hemoglobin |


DocUUID: 37fdb6e0-13e6-4166-b11d-9b0fadb51359


| Abbreviation or Specialist Term | Explanation |
|---|---|
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean corpuscular volume |
| MDRD | Modification of diet in renal disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Myocardial infarction |
| MRI | Magnetic resonance imaging |
| Na | Sodium |
| NA | Not applicable |
| NLA | National Lipid Association |
| NOAEL | No-observed-adverse-effect level |
| non-HDL-C | Non-high-density lipoprotein cholesterol |
| OLE | Open-label extension (study) |
| Parent study | Study 1002-040 |
| PCSK9 | Proprotein convertase subtilisin/kexin type 9 |
| PE | Physical exam |
| PK | Pharmacokinetic(s) |
| PT | Prothrombin time |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SOC | System organ class |
| SP | Safety population |
| SUSARS | Suspected and unexpected serious adverse reactions |
| T2DM | Type 2 diabetes mellitus |
| TB | Total bilirubin |
| TC | Total cholesterol |
| TEAE | Treatment-emergent adverse event |
| TG | Triglycerides |
| TQT | Thorough QT/QTc |
| ULN | Upper limit of normal |
| US | United States |
| WBC | White blood cell |
| WHO | World Health Organization |


DocUUID: 37fdb6e0-13e6-4166-b11d-9b0fadb51359

#### 2 Introduction

The purpose of this document is to describe the statistical methods, data derivations and data summaries to be employed in ETC-1002-050. The preparation of this statistical analysis plan (SAP) has been based on International Conference on Harmonisation (ICH) E3 and E9 Guidelines and in reference to Protocol ETC-1002-050 (Protocol Amendment 2, 10 May 2017).

The SAP will supersede the protocol in the event of any differences between the two documents in the plans for data analysis, and the protocol will be amended if appropriate. The SAP will be included as an appendix in the clinical study report for this protocol.

## 3 Study Objectives and Endpoints

## 3.1 Objectives

- The primary objective for this study is to characterize the safety and tolerability of long-term administration of bempedoic acid (ETC-1002) 180 mg
- The secondary objective is to characterize the efficacy of long-term administration of bempedoic acid 180 mg/day as assessed by changes in low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-high-density lipoprotein cholesterol (non-HDL-C), apolipoprotein B (ApoB), total cholesterol (TC), triglycerides TG and high-sensitivity C-reactive protein (hs-CRP) in patients with hyperlipidemia

## 3.2 Primary Endpoint

• The primary endpoint for this study is patient incidence of AEs

## 3.3 Secondary Endpoints

- Percent change from baseline in LDL-C at Weeks 52 and 78
- Change from baseline in LDL-C at Weeks 52 and 78
- Percent change from baseline in non-HDL-C at Weeks 52 and 78
- Percent change from baseline in TC at Weeks 52 and 78
- Percent change from baseline in ApoB at Weeks 52 and 78
- Percent change from baseline in hs-CRP at Weeks 52 and 78
- Percent change from baseline in TG at Weeks 52 and 78


• Percent change from baseline in HDL-C at Weeks 52 and 78

#### 3.3.1 Adverse Events

The evaluation of AEs will include only incidence of treatment-emergent AEs (TEAEs), defined as AEs that begin or worsen on or after the date of first dose of study drug administration in OLE period and until 30 days after last dose of study drug. Clinical endpoints (details see section 4.2) will be collected and adjudicated by an independent Clinical Events Committee (CEC). Clinical endpoints will also be reported as SAEs. Adverse events of special interest (AESI) will further be examined (See Section 5.4.2 for more information).

### 3.3.2 Clinical Safety Laboratories

The evaluation of clinical safety laboratories, including blood hematology, chemistry, coagulation, and urinalysis, will be based on the observed values. Observed values, changes and percent change from baseline of both the parent study and OLE study will be summarized for all post-baseline study visits.

#### 3.3.3 Vital Signs

The evaluation of vital signs (including heart rate, systolic blood pressure, diastolic blood pressure, height, and weight will be based on the observed values. For vital signs, observed values, and changes from baseline of both the parent study and OLE study will be summarized for all post-baseline study visits.

#### 3.3.4 PE

Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant.'

## 3.4 Lipids

After enrollment, patients will return to clinic at week 12, 52, 78/EOT and 82/EOS. Clinical laboratory samples will be collected and analyzed for calculated LDL-C and lipid and cardiometabolic biomarkers including non-HDL-C, HDL-C, TC, ApoB, and TG at baseline and all clinic visits for evaluation of bempedoic acid effects on lipids and cardiometabolic parameters.

## 3.5 Pharmacokinetic (PK) and Other Biomarkers

NA.

## 4 Study Design

## 4.1 Study Design

This is a multicenter OLE study designed to assess the long-term safety and efficacy of bempedoic acid (ETC-1002) 180 mg. All patients will receive open-label bempedoic acid 180 mg for up to 1.5 years after rolling over from the parent study (Study 1002-040) followed by a follow-up period off study drug for 4 weeks. Investigators, site staff, patients, and the study team will be masked to study lipid levels until the Week 12 study visit, after which time lipid values will be made available.

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other ongoing studies of bempedoic acid. A blinded independent expert Clinical Events Committee (CEC) will adjudicate designated clinical endpoints across the program, including all major adverse cardiac events (MACE) and non-MACE endpoints defined as: cardiovascular (CV) death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction [MI] (MACE), nonfatal stroke (MACE), hospitalization for unstable angina (MACE), coronary revascularization (MACE), noncoronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE) using standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs as well as a clinical endpoint.

The study will be conducted at approximately 125 clinical sites in the United States, Canada, Germany, Netherlands, Poland, and United Kingdom. The study will end when the last randomized patient completes their last study visit (last patient last visit [LPLV] for last randomized patient). The estimated overall duration of the study (first patient first visit [FPFV] to LPLV) is approximately 2.5 years.

Parent Study
Patients on ETC-1002
or Placebo and
Background Therapy

1.5 Years

4 weeks
Washout

Figure 1. Study 1002-040 Study Design

### 4.2 Study Treatments and Assessments

Day 1 for this study should occur on the same day as the end of study visit for the parent study (1002-040). Patients who provide informed consent and sign the ICD will be eligible to enroll in the study.

The schedule of study events is provided in Appendix 1. However, a patient can be seen at any time for reasons of safety.


The investigational products were listed in Table 1 below:

**Table 1: Investigational Medicinal Products** 

| | Investigational Medicinal Product |
|---|---|
| Product Name: | Bempedoic acid |
| Dosage Form: | Film-coated tablets |
| Unit Dose: | 180 mg |
| Container/Closure <sup>a</sup> | 100-count bottle with screw on, child proof cap |
| Route of Administration: | Oral, daily with or without food |
| Physical Description: | |
| Manufacturer<br>(Fill/Finish): | |

Study drug should be taken once a day (once every 24 hours) at approximately the same time every day and may be taken with or without food. Patients will fast (no food or drink, other than water) for a minimum of 10 hours prior to collection of all laboratory samples.

Please see Pharmacy Manual for detailed storage requirements and instructions.

Patients who withdraw from investigational medicinal product (IMP) treatment will be asked to continue to be followed for safety using the protocol-specified visit schedule and procedures. For details of study assessments, see Appendix 1: Schedule of Events (Subject Visit Schedule).

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other any ongoing studies of ETC-1002. All clinical endpoints, including all major cardiac events (MACE) and non-MACE endpoints defined as: CV death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction (MI) (MACE), nonfatal stroke (MACE), hospitalization for unstable angina (MACE), coronary revascularization (MACE), non-coronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE), will be adjudicated by an independent blinded expert Clinical Events Committee (CEC), using


standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs.

### 4.3 Randomization and Blinding

- Randomization is not applicable for this OLE study.
- Laboratory results for lipid panel and hs-CRP will be masked to investigators, patients, and the study team until the Week 12 visit is completed. All site staff involved with this trial should refrain from obtaining lipid panels between date of last study medication (bempedoic acid or placebo) dose at end of parent study Week 52 (Visit T7) and Week 12 in this OLE trial.

## 4.4 Sample Size Justification

The number of patients entering this study will depend on the number of patients completing Study 1002-040 and their willingness to enroll.

## 4.5 Interim Analyses, Final Analyses and Unblinding

An interim analysis will be conducted in 2H, 2018 in order to provide safety assessment to support NDA submission. Another interim analysis for Day120 safety update will be approximately 120 days after the NDA cutoff. The endpoints and analyses are the same as the defined in final analysis if applicable.

The final analysis will be performed after the database is locked, and the database released.

## 4.6 Change from Planned Analyses

There is no change from planned analyses for this study.

## 5 Statistical and Analytical Plans

#### 5.1 General Statistical Considerations

The treatment groups will be displayed as previous treatment in parent study as well as overall treatment group in OLE study.

In general, all safety and efficacy data will be reported as observed. No imputation will be performed for missing data. Descriptive statistics (n, mean, standard deviation [SD] or Standard Error [SE], median, Q1, Q3, minimum, and maximum) will be calculated for continuous data. Minimum and maximum will be presented same number of decimal places as reported/collected, one additional decimal place for mean and median, and two additional decimal places for SD.


Categorical data will be summarized using n and percentage based on number of non-missing values. Percentage will be presented with one decimal place. The number of missing values will be presented as a separate category with no percentage, but only if 1 or more patients are missing data for the summary. Otherwise, all categories will be presented (even if no patients are counted in the category). Counts of zero in any category will be presented without percentage. Ninety-five percent (95%) confidence intervals (CIs) will be calculated for select continuous and categorical endpoint estimates. All patients will be summarized together as well as by their prior treatment group in the parent study.

Data will be presented on listings in order of patient/subject, assessment date and assessment (in order collected on CRF, unless specified otherwise). Dates will be presented in format DDMMMYYYY.

Relative day calculations will be [date of interest – relative date + (date of interest >= relative date)]. This calculation will result in dates prior to the relative date being presented as negative days, and those occurring on or after the relative date as Day 1 or later, i.e., there will be no Day 0.

Two sets of baseline are defined for any laboratory parameters and vital signs: baseline in parent study (1002-040) and baseline in OLE study (1002-050). The parent baseline values will be directly extracted from parent study database and baseline for the OLE study is defined as the last non-missing value on or prior to the date of first dose in the OLE. If last dose of study treatment is missing, then the date of last visit at which study assessments were obtained on CRF will be used in its place.

The visit schedules and window are shown below.

| Visit | Day 1/Week 0 | Week 12 | Week 24 | Week 36 | Week 52 | Week 64 | Week<br>78/EOT | Week<br>82/EOS |
|---|---|---|---|---|---|---|---|---|
| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOT | 19/EOS |
| Slotted Study<br>Week | EOS Parent | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 | Wk 82 |
| Target Study<br>Day | 1 | 84 | 168 | 252 | 364 | 448 | 546 | 574 |
| Analysis<br>Window | 1 | [2,126] | [127,210] | [211,308] | [309,406] | [407,497] | [498,562] | [563,∞] |
| Protocol<br>defined visit<br>Windows | [30 Days, Pre<br>M0] | 84±7 | 168±7 | 252±7 | 364±7 | 448±7 | 546±7 | 574±14 |


## 5.2 Statistical Analysis Plans

#### 5.2.1 Analysis Sets

#### 5.2.1.1 Safety Population (SP)

The Safety Population (SP) is defined as all enrolled patients who received at least 1 dose of bempedoic acid during the OLE period and will be used for demographics and baseline characteristics, treatment exposure, concomitant medications, and all safety summaries.

#### **5.2.1.2** Completer Analysis Set (CAS)

The completer analysis set is defined as patients who completed the full 78 weeks treatment as per end of treatment CRF page.

#### 5.2.2 Protocol Violations and Deviations

A full list of protocol violations and deviations will be compiled and reviewed by the clinical team to identify key versus non-key violations/deviations before final database lock. For violations at study entry, patients will be assessed against the inclusion and exclusion criteria of the protocol. For on-study deviations, compliance with the protocol will be examined with regard to prohibited therapies, and timing and availability of planned assessments. The final list of protocol deviation will be approved by the study team prior to interim analysis cut of or database lock and will be used to generate the PD deviation summary and listing.

#### 5.2.3 Subject Disposition

The number of patients enrolled, and included in each analysis population, along with IMP and study completion status, will be summarized by the treatment group in parent ETC-1002-040 study and overall. In addition, the number of patients who withdraw from the study and withdraw from study drug will be summarized by discontinuation reason.

#### 5.2.4 Demographic and Baseline Characteristics

Demographic collected from the parent study will be used for this study. Two sets of baseline values will be defined: baseline of parent study and OLE study. The parent study baseline will be taken directly from the parent study, and the OLE baseline is defined as last non-missing value prior to the first dose of IMP in the OLE study. The following demographic and both baseline characteristics will be summarized by previous treatment group in parent study, as well as overall, for safety population:

age group (18-40, 41-64, 65-74, and >=75), gender, race, ethnicity, region (North America, and EU), height (cm), weight (kg), body mass index (kg/m<sup>2</sup>) ( $< 25, 25 - < 30, \ge 30 \text{ kg/m}^2$ ), waist circumference, systolic and diastolic blood pressure, fasting lipid parameters (TC, LDL-C, HDL-C, non-HDL-C and TG), apoB, hs-CRP).


Cardiovascular risk factors from the parent study: ASCVD (Yes/No), HeFH (Yes/No), baseline statin intensity (derived) (low or moderate, high), eGFR category, tobacco history, alcohol history, history of diabetics, history of hypertension.

Data will be summarized using descriptive statistics for continuous variables and using counts and percentages for categorical variables by treatment group and overall.

The baseline estimated glomerular filtration rate (eGFR) categories are: normal: ≥90 mL/min/1.73m<sup>2</sup>; mild Renal Impairment: 60-89 mL/min/1.73m<sup>2</sup>; moderate Renal Impairment: 30-59 mL/min/1.73m<sup>2</sup>, and severe Renal Impairment (15-29 mL/min/1.73m<sup>2</sup>).

#### 5.2.5 Subgroup Variables

Subgroups defined by below variables will be evaluated for safety and the LDL-C efficacy endpoint.

- 1) Gender (male vs. female)
- 2) Age ( $< 65 \text{ yrs. vs.} \ge 65 \text{ yrs. and} < 75 \text{ yrs. vs.} \ge 75 \text{ yrs.}$ )
- 3) Baseline CVD risk category (HeFH (with/without ASCVD) vs. ASCVD only)
- 4) Baseline statin intensity (low vs. moderate vs. high)
- 5) Race (White vs. other)
- 6) Baseline LDL category (< 100 mg/dL vs. ≥100 mg/dL) (efficacy only)
- 7) History of diabetes (yes vs. no)
- 8) Body Mass Index (BMI) ( $< 25, 25 < 30, \ge 30 \text{ kg/m}^2$ )
- 9) Region (North America, EU)

In case the number of patients within a subgroup is too small, e.g. less than 5% of the overall population, the analyses may not be performed or the subgroup levels may be combined.

#### **5.2.6** Medical History

General medical history, cardiovascular history/risk factors, previous statin use and statin tolerance history will be summarized by previous treatment group in parent study, as well as overall in OLE study for safety population and presented in a by-patient listing. Where appropriate, terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 or later.

If a patient is entering the study beyond the 30 day rollover window, new medical history that occur between more than 30 days after the end of the parent study and treatment start in OLE study (exclusive) that period will be collected and presented in a by-patient listing.


#### **5.2.7** Concomitant Medications

Concomitant medications are defined as medications that were ongoing at the time of study drug initiation in this OLE study or new medications that started post study drug initiation and within 30 days following the date of the last dose of study drug.

Medications, including lipid modifying therapy (LMT) medications, will be coded using WHO Drug (March, 2017, or later if appropriate). The frequency of use of concomitant medications will be summarized by previous treatment group in parent study, as well as overall in OLE study, for the safety population according to Anatomical Therapeutic Chemical (ATC) class and preferred term. Concomitant medications will be listed for each patient. Concomitant LMT medications will be summarized by ATC class and medication name and listed separately in a similar fashion.

#### 5.2.8 Study Drug Exposure and Compliance

The length of exposure to study drug will be calculated as the number of days from the first dose of study drug to the last dose of study drug, regardless if the patient missed one or more doses of study drug. Length of exposure will be summarized by previous treatment group in parent study and overall in OLE study using descriptive statistics for the safety population.

The number and percentage of patients who were compliant with taking study drug will be summarized by previous treatment group in parent study and overall in OLE study and post-baseline time point for the safety population for the following categories 0 - <80%; >= 80%. Overall compliance will be calculated as: 100\* (Total Number of Tablets Dispensed – Total Number of Tablets Returned) / (Treatment Duration in Days).

The study drug administration and compliance data, including reasons for poor compliance, will be listed for each patient.

## 5.3 Efficacy Endpoints and Analyses

Given the primary objective of the study being long term safety, efficacy analyses will be using the safety population (SP). The efficacy data will be summarized by previous treatment group in parent study as well as an overall group.

For each efficacy parameter, descriptive summary statistics at each visit will be provided for the actual value, change from baseline and percent change from baseline for both conventional and International System of Units (SI). Two sets of summaries will be provided using the baseline from the parent study and from the OLE study. The visits to be included in the overtime summary are baseline of parent study (1002-040), baseline of OLE study, week 12, week 52, week 78, and Week 82. There will be no imputation for missing data, all summaries will use observed data. Ninety-five percent (95%) CI will be provided for the estimates at post-baseline visits.


In addition, efficacy parameters will also be summarized using the Completer Analysis Set (CAS).

For LDL-C, Same descriptive summary statistics at each visit will be provided within subgroups for the actual value, change from baseline and percent change from baseline.

Efficacy data (actual value, change and percent change from baseline) from all visits will be presented using descriptive statistics using both conventional and standard units.

Figures (mean+/-se or median/IQR) supporting the summary tables will be provided for each efficacy parameter. Efficacy data from all visits will be provided in listings as well.

## 5.4 Safety Data Endpoints and Analyses

The safety and tolerability of ETC-1002 will be assessed by examination of TEAEs, physical exams, vital signs, clinical laboratory values (serum chemistry, hematology, coagulation and urinalysis), and weight. SP will be used for all safety analyses.

Unless otherwise stated, descriptive summaries will be displayed by previous treatment group actually received in parent study and overall group.

#### 5.4.1 Adverse Events (AEs)

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 or later and will be categorized by system organ class (SOC) and preferred term (PT). Summary tables will focus on TEAEs; however, listings will include all AEs (with non-TEAEs flagged). An additional AE listing will be provided for AEs occurred during rollover period.

In summary tables, TEAEs will be counted as "Not Related" if relationship to study drug was recorded as 'Not Related' or "Unlikely". Events will be counted as "Related" if relationship to study drug was recorded as 'Possible', 'Probable', 'Definite' or if relationship to study drug is missing.

The severity of the AE will be characterized as mild, moderate, or severe, to the following definitions:

- Mild: Events are usually transient and do not interfere with the patient's daily activities
- Moderate: Events introduce a low level of inconvenience or concern to the patient and may interfere with daily activities
- Severe: Events interrupt the patient's usual daily activity, are incapacitating with inability to do usual activities, or significantly affect clinical status and warrant intervention and/or close follow-up


Overviews of TEAEs will include total number of TEAEs and patient incidence of TEAE, TE SAE, related TEAE, related TE SAE, withdrew due to TEAE, AE with fatal outcome. Individual TEAE summary will be presented by previous treatment group in parent study and overall containing the following counts and percentages for:

- patients with TEAEs
- patients with TEAE by PT
- patients with TEAEs by SOC, PT and maximum severity
- patients with treatment-related TEAEs
- patients with treatment-related TEAEs by PT
- patients with treatment-related TEAEs by SOC and PT
- patients with treatment-emergent serious adverse events (TE SAEs)
- patients with TE SAEs by PT
- patients with TE SAEs by SOC, PT and maximum severity
- patients with treatment-related TE SAEs
- patients with treatment-related TE SAEs by SOC and PT
- TEAEs leading to discontinuation of IMP
- Fatal AEs by SOC and PT

In addition, summary tables will be provided, by prior treatment group and overall, for the number and percent of patients experiencing:

- adjudicated major adverse cardiovascular events and mortality (MACE) by event type
- non-CV deaths (non-MACE),
- nonfatal myocardial infarction [MI] (MACE),
- nonfatal stroke (MACE),
- hospitalization for unstable angina (MACE),
- coronary revascularization (MACE),
- noncoronary arterial revascularization (non-MACE),
- hospitalization for heart failure (non-MACE) using standardized definitions.

The TEAE, related TEAE, TE SAE, and AESI summaries by SOC, PT and maximum severity will be provided for relevant subgroups described in 5.2.5 with the exception of baseline LDL category.

The AE overview summaries will count a patient at most once in each AE category (at the "highest/most extreme" designation of each category regardless of preferred term) and percentages will be based on the total number of patients in the safety population.

In addition to a comprehensive listing of all AEs (with non-TEAEs flagged), separate listings will be generated for SAEs, AEs resulting in withdrawal of study drug, and AEs with a fatal outcome, investigator reported major adverse cardiovascular events and mortality, and adjudicated major adverse cardiovascular events and mortality.


#### 5.4.2 Adverse Events of Special Interest

Adverse events of special interest (AESI) will be identified based on a pre-defined list of preferred terms provided by the sponsor (Appendix 2).

AESI will be presented in a listing and summarized by SOC, PT and previous treatment group in parent study and overall in OLE study. A separate table for treatment emergent AESI resulting in the discontinuation of study drug will be summarized by SOC, PT, and previous treatment group in the parent study and overall in OLE study.

In addition to adverse events, AESI is also being evaluated based on safety lab parameters. The details are provided in 5.4.5.

#### 5.4.3 Clinical Cardiovascular Endpoints

Clinical cardiovascular endpoints will be monitored and adjudicated by an independent blinded expert CEC for this study and other ongoing studies the ETC-1002 program. Adjudicated clinical endpoints that are treatment-emergent will be summarized by event type and previous treatment group in parent study and overall in OLE study. All events will be provided in a listing. Additional details regarding clinical endpoints and clinical endpoint definitions will be included in CEC charter.

#### **5.4.4** Neurocognitive Events

Neurocognitive events will be identified and evaluated by routine safety monitoring of PE findings and AEs. Summarization of neurocognitive events will occur using pre-specified MedDRA terms and will be performed by SOC, severity, and relationship to study drug by previous treatment group in parent study and overall in OLE study.

#### 5.4.5 Laboratory Evaluations

Two sets of baseline for safety parameters are defined, similar to that for the efficacy parameters, baseline from the parent study and the baseline from the OLE study.

Continuous laboratory parameters (serum chemistry, hematology, coagulation (only for those patients receiving anti-coagulation), urinalysis, urinalysis [microscopic]) listed in Table 4 will be summarized using descriptive statistics at each scheduled visit starting from the baseline of the parent study. The similar on-treatment and completer analysis set approach for efficacy analysis described in section 5.3 will be used for safety laboratory analysis. All analysis will use conventional unit and SI unit will be provided for selected parameters.

Fasting serum glucose and HbA1c will be summarized using descriptive statistics for the observed value and the change, percent change from baseline by history of diabetics. Missing values for any of the laboratory evaluations will not be imputed; that is, only observed case data will be used.


Categorical urinalysis data will be listed, but will not be summarized.

As part of the AESI evaluation, below safety lab abnormality will be summarized by treatment group. All post-baseline lab values during the on-treatment period are being considered. Further details are provided in Section 5.4.6.1 through 5.4.6.4.

- ALT or AST ( $> 3 \times ULN$  and  $> 5 \times ULN$ )
- TB (>  $2 \times ULN$ )
- Potential Hy's Law case: (ALT and/or AST  $> 3 \times$  ULN with concurrent TB  $> 2 \times$  ULN)
- CK (>  $5 \times ULN$ ) and (> $10 \times ULN$ )
- Fasting Serum Glucose (mg/dL) ( $\leq$  50, and  $\geq$  126) by history of diabetics
- HbA1C ( $\geq$  6.5%) by history of diabetics
- Creatinine (change from baseline for >1 mg/dL)
- eGFR (< 15 mL/min/1.73m<sup>2</sup>, 15 –29 mL/min/1.73m<sup>2</sup>)
- Hgb (g/dL) (decrease from baseline for  $\geq 2$  g/dL)
- Hgb (< 8 g/dL)

The number and percentage of patients with the following laboratory abnormalities will be summarized by the parent study baseline statin intensity, previous treatment group in the parent study, and overall in the OLE study:

- ALT or AST ( $> 3 \times ULN$  and  $> 5 \times ULN$ )
- TB (>  $2 \times ULN$ )
- Potential Hy's Law case: (ALT and/or AST  $> 3 \times$  ULN with concurrent TB  $> 2 \times$  ULN)
- CK (>  $5 \times ULN$ ) and (> $10 \times ULN$ )
- Creatinine (change from baseline for > 1 mg/dL)
- eGFR (< 15 mL/min/1.73m<sup>2</sup>, 15 –29 mL/min/1.73m<sup>2</sup>)
- Hgb (g/dL) (decrease from baseline for  $\geq 2$  g/dL)
- Hgb (< 8 g/dL)


**Table 2:** Clinical Laboratory Parameters (Safety)

| Clinical Laboratory Test | Clinical Laboratory Test |
|---|---|
| <ul><li>Hematology</li><li>Hematocrit (Hct)</li></ul> | Blood Chemistry (serum, fasting) • Albumin (Alb) |
| <ul> <li>Hemoglobin (Hgb)</li> <li>Mean corpuscular hemoglobin (MCH)</li> <li>Mean corpuscular hemoglobin concentration (MCHC)</li> <li>Mean corpuscular volume (MCV)</li> </ul> | <ul> <li>Albumin (Alb)</li> <li>Alkaline phosphatase (ALK-P)</li> <li>Alanine aminotransferase (ALT; SGPT)</li> <li>Aspartate aminotransferase (AST; SGOT)</li> <li>Blood urea nitrogen (BUN)</li> </ul> |
| <ul> <li>Platelet count</li> <li>Red blood (RBC) cell count</li> <li>White blood (WBC) cell count with differential (absolute and %)</li> </ul> | <ul> <li>Calcium (Ca)</li> <li>Carbon dioxide (CO2)</li> <li>Chloride (Cl)</li> <li>Creatinine</li> </ul> |
| Urinalysis (Dipstick) Clarity Bilirubin Color Glucose Ketones Leukocyte esterase Nitrate Occult blood pH Protein Specific gravity Urobilinogen | <ul> <li>Creatine kinase (CK)</li> <li>Glucose</li> <li>Lactate dehydrogenase (LDH)</li> <li>Phosphorus</li> <li>Potassium (K)</li> <li>Sodium (Na)</li> <li>Total and direct bilirubin (TB)a</li> <li>Total protein</li> <li>Uric acid</li> <li>Coagulation—only in patients receiving anticoagulant therapy that in the investigator's judgment require monitoring at Month 0 and 3 to 5 days post-Month 0</li> <li>Prothrombin time (PT)</li> </ul> |
| Urinalysis (Microscopic)-only if urine dipstick abnormal Bacteria Casts Crystals Epithelial cells RBC WBC | International normalized ration (INR) Other Labs: • Urine pregnancy test • Hemoglobin A <sub>IC</sub> (HbA <sub>IC</sub> ) |

 $<sup>^{\</sup>rm a}$  If TB  ${\ge}1.2\times$  ULN, a reflex indirect (unconjugated) bilirubin will be obtained.


The number and percentage of patients with laboratory abnormalities (i.e., laboratory values outside the stated laboratory normal range) will be summarized at each time point (i.e., including baseline and post-baseline time points) for each laboratory parameter. The determination of laboratory abnormalities will take into account any unscheduled laboratory assessments. Additional lab-related summaries will be provided as follows for hepatic safety, musculoskeletal safety, diabetes and glycemia, and renal safety.

#### **5.4.5.1 Hepatic Safety**

For liver-associated enzymes and total bilirubin (TB), the number and percent of patients with abnormal values for ALT ( $>3 \times ULN$ ,  $>5 \times ULN$ ), AST ( $>3 \times ULN$ ,  $>5 \times ULN$ ), and TB ( $>2 \times ULN$ ) will be summarized by overall, normal baseline ALT/AST/TB and abnormal baseline ALT/AST/TB.

Hy's law criteria (>  $3 \times \text{upper limit}$  of normal [ULN] for either ALT or AST, with accompanying TB >  $2 \times \text{ULN}$ ) will also be applied to the data; any potential Hy's law cases will be listed separately. In the case of patients with Gilbert's disease, TB will be fractionated and the determination of  $2 \times \text{ULN}$  will be based upon direct (conjugated) bilirubin.

The number and percentage of patients experiencing a single incident or confirmed and repeated incidence of abnormal liver function test values for ALT (>3 × ULN, >5 × ULN), AST (>3 × ULN, >5 x ULN), CK (>5 × ULN, >10 × ULN) and either ALT and/or AST (>3 × ULN, >5 × ULN) will be summarized by the previous treatment group in the parent study and overall in the OLE study. A single incident is defined as the patient experiencing only one abnormal incident of the liver function test value. Repeated and confirmed incidence is defined as the patient experiencing at least one of the following: the last onstudy liver function test value is abnormal, the last on-treatment liver function test value is abnormal liver function test value for the same test.

A separate listing for direct TB will be provided for those who have Gilbert's syndrome.

#### **5.4.5.2** Musculoskeletal Safety

CK levels will be summarized by the value and change from baseline in the value, by treatment group and visit as well as baseline eGFR category. In addition, the number and percent of patients with abnormal CK values (>5 X ULN, >10 × ULN) will be summarized. These summaries of patients with abnormal CK will be performed overall, normal baseline CK, and abnormal baseline CK.

#### 5.4.5.3 Diabetes and Glycemia

For fasting glucose and HbA1C (%), a shift table from baseline with the number and percent of patients will be categorized as below:

Fasting glucose: >= 126 mg/dL; 100-125 mg/dL, and < 100 mg/dL; HbA1C (%): >=6.5%; >5.5 to <=6.4% and <=5.5%.

110A1C (70). >-0.570, >5.5 to <-0.470 and <-5.570.


These tables will be summarized by history of Diabetes.

Descriptive summary for fasting serum glucose and HbA1C will be provided by history of diabetics, previous treatment group in parent study and overall at each scheduled visit.

#### 5.4.5.4 Renal Safety

Shift tables of eGFR category from baseline over the study, will be provided by previous treatment group in parent study and overall.

In addition, renal function abnormality will be identified as: (1) A creatinine change from baseline of > 1 mg/dL (2) eGFR value <30 mL/min/1.73m2. A shift table from baseline with the number and percent of patients using the two categories will be presented.

#### 5.4.6 Physical Examinations (PEs)

Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant'. Baseline is defined as the last value prior to the first dose of study medication in OLE study. Only changes from baseline physical examination findings that meet the definition of an AE will be recorded on the AE page of the eCRF and will be summarized with other AE outcomes.

#### 5.4.7 Vital Signs

Actual values and changes from baseline of both parent study and OLE study in vital signs (heart rate, systolic blood pressure, diastolic blood pressure, weight, height [baseline only], and BMI) will be summarized using descriptive statistics by previous treatment group in parent study, overall and post-baseline time point.

Vital signs data will be listed for each patient, with increases from baseline of >15 mmHg in systolic or diastolic blood pressure flagged.

# 6 DMC Analyses

Refer to DMC charter.

#### 7 Reference

1. Sharrett AR, Ballantyne CM, Coady SA, Heiss G, Sorlie PD, Catellier D, et al. Atherosclerosis Risk in Communities Study Group. Coronary Heart Disease


Prediction from Lipoprotein Cholesterol Levels, Triglycerides, Lipoprotein(A), Apolipoproteins A-I and B, and HDL Density Subfractions. The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2001;104:1108-13.

- 2. World Health Organization (WHO) Fact Sheet No 317 Updated January 2015.
- 3. Robinson JG. Management of Familial Hypercholesterolemia: A Review of the recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Managed Care Pharm. 2013;19(2):139-49.
- 4. Pharmacokinetics in Patients with Impaired Renal Function Study Design, Data Analysis, and Impact on Dosing and Labeling. FDA Draft Guidance. March 2010
- 5. Haase A, Goldberg AC. Identification of people with heterozygous familial hypercholesterolemia. Curr Opin Lipidol. 2012;23:282-9.
- 6. Glynn RJ, Laird NM, and Rubin DB. (1986). Selection modelling versus mixture modelling with nonignorable nonresponse. In H. Wainer (ed.), Drawing Inferences from Self-Selected Samples, pp. 115–142. New York: Springer.


# 8 Appendices

## 8.1 Appendix 1: Schedule of Events (Subject Visit Schedule)

| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOT <sup>1</sup> | 19/EOS <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|
| Week | EOS | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 | Wk 82 |
| | Parent | | | | | | | |
| Visit Window | 30 Days | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days | +14 days |
| | pre-M0 | | | | | | | |
| In-clinic Visit | X | X | | | X | | X | X |
| <b>Phone Visit</b> | | | X | X | | X | | |
| Procedure | | | | | | | | |
| Informed Consent | X | | | | | | | |
| Enrollment Criteria | X | | | | | | | |
| Medical History | X | | | | | | | |
| Concomitant | X | X | X | X | X | X | X | X |
| Medications | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X |
| Recording | | | | | | | | |
| Physical Exam | X | | | | X | | X | |
| Weight <sup>3</sup> | X | X | | | X | | X | X |
| Vital Signs <sup>4</sup> | X | X | | | X | | X | X |
| Urine Pregnancy Test <sup>5</sup> | X | | | | | | | |
| Clinical Safety Labs <sup>6</sup> | X | X | | | X | | X | X |
| Basic Fasting Lipids <sup>7</sup> | X | X | | | X | | X | X |
| Coagulation <sup>8</sup> | X | | | | | | | |
| ApoB and hsCRP | X | X | | | X | | X | X |
| HbA <sub>1C</sub> | X | | | | X | | X | X |
| IWRS Contact <sup>9</sup> | X | X | | _ | X | | X | |
| Drug Dispensing | X | X | | | X | | | |
| Drug Return/ | _ | X | | _ | X | | X | |
| Compliance | | | | | | | | |

NOTE: For patients who withdraw from study drug treatment, but consent to be followed for safety assessments and return to clinic for these visit, the visits will occur according to the protocol schedule. Safety assessments should include clinical safety and basic lipid laboratories, adverse events (AEs), physical examination (PE), and vital signs. For patients who withdraw from study drug treatment, but consent to be followed for safety assessments by phone, the telephone contacts will occur according the protocol schedule with information regarding current health status and to collect information on AEs (eg, recent procedures, hospitalizations, and if the patient has died, the cause of death). If a patient does not provide consent to be followed for safety assessments per the protocol (either by returning to clinic or by phone), Visit Week 78/End of Treatment (EOT) will be scheduled as soon as possible and the patient will be asked to come back 4 weeks after last investigational medicinal product (IMP) dose for Visit Week 82/End of Study (EOS). No further visits will be scheduled.


<sup>&</sup>lt;sup>1</sup> All procedures will be completed for all patients at either EOT or early withdrawal.

<sup>&</sup>lt;sup>2</sup> All procedures will be completed for all patients 4 weeks after last IMP dose if completing the study or early withdrawal.

<sup>&</sup>lt;sup>3</sup> Body weight will be measured in the morning while fasting, using consistent scales, after voiding, and without shoes and outerwear (eg, coats).

<sup>&</sup>lt;sup>4</sup> Vital signs will include diastolic blood pressure (DBP), systolic blood pressure (SBP), heart rate (HR) and will be collected prior to any blood sample collection. Patient will rest for 5 minutes prior to assessments


DocUUID: 37fdb6e0-13e6-4166-b11d-9b0fadb51359

<sup>&</sup>lt;sup>5</sup> Urine pregnancy test in women of childbearing potential only

<sup>&</sup>lt;sup>6</sup> Clinical safety labs include hematology, blood chemistry, and urinalysis at all visits. Please refer to laboratory manual for detailed schedule of tests.

<sup>&</sup>lt;sup>7</sup> Basic fasting lipids include total cholesterol (TC), calculated low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-HDL-C,), and triglycerides (TG).

<sup>&</sup>lt;sup>8</sup> Only in patients receiving anticoagulant therapy that in the investigator's judgment require monitoring at Month 0 and 3 to 5 days post-Month 0

<sup>&</sup>lt;sup>9</sup> Interactive web response system (IWRS) contact at either an early withdrawal or an EOS visit to register study discontinuation visit date

# 8.2 Appendix 2: Adverse Event of Special Interest (AESI)

| Adverse Event Terms per Protocol | Associated MedDRA Preferred Terms |
|---|---|
| Creatine kinase elevations | Blood creatine phosphokinase abnormal |
| Creatine kinase elevations | Blood creatine phosphokinase achiernal Blood creatine phosphokinase increased |
| Creatine kinase elevations Creatine kinase elevations | Blood creatine phosphokinase MM abnormal |
| Creatine kinase elevations Creatine kinase elevations | Blood creatine phosphokinase MM increased |
| New onset or worsening diabetes mellitus | Blood glucose abnormal |
| | <u> </u> |
| New onset or worsening diabetes mellitus | Blood glucose increased Diabetes mellitus |
| New onset or worsening diabetes mellitus | |
| New onset or worsening diabetes mellitus | Diabetes mellitus inadequate control |
| New onset or worsening diabetes mellitus | Diabetic ketoacidosis |
| New onset or worsening diabetes mellitus | Glucose tolerance impaired |
| New onset or worsening diabetes mellitus | Glucose urine present |
| New onset or worsening diabetes mellitus | Glycosuria |
| New onset or worsening diabetes mellitus | Glycosylated haemoglobin increased |
| New onset or worsening diabetes mellitus | Hyperglycaemia |
| New onset or worsening diabetes mellitus | Impaired fasting glucose |
| New onset or worsening diabetes mellitus | Ketoacidosis |
| New onset or worsening diabetes mellitus | Ketosuria |
| New onset or worsening diabetes mellitus | Ketosis |
| New onset or worsening diabetes mellitus | Type 2 diabetes mellitus |
| New onset or worsening diabetes mellitus | Urine ketone body present |
| Hepatic disorders | Alanine aminotransferase abnormal |
| Hepatic disorders | Alanine aminotransferase increased |
| Hepatic disorders | Aspartate aminotransferase abnormal |
| Hepatic disorders | Aspartate aminotransferase increased |
| Hepatic disorders | Blood bilirubin abnormal |
| Hepatic disorders | Blood bilirubin increased |
| Hepatic disorders | Hepatic enzyme abnormal |
| Hepatic disorders | Hepatic enzyme increased |
| Hepatic disorders | Hypertransaminaseaemia |
| Hepatic disorders | Liver function test abnormal |
| Hepatic disorders | Liver function test increased |
| Hepatic disorders | Transaminases abnormal |
| Hepatic disorders | Transaminases increased |
| Hypoglycemia | Blood glucose abnormal |
| Hypoglycemia | Blood glucose decreased |
| Hypoglycemia | Hypoglycaemia |
| Hypoglycemia | Hypoglycaemic coma |
| Hypoglycemia Hypoglycemia | Hypoglycaemic encephalopathy |
| Hypoglycemia Hypoglycemia | Hypoglycaemic seizure |
| Hypoglycemia Hypoglycemia | Shock hypoglycaemic |
| Metabolic acidosis | Metabolic acidosis |
| Muscular disorders | Muscular weakness |
| | Muscle necrosis |
| Muscular disorders | iviuscie necrosis |


| Muscular disorders | Muscle spasms |
|---|---|
| Muscular disorders | Myalgia |
| Muscular disorders | Myoglobin blood increased |
| Muscular disorders | Myoglobin blood present |
| Muscular disorders | Myoglobin urine present |
| Muscular disorders | Myoglobinaemia |
| Muscular disorders | Myoglininuria |
| Muscular disorders | Myopathy |
| Muscular disorders | Myopathy toxic |
| Muscular disorders | Necrotizing myositis |
| Muscular disorders | Pain in extremity |
| Muscular disorders | Rhabdomyolysis |
| Neurocognitive/Neurologic disorders | Amnesia |
| Neurocognitive/Neurologic disorders | Cognitive disorder |
| Neurocognitive/Neurologic disorders | Confusional state |
| Neurocognitive/Neurologic disorders | Disorientation |
| Neurocognitive/Neurologic disorders | Memory impairment |
| Neurocognitive/Neurologic disorders | Mental status changes |
| Renal disorders | Acute kidney injury |
| Renal disorders | Acute prerenal failure |
| Renal disorders | Blood creatinine abnormal |
| Renal disorders | Blood creatinine increased |
| Renal disorders | Blood urea abnormal |
| Renal disorders | Blood urea increased |
| Renal disorders | Blood urea nitrogen/Creatinine ratio increased |
| Renal disorders | Creatinine renal clearance abnormal |
| Renal disorders | Creatinine renal clearance decreased |
| Renal disorders | Glomerular filtration rate abnormal |
| Renal disorders | Glomerular filtration rate decreased |
| Renal disorders | Gout |
| Renal disorders | Oliguria |
| Renal disorders | Prerenal failure |
| Renal disorders | Renal failure |
| Renal disorders | Renal function test abnormal |
| Renal disorders | Renal impairment |


DocUUID: 37fdb6e0-13e6-4166-b11d-9b0fadb51359

### Statistical Analysis Plan for Study 1002-050, 120 Day Safety Update Interim Analysis

Title: A MULTICENTER OPEN-LABEL EXTENSION (OLE) STUDY

TO ASSESS THE LONG-TERM SAFETY AND EFFICACY OF

BEMPEDOIC ACID (ETC-1002) 180 MG

**Protocol:** ETC-1002-050

Clinical Phase: 3

**Product:** ETC-1002 **Date:** 23-May-2019




#### Statistical Analysis Plan for Study 1002-050, Day 120 Safety Update Interim Analysis

An interim analysis for Day120 safety update will happen ≥ 4 months after the cutoff for the NDA submission (15-Mar-2019). The set of tables, listings and figures that were run for the NDA submission will be run again for the Day 120 safety update with additional tables and listings as described here. In addition, all of the subject incidence treatment-emergent adverse event (TEAE) tables as specified in the original SAP (dated as 05-Dec-2018), will be replaced with exposure-adjusted tables.

The lipid modifying treatment (LMT) use at the study baseline will be summarized by anatomic therapeutic chemical class and preferred term by treatment group in the parent study (1002-040) for the safety population.

The summary tables will be generated for incremental adverse events, serious adverse events, death, adverse events leading to discontinuation of investigational product and major adverse cardiac event by treatment group in the parent study (1002-040) for the safety population.

To calculate exposure-adjusted subject incidence, the number of subjects with at least one incidence of a given treatment-emergent adverse event (TEAE) will be used as the numerator, and the exposure-years for all the subjects for that treatment-emergent adverse event will be used as the denominator. The exposure-years will be calculated as total person time (in person-years) at risk from on or after the first dose of IMP and up to last date of IMP+30 days or end of study date or analysis cut-off date whichever is earlier for subjects who did not have a given TEAE. For a subject with the TEAE, the exposure-year will be calculated as total person time from on or after first dose of IMP to the onset date of first occurrence of the given TEAE. In the tables by maximum severity, the first occurrence to the maximum severity of the TEAE will be used for the exposure calculation.

The tables and listings for the Day 120 analyses:

| Number | Title | Population |
|---|---|---|
| | Patient Diaposition | The Enrolled |
| Table 14.1.1.1 | Patient Disposition | Patients |
| | Major Protocol Deviction | Safety |
| Table 14.1.1.2 | Major Protocol Deviation | Population |
| | Demographic and Baseline Characteristics from | Safety |
| Table 14.1.2.1 | the Parent ETC-1002-040 Study | Population |
| | Demographic and Baseline Characteristics from | Safety |
| Table 14.1.2.1.1 | OLE Study | Population |
| | Madicallictory | Safety |
| Table 14.1.3.1 | Medical History | Population |
| | Condinues sules History | Safety |
| Table 14.1.4.1 | Cardiovascular History | Population |
| | Concomitant Non-statin Medications by Anatomic | Safety |
| Table 14.1.6.1 | Therapeutic Chemical Class and Preferred Term | Population |
| | Concomitant Statin Medications by Anatomic | Safety |
| Table 14.1.6.2 | Therapeutic Chemical Class and Preferred Term | Population |
| | LMT Category at OLE Study (ETC-1002-050) | Cofoty |
| | Baseline by Anatomic Therapeutic Chemical Class | Safety |
| Table 14.1.6.3 | and Preferred Term | Population |
| | IMD Eveneure | Safety |
| Table 14.1.7 | IMP Exposure | Population |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline (Observed | Population |
| Table 14.2.1 | Data, Conventional Unit) | |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline by Gender | Population |
| Table 14.2.1.1 | (Observed Data, Conventional Unit) | |


| | Low-density Lipoprotein Cholesterol (LDL-C) | |
|---|---|---|
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline by Age | Population |
| Table 14.2.1.2 | (Observed Data, Conventional Unit) | |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline by | Population |
| | Baseline CVD Risk Category (Observed Data, | Гориналогі |
| Table 14.2.1.3 | Conventional Unit) | |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline by | Population |
| | Baseline Statin Intensity Category (Observed Data, | |
| Table 14.2.1.4 | Conventional Unit) | |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| T-1-1-44045 | Parent Study (ETC-1002-040) Baseline by Race | Population |
| Table 14.2.1.5 | (Observed Data, Conventional Unit) | |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline by | Population |
| Table 14.2.1.6 | Baseline LDL Category (Observed Data, Conventional Unit) | |
| Table 14.2.1.0 | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline by History | Population |
| Table 14.2.1.7 | of Diabetes (Observed Data, Conventional Unit) | . opaiation |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | |
| | Parent Study (ETC-1002-040) Baseline by | Safety |
| | Baseline BMI Group (Observed Data, Conventional | Population |
| Table 14.2.1.8 | Unit) | |


| | Low-density Lipoprotein Cholesterol (LDL-C) Values and Changes and Percent Changes from | Safety |
|---|---|---|
| | Parent Study (ETC-1002-040) Baseline by Region | Population |
| Table 14.2.1.9 | (Observed Data, Conventional Unit) | |
| | High-density Lipoprotein Cholesterol (HDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline (Observed | Population |
| Table 14.2.2 | Data, Conventional Unit) | |
| | Non-High-density Lipoprotein Cholesterol (Non - | |
| | HDL-C) Values and Changes and Percent | Safety |
| | Changes from Parent Study (ETC-1002-040) | Population |
| Table 14.2.3 | Baseline (Observed Data, Conventional Unit) | |
| | Total Cholesterol (TC) Values and Changes and | |
| | Percent Changes from Parent Study (ETC-1002- | Safety |
| Table 14.2.4 | 040) Baseline (Observed Data, Conventional Unit) | Population |
| | Triglycerides (TG) Values and Changes and | |
| | Percent Changes from Parent Study (ETC-1002- | Safety |
| Table 14.2.5 | 040) Baseline (Observed Data, Conventional Unit) | Population |
| | Apolipoprotein B (apo-B) Values and Changes and | 0-6-6- |
| | Percent Changes from Parent Study (ETC-1002- | Safety |
| Table 14.2.6 | 040) Baseline (Observed Data, Conventional Unit) | Population |
| | High-sensitivity C-reactive Protein (hs-CRP) Values | |
| | and Changes and Percent Changes from Parent | Safety |
| | Study (ETC-1002-040) Baseline (Observed Data, | Population |
| Table 14.2.7 | Conventional Unit) | |
| | Low-density Lipoprotein Cholesterol (LDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline (Standard | Population |
| Table 14.2.8.1 | Unit) | |
| | High-density Lipoprotein Cholesterol (HDL-C) | |
| | Values and Changes and Percent Changes from | Safety |
| | Parent Study (ETC-1002-040) Baseline (Standard | Population |
| Table 14.2.8.2 | Unit) | |

| Table 14.2.8.3 | Non-High-density Lipoprotein Cholesterol (Non-HDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |
|---|---|---|
| Table 14.2.8.4 | Total Cholesterol (TC) Values and Changes and Percent Changes from Parent Study (ETC-1002- 040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.2.8.5 | Triglycerides (TG) Values and Changes and Percent Changes from Parent Study (ETC-1002- 040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.2.8.6 | Apolipoprotein B (apo-B) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.2.8.7 | High-sensitivity C-reactive Protein (phCRP) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.2.9.1 | Low-density Lipoprotein Cholesterol (LDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Conventional Unit) | Completer<br>Analysis Set |
| Table 14.2.9.2 | High-density Lipoprotein Cholesterol (HDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Conventional Unit) | Completer<br>Analysis Set |
| Table 14.2.9.3 | Non-High-density Lipoprotein Cholesterol (Non-HDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline by Age (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.9.4 | Total Cholesterol (TC) Values and Changes and Percent Changes from Parent Study (ETC-1002- 040) Baseline (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.9.5 | Triglycerides (TG) Values and Changes and Percent Changes from Parent Study (ETC-1002- | Completer<br>Analysis Set |

| | 040) Baseline (Conventional Unit) | |
|---|---|---|
| Table 14.2.9.6 | Apolipoprotein B (apo-B) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Conventional Unit) | Completer<br>Analysis Set |
| Table 14.2.9.7 | High-sensitivity C-reactive Protein (phCRP) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Conventional Unit) | Completer<br>Analysis Set |
| Table 14.2.10.1 | Low-density Lipoprotein Cholesterol (LDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.10.2 | High-density Lipoprotein Cholesterol (HDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.10.3 | Non-High-density Lipoprotein Cholesterol (Non-HDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.10.4 | Total Cholesterol (TC) Values and Changes and<br>Percent Changes from Parent Study (ETC-1002-<br>040) Baseline (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.10.5 | Triglycerides (TG) Values and Changes and Percent Changes from Parent Study (ETC-1002- 040) Baseline (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.10.6 | Apolipoprotein B (apo-B) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Completer<br>Analysis Set |
| Table 14.2.10.7 | High-sensitivity C-reactive Protein (phCRP) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Completer<br>Analysis Set |


| Table 14.2.11.1 | Low-density Lipoprotein Cholesterol (LDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Observed Data, Conventional Unit) | Safety<br>Population |
|---|---|---|
| Table 14.2.11.2 | High-density Lipoprotein Cholesterol (HDL-C) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Conventional Unit) | Safety<br>Population |
| Table 14.2.11.3 | Non-High-density Lipoprotein Cholesterol (Non - HDL-C) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Conventional Unit) | Safety<br>Population |
| Table 14.2.11.4 | Total Cholesterol (TC) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Conventional Unit) | Safety<br>Population |
| Table 14.2.11.5 | Triglycerides (TG) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Conventional Unit) | Safety<br>Population |
| Table 14.2.11.6 | Apolipoprotein B (apo-B) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Conventional Unit) | Safety<br>Population |
| Table 14.2.11.7 | High-sensitivity C-reactive Protein (hs-CRP) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Conventional Unit) | Safety<br>Population |
| Table 14.2.12.1 | Low-density Lipoprotein Cholesterol (LDL-C) Values and Changes and Percent Changes from Parent Study (ETC-1002-040) Baseline (Observed Data, Standard Unit) | Safety<br>Population |
| Table 14.2.12.2 | High-density Lipoprotein Cholesterol (HDL-C) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Standard Unit) | Safety<br>Population |

| Table 14.2.12.3 | Non-High-density Lipoprotein Cholesterol (Non - HDL-C) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Standard Unit) | Safety<br>Population |
|---|---|---|
| Table 14.2.12.4 | Total Cholesterol (TC) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Standard Unit) | Safety<br>Population |
| Table 14.2.12.5 | Triglycerides (TG) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Standard Unit) | Safety<br>Population |
| Table 14.2.12.6 | Apolipoprotein B (apo-B) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Standard Unit) | Safety<br>Population |
| Table 14.2.12.7 | High-sensitivity C-reactive Protein (hs-CRP) Values and Changes and Percent Changes from Baseline (Baseline in OLE Study) (Observed Data, Standard Unit) | Safety<br>Population |
| Table 14.3.1.1.1 | Overview of Treatment-emergent Adverse Events | Safety<br>Population |
| Table 14.3.1.1.1.2 | Overview of Treatment-emergent Adverse Events by Gender | Safety<br>Population |
| Table 14.3.1.1.1.3 | Overview of Treatment-emergent Adverse Events by Age | Safety<br>Population |
| Table 14.3.1.1.1.4 | Overview of Treatment-emergent Adverse Events by Baseline CVD risk Category | Safety<br>Population |
| Table 14.3.1.1.5 | Overview of Treatment-emergent Adverse Events by Baseline Statin Intensity | Safety<br>Population |
| Table 14.3.1.1.1.6 | Overview of Treatment-emergent Adverse Events by Race | Safety Population |
| Table 14.3.1.1.7 | Overview of Treatment-emergent Adverse Events by History of Diabetes Overview of Treatment-emergent Adverse Events | Safety Population Safety |
| Table 14.3.1.1.1.8 | by Baseline BMI Group | Population |

| | Overview of Treatment-emergent Adverse Events | Safety |
|---|---|---|
| Table 14.3.1.1.1.9 | by Region | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.1 | Events (TE SAE) | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.2 | Events (TE SAE) by Gender | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.3 | Events (TE SAE) by Age | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.4 | Events (TE SAE) by Baseline CVD risk category | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.5 | Events (TE SAE) by Baseline Statin Intensity | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.6 | Events (TE SAE) by Race | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.7 | Events (TE SAE) by History of Diabetes | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.8 | Events (TE SAE) by Baseline BMI Group | Population |
| | Overview of Treatment-emergent Serious Adverse | Safety |
| Table 14.3.1.1.2.9 | Events (TE SAE) by Region | Population |
| | Overview of Treatment-emergent Adverse Events | Safety |
| Table 14.3.1.2.2 | Resulting in Withdrawal of Study Drug | Population |
| | Incremental Treatment-emergent Adverse Events | C-f-tr |
| Table | by System Organ Class, Preferred Term, and | Safety |
| 14.3.1.3.1.1a | Maximum Severity | Population |
| | Incremental Treatment-emergent Serious Adverse | Sofoty |
| Table | Events by System Organ Class, Preferred Term | Safety |
| 14.3.1.3.2.1a | and Maximum Severity | Population |
| | Incremental Treatment-emergent Adverse Events | |
| | Resulting in Discontinuation of IMP by System | Safety |
| Table | Organ Class, Preferred Term and Maximum | Population |
| 14.3.1.3.3.3a | Severity | |


DocUUID: 8adc0e63-e069-47db-8837-9177fe71f2a0

| Table<br>14.3.1.3.3.4a | Incremental Treatment-emergent Fatal Adverse Events by System Organ Class, Preferred Term, and Maximum Severity | Safety<br>Population |
|---|---|---|
| Table 14.3.2.2.1a | Incremental Treatment-emergent and Positively Adjudicated Adverse Cardiovascular Events by Event Type | Safety<br>Population |
| Table 14.3.2.2.2 | Exposure-Adjusted Subject Incidence of Treatment-emergent and Positivrely Adjudicated Adverse Cardiovascular Events by Event Type | Safety<br>Population |
| Table 14.3.3.1.1 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety<br>Population |
| Table 14.3.3.1.2 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population - by Gender |
| Table 14.3.3.1.3 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population - by Age |
| Table 14.3.3.1.4 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population – by Baseline CVD risk Category |
| Table 14.3.3.1.5 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population – by Baseline Statin Intensity |
| Table 14.3.3.1.6 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population – by Race |
| Table 14.3.3.1.7 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population – by History of |


| | | Diabetes |
|---|---|---|
| Table 14.3.3.1.8 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population – by Baseline Body Mass Index (BMI) Group |
| Table 14.3.3.1.9 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by System Organ Class,<br>Preferred Term and Maximum Severity | Safety Population – by Region |
| Table 14.3.3.2.1 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Safety<br>Population |
| Table 14.3.3.2.2 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Safety<br>Population - by<br>Gender |
| Table 14.3.3.2.3 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Safety<br>Population - by<br>Age |
| Table 14.3.3.2.4 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Safety Population – by Baseline CVD risk Category |
| Table 14.3.3.2.5 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Safety Population – by Baseline Statin Intensity |


DocUUID: 8adc0e63-e069-47db-8837-9177fe71f2a0


| Table 14.3.3.2.6 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Safety<br>Population –<br>by Race |
|---|---|---|
| | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum | Safety Population – by History of |
| Table 14.3.3.2.7 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Diabetes Safety Population – by Baseline Body Mass Index (BMI) |
| Table 14.3.3.2.8 Table 14.3.3.2.9 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by System<br>Organ Class, Preferred Term and Maximum<br>Severity | Group Safety Population – by Region |
| Table 14.3.3.3.3 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events Resulting in<br>Discontinuation of IMP by System Organ Class,<br>Preferred Term and Maximum Severity | Safety<br>Population |
| Table 14.3.3.4.1 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety<br>Population |
| Table 14.3.3.4.2 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety<br>Population - by<br>Gender |
| Table 14.3.3.4.3 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term | Safety<br>Population - by<br>Age |

| | and Maximum Severity | |
|---|---|---|
| Table 14.3.3.4.4 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety Population – by Baseline CVD risk Category |
| Table 14.3.3.4.5 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety Population – by Baseline Statin Intensity |
| Table 14.3.3.4.6 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety Population – by Race |
| Table 14.3.3.4.7 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety Population – by History of Diabetes |
| Table 14.3.3.4.8 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety Population – by Baseline Body Mass Index (BMI) Group |
| Table 14.3.3.4.9 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) by System Organ Class, Preferred Term<br>and Maximum Severity | Safety Population – by Region |
| Table 14.3.3.5.1 | Exposure-Adjusted Incidence of Related Treatment-emergent Adverse Events by System Organ Class and Preferred Term | Safety<br>Population |


| | Exposure-Adjusted Incidence of Related | Safety |
|---|---|---|
| | Treatment-emergent Adverse Events by System | Population - by |
| Table 14.3.3.5.2 | Organ Class and Preferred Term | Gender |
| | Exposure-Adjusted Incidence of Related | Safety |
| | Treatment-emergent Adverse Events by System | Population - by |
| Table 14.3.3.5.3 | Organ Class and Preferred Term | Age |
| | | Safety |
| | Exposure-Adjusted Incidence of Related | Population – |
| | Treatment-emergent Adverse Events by System | by Baseline |
| | Organ Class and Preferred Term | CVD risk |
| Table 14.3.3.5.4 | | Category |
| | | Safety |
| | Exposure-Adjusted Incidence of Related | Population – |
| | Treatment-emergent Adverse Events by System | by Baseline |
| Table 14.3.3.5.5 | Organ Class and Preferred Term | Statin Intensity |
| | Exposure-Adjusted Incidence of Related | Safety |
| | Treatment-emergent Adverse Events by System | Population – |
| Table 14.3.3.5.6 | Organ Class and Preferred Term | by Race |
| | Formation Adjusted Institutes of Deleted | Safety |
| | Exposure-Adjusted Incidence of Related | Population – |
| | Treatment-emergent Adverse Events by System | by History of |
| Table 14.3.3.5.7 | Organ Class and Preferred Term | Diabetes |
| | | Safety |
| | Experime Adjusted Incidence of Deleted | Population – |
| | Exposure-Adjusted Incidence of Related | by Baseline |
| | Treatment-emergent Adverse Events by System | Body Mass |
| | Organ Class and Preferred Term | Index (BMI) |
| Table 14.3.3.5.8 | | Group |
| | Exposure-Adjusted Incidence of Related | Safety |
| | Treatment-emergent Adverse Events by System | Population – |
| Table 14.3.3.5.9 | Organ Class and Preferred Term | by Region |
| | Exposure-Adjusted Incidence of Related | Safety |
| Table 14.3.3.6.2 | Treatment-emergent Adverse Events of Special | Population |

| | Interest (AESIs) by System Organ Class and Preferred Term | |
|---|---|---|
| Table 14.3.3.6.3 | Exposure-Adjusted Incidence of Related Treatment-emergent Serious Adverse Events by System Organ Class and Preferred Term | Safety<br>Population |
| Table 14.3.3.6.4 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events of Special Interest<br>(AESIs) Resulting in Discontinuation of IMP by<br>System Organ Class and Preferred Term | Safety<br>Population |
| Table 14.3.3.7.1 | Exposure-Adjusted Incidence of Treatment-<br>emergent Adverse Events by Preferred Term | Safety<br>Population |
| Table 14.3.3.7.2 | Exposure-Adjusted Incidence of Treatment-<br>emergent Serious Adverse Events by Preferred<br>Term | Safety<br>Population |
| Table 14.3.3.7.3 | Exposure-Adjusted Incidence of Related Treatment-emergent Adverse Events by Preferred Term | Safety<br>Population |
| Table 14.3.3.8.1 | Exposure-Adjusted Subject Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term | Safety<br>Population |
| Table 14.3.3.8.2 | Exposure-Adjusted Subject Incidence of Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term | Safety<br>Population |
| Table 14.3.3.8.3 | Exposure-Adjusted Subject Incidence of Fatal Treatment-emergent Adverse Events by System Organ Class and Preferred Term | Safety<br>Population |
| Table 14.3.4.1.1.1 | Serum Chemistry Laboratory Values and Changes from Baseline (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.1.1.2 | Hematology Laboratory Values and Changes from Baseline (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.1.1.3 | Coagulation Laboratory Values and Changes from Baseline (Conventional Unit) | Safety<br>Population |


DocUUID: 8adc0e63-e069-47db-8837-9177fe71f2a0

| | Urinalysis Laboratory Values and Changes from | Safety |
|---|---|---|
| Table 14.3.4.1.1.4 | Baseline (Conventional Unit) | Population |
| Table 14.3.4.1.1.5 | Alanine Aminotransferase (ALT), Aspartame Aminotransferase (AST) and Total Bilirubin Values and Changes from Baseline (Conventional Unit) | Safety<br>Population |
| | Creatinine Kinase Values and Changes from | Safety |
| Table 14.3.4.1.1.6 | Baseline (Conventional Unit) | Population |
| Table 14.3.4.1.1.7 | Creatinine Kinase Values and Changes from Baseline by Treatment and Baseline Estimated Glomerular Filtration Rate (eGFR) Category (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.1.1.8 | HbA1C and Fasting Glucose Laboratory Values and Changes from Baseline by History of Diabetics (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.1.2.1 | Serum Chemistry Laboratory Values and Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.3.4.1.2.2 | Hematology Laboratory Values and Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.3.4.1.2.3 | Coagulation Laboratory Values and Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.3.4.1.2.4 | Urinalysis Laboratory Values and Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |
| Table 14.3.4.1.2.5 | Alanine Aminotransferase (ALT), Aspartame Aminotransferase (AST) and Total Bilirubin Values and Changes from Baseline (Standard Unit) | Safety<br>Population |
| Table 14.3.4.1.2.6 | Creatinine Kinase Values and Changes from Parent Study (ETC-1002-040) Baseline (Standard Unit) | Safety<br>Population |


| Table 14.3.4.1.2.7 | Creatinine Kinase Values and Changes from Parent Study (ETC-1002-040) Baseline by Treatment and Baseline Estimated Glomerular Filtration Rate (eGFR) Category (Standard Unit) | Safety<br>Population |
|---|---|---|
| Table 14.3.4.1.2.8 | HbA1C and Fasting Glucose Laboratory Values and Changes from Parent Study (ETC-1002-040) Baseline by History of Diabetics (Standard Unit) | Safety<br>Population |
| Table 14.3.4.2.1 | Serum Chemistry Laboratory Abnormalities | Safety<br>Population |
| Table 14.3.4.2.2 | Hematology Laboratory Abnormalities | Safety<br>Population |
| Table 14.3.4.2.3 | Coagulation Laboratory Abnormalities | Safety Population - Patients Using Anticoagulatio n Medication |
| Table 14.3.4.2.4 | Urinalysis Laboratory Abnormalities | Safety<br>Population |
| Table 14.3.4.2.5 | Alanine Aminotransferase (ALT) Abnormalities (Overall, by Normal Baseline ALT and by Abnormal Baseline ALT) | Safety<br>Population |
| Table 14.3.4.2.6 | Aspartate Aminotransferase (AST) Abnormalities (Overall, by Normal Baseline AST and by Abnormal Baseline AST) | Safety<br>Population |
| Table 14.3.4.2.7 | Total Bilirubin (TB) Abnormalities (Overall, by Normal Baseline TB and by Abnormal Baseline TB) | Safety<br>Population |
| Table 14.3.4.2.8 | Creatinine Kinase Laboratory Abnormalities (Overall, by Normal Baseline CK and by Abnormal Baseline CK) | Safety<br>Population |
| Table 14.3.4.2.9.1 | Laboratory Abnormalities of Fasting Glucose by History of Diabetes Laboratory Abnormalities of HbA1C by History of | Safety Population Safety |
| Table 14.3.4.2.9.2 | Diabetes | Population |


| Table 14.3.4.2.10 | Laboratory Abnormalities of Renal Function | Safety<br>Population |
|---|---|---|
| Table 14.3.4.2.11 | Laboratory Parameters of Interest: Laboratory Abnormalities by Derived Baseline Statin Intensity of Parent Study (1002-040) | Safety<br>Population |
| Table 14.3.4.3.1.1 | Serum Chemistry Laboratory Values and Changes from Baseline (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.1.2 | Hematology Laboratory Values and Changes from Baseline (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.1.3 | Coagulation Laboratory Values and Changes from Baseline (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.1.4 | Urinalysis Laboratory Values and Changes from Baseline (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.1.5 | Alanine Aminotransferase (ALT), Aspartame Aminotransferase (AST) and Total Bilirubin Values and Changes from Baseline (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.1.6 | Creatinine Kinase Values and Changes from Baseline (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.1.7 | Creatinine Kinase Values and Changes from Baseline by Treatment and Baseline Estimated Glomerular Filtration Rate (eGFR) Category (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.1.8 | HbA1C and Fasting Glucose Laboratory Values and Changes from Baseline (Baseline in OLE Study) (Conventional Unit) | Safety<br>Population |
| Table 14.3.4.3.2.1 | Serum Chemistry Laboratory Values and Changes from Baseline (Baseline in OLE Study) (Standard | Safety<br>Population |

| | Unit) | |
|---|---|---|
| | Hematology Laboratory Values and Changes from | Safety |
| Table 14.3.4.3.2.2 | Baseline (Baseline in OLE Study) (Standard Unit) | Population |
| | Coagulation Laboratory Values and Changes from | Safety |
| Table 14.3.4.3.2.3 | Baseline (Baseline in OLE Study) (Standard Unit) | Population |
| | Urinalysis Laboratory Values and Changes from | Safety |
| Table 14.3.4.3.2.4 | Baseline (Baseline in OLE Study) (Standard Unit) | Population |
| | Alanine Aminotransferase (ALT), Aspartame | |
| | Aminotransferase (AST) and Total Bilirubin Values | Safety |
| | and Changes from Baseline (Baseline in OLE | Population |
| Table 14.3.4.3.2.5 | Study) (Standard Unit) | |
| | Creatinine Kinase Values and Changes from | Safety |
| Table 14.3.4.3.2.6 | Baseline (Baseline in OLE Study) (Standard Unit) | Population |
| | Creatinine Kinase Values and Changes from | |
| | Baseline by Treatment and Baseline Estimated | Safety |
| | Glomerular Filtration Rate (eGFR) Category | Population |
| Table 14.3.4.3.2.7 | (Baseline in OLE Study) (Standard Unit) | |
| | HbA1C and Fasting Glucose Laboratory Values | Safety |
| | and Changes from Baseline (Baseline in OLE | Population |
| Table 14.3.4.3.2.8 | Study) (Standard Unit) | Fopulation |
| | Estimated Glomerular Filtration Rate (eGFR) | Safety |
| | Values and Change from Parent Study (ETC-1002- | Population |
| Table 14.3.6.1.1 | 040) Baseline | 1 opulation |
| | Estimated Glomerular Filtration Rate (eGFR) | Safety |
| | Values and Change from Baseline (Baseline in | Population |
| Table 14.3.6.1.2 | OLE Study) | . opalation |
| | Shift Table of Estimated Glomerular Filtration Rate | Safety |
| | (eGFR) Category from Baseline of Parent Study | Population |
| Table 14.3.6.2.1 | (ETC-1002-040) over the Study | - |
| | Shift Table of Estimated Glomerular Filtration Rate | Safety |
| | (eGFR) Category from Baseline of OLE Study over | Population |
| Table 14.3.6.2.2 | the Study | . openation |


| | Shift Table of Urine Protein from Baseline of Parent | Safety |
|---|---|---|
| Table 14.3.6.3.1 | Study (ETC-1002-040) over the Study | Population |
| | Shift Table of Urine Protein from Baseline of OLE | Safety |
| Table 14.3.6.3.2 | Study over the Study | Population |
| | Post-Baseline of OLE Abnormal Liver Function | Safety |
| Table 14.3.6.4 | Summary | Population |
| | Vital Signs Values and Changes from Parent Study | Safety |
| Table 14.3.7 | (ETC-1002-040) Baseline | Population |
| | Vital Signs Values and Changes from OLE Study | Safety |
| Table 14.3.7.2 | (ETC-1002-050) Baseline | Population |
| | Detient Diemonitien | All Enrolled |
| Listing 16.2.1 | Patient Disposition | Patients |
| | Protocol Deviations | Safety |
| Listing 16.2.2 | Flotocol Deviations | Population |
| | Cardiovascular History and Cardiovascular Risk | Safety |
| Listing 16.2.3.2 | Factors | Population |
| | Medical History from Parent Study ETC-1002-040 | Safety |
| Listing 16.2.4.5 | Wedical History Holli Parent Study ETC-1002-040 | Population |
| | | Safety |
| | | Population |
| | | (Patients |
| | Now Medical History during Polloyer Period | Entered the |
| | New Medical History during Rollover Period | OLE Study |
| | | beyond 30-Day |
| | | Rollover |
| Listing 16.2.4.5.2 | | Window) |
| | Concomitant Non-statin Medications | Safety |
| Listing 16.2.4.6 | Concomitant Non-statin Medications | Population |
| | | Safety |
| Listing 16.2.4.7 | Concomitant Statin Medications | Population |
| | | Safety |
| Listing 16.2.5.1 | Exposure | Population |
| Listing 16.2.5.2 | IMP Administration | Safety |


| | | Population |
|---|---|---|
| Listing 16.2.6.1 | Lipids | FAS |
| | A diverse Trents | Safety |
| Listing 16.2.7.1 | Adverse Events | Population |
| | Adverse Events Occurred during Rollover Period | Safety |
| | (Between End of Parent Study and Treatment Start | |
| Listing 16.2.7.1.2 | of OLE Study) | Population |
| | Cariava Advaraa Evanta | Safety |
| Listing 16.2.7.2 | Serious Adverse Events | Population |
| | In any manufal Listing of Conjess Advance Frants | Safety |
| Listing 16.2.7.2.1 | Incremental Listing of Serious Adverse Events | Population |
| | A share a Farente De coltina e in Mith de cord of IMD | Safety |
| Listing 16.2.7.3 | Adverse Events Resulting in Withdrawal of IMP | Population |
| | Incremental Listing of Adverse Events Resulting in | Safety |
| Listing 16.2.7.3.1 | Withdrawal of Study Drug | Population |
| | Deleted Treetment annual Advance Frents | Safety |
| Listing 16.2.7.4 | Related Treatment-emergent Adverse Events | Population |
| | Dootho | Safety |
| Listing 16.2.7.5 | Deaths | Population |
| | In an area whell lieding of Doothe | Safety |
| Listing 16.2.7.5.1 | Incremental Listing of Deaths | Population |
| | A house 5 Secretarist On a sight heteroact | Safety |
| Listing 16.2.7.7 | Adverse Events of Special Interest | Population |
| | Adjudicated Major Adverse Cardiovascular Events | Safety |
| Listing 16.2.7.8 | and Mortality (MACE) and Non-MACE Events | Population |
| | Cotogorical Uringhaia Safety Laboratory | Safety |
| Listing 16.2.8.1.1 | Categorical Urinalysis Safety Laboratory | Population |
| | Chamistay Safaty Laborate | Safety |
| Listing 16.2.8.1.2 | Chemistry Safety Laboratory | Population |
| | Homotology Sofoty Laboratary | Safety |
| Listing 16.2.8.1.3 | Hematology Safety Laboratory | Population |
| | Consulation Cofety Laboratory | Safety |
| Listing 16.2.8.1.4 | Coagulation Safety Laboratory | Population |


| | | Cofoty |
|---|---|---|
| Listing 40 0 0 4 5 | Urinalysis Safety Laboratory | Safety |
| Listing 16.2.8.1.5 | | Population |
| | Safety Laboratory Abnormalities | Safety |
| Listing 16.2.8.1.6 | , , | Population |
| | Safety Laboratory Parameters of Interest | Safety |
| Listing 16.2.8.1.7 | carety Euperatory Furameters of Interest | Population |
| | Direct Bilirubin Values in Subjects with Gilbert's | Safety |
| Listing 16.2.8.1.8 | Disease | Population |
| | D T / | Safety |
| Listing 16.2.8.1.9.1 | Serum Pregnancy Test | Population |
| | | Safety |
| Listing 16.2.8.1.9.2 | Urine Pregnancy Test | Population |
| | | Safety |
| Listing 16.2.10 | Physical Examination | Population |
| | | Safety |
| Listing 16.2.11 | Vital Signs | Population |
| 2.04.19 | Mean (+/- SE) Low-density Lipoprotein Cholesterol | Safety |
| Figure 14.2.1 | (LDL-C) Values by Visit (Observed Data) | Population |
| riguic 14.2.1 | Mean (+/- SE) High-density Lipoprotein Cholesterol | Safety |
| Figure 14.2.2 | | |
| Figure 14.2.2 | (HDL-C) Values by Visit (Observed Data) | Population |
| | Mean (+/- SE) Non-High-density Lipoprotein | Safety |
| | Cholesterol (Non - HDL-C) Values by Visit | Population |
| Figure 14.2.3 | (Observed Data) | |
| | Mean (+/- SE) Total Cholesterol (TC) Values by | Safety |
| Figure 14.2.4 | Visit (Observed Data) | Population |
| | Median (IQR) Triglycerides (TG) Values by Visit | Safety |
| Figure 14.2.5.2 | (Observed Data) | Population |
| | Mean (+/- SE) Apolipoprotein B (apo-B) Values by | Safety |
| Figure 14.2.6 | Visit (Observed Data) | Population |
| | Median (IQR) High-sensitivity C-reactive Protein | Safety |
| Figure 14.2.7.2 | (hs-CRP) Values by Visit (Observed Data) | Population |


DocUUID: 8adc0e63-e069-47db-8837-9177fe71f2a0

### Statistical Analysis Plan

Title: A MULTICENTER OPEN-LABEL EXTENSION (OLE) STUDY

TO ASSESS THE LONG-TERM SAFETY AND EFFICACY OF

BEMPEDOIC ACID (ETC-1002) 180 MG

**Protocol:** ETC-1002-050

Clinical Phase: 3

**Product:** ETC-1002

**Version (Date):** Statistical Analysis Plan – Version 1.3

**Status:** Final

#### Prepared by:




## **Table of Contents**

| I | List of Abbreviations | . 4 |
|---|------------------------------------------------------|-----|
| 2 | Introduction | 6 |
| 3 | Study Objectives and Endpoints | . 6 |
| | 3.1 Objectives | . 6 |
| | 3.2 Endpoint | 6 |
| | Primary Endpoint (Safety) | . 6 |
| | Secondary Endpoints (Efficacy) | . 6 |
| | 3.2.1 Adverse Events | 7 |
| | 3.2.2 Clinical Safety Laboratories | 7 |
| | 3.2.3 Vital Signs | . 7 |
| | 3.2.4 Physical Exam | . 8 |
| | 3.2.5 Lipids | . 8 |
| 4 | Study Design | . 8 |
| | 4.1 Study Design | . 8 |
| | 4.2 Study Treatments and Assessments | . 9 |
| | 4.3 Randomization and Blinding | |
| | 4.4 Sample Size Justification | |
| | 4.5 Interim Analyses, Final Analyses, and Unblinding | |
| | 4.6 Change from Planned Analyses in Protocol | 11 |
| 5 | Statistical and Analytical Plans | |
| | 5.1 General Statistical Considerations | |
| | 5.2 Statistical Analysis Plans | |
| | 5.2.1 Analysis Sets | |
| | 5.2.1.1 Safety Population (SP) | |
| | 5.2.1.2 Completer Analysis Set (CAS) | 12 |
| | 5.2.2 Protocol Violations and Deviations | |
| | 5.2.3 Subject Disposition | |
| | 5.2.4 Demographic and Baseline Characteristics | |
| | 5.2.5 Subgroup Variables | |
| | 5.2.6 Medical History | |
| | 5.2.7 Concomitant Medications | |
| | 5.2.8 Study Drug Exposure and Compliance | |
| | 5.3 Efficacy Endpoints and Analyses | |
| | 5.4 Safety Data Endpoints and Analyses | |
| | 5.4.1 Adverse Events (AEs) | |
| | 5.4.2 Adverse Events of Special Interest | |
| | 5.4.2.1 Neurocognitive Events | |
| | 5.4.3 Clinical Cardiovascular Endpoints | |
| | 5.4.4 Laboratory Evaluations | |
| | 5.4.4.1 Hepatic Safety | |
| | 5.4.4.2 Musculoskeletal Safety | |
| | 5.4.4.3 Diabetes and Glycemia | 21 |

Confidential

| | 5.4 | .4.4 Renal Safety | 22 |
|---|------|--------------------------------------------------------|----|
| | | Physical Examination (PE) | |
| | | Vital Signs and Weight | |
| 6 | | Analyses | |
| | | ence | |
| 8 | Appe | ndices | 24 |
| | | ppendix 1: Schedule of Events (Subject Visit Schedule) | |
| | | ppendix 2: Adverse Event of Special Interest (AESI) | |

# 1 List of Abbreviations

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ALB | Albumin |
| ALK-P | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| ApoB | Apolipoprotein B |
| ASCVD | Atherosclerotic cardiovascular diseases |
| AST | Aspartate aminotransferase |
| BMI | Body mass index |
| BP | Blood pressure |
| BUN | Blood urea nitrogen |
| Ca | Calcium |
| CAS | Completer Analysis Set |
| CEC | Clinical Event Committee |
| CI | Confidence interval |
| CK | Creatine kinase |
| Cl | Chloride |
| CO <sub>2</sub> | Carbon dioxide |
| CV | Cardiovascular |
| DBP | Diastolic blood pressure |
| DMC | Data Monitoring Committee |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| eGFR | Estimated glomerular filtration rate |
| EOS | End of Study |
| ETC-1002 | Bempedoic acid |
| FDA | Food and Drug Administration |
| FPFV | First patient first visit |
| HbA <sub>1C</sub> | Glycosylated hemoglobin, Type A <sub>1C</sub> |
| Het | Hematocrit |
| HDL-C | High-density lipoprotein cholesterol |
| HeFH | Heterozygous familial hypercholesterolemia |
| Hgb | Hemoglobin |
| hs-CRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonisation |


| Abbreviation or Specialist Term | Explanation |
|---|---|
| IMP | Investigational medicinal product |
| ITT | Intention-to-treat |
| IWRS | Interactive web response system |
| K | Potassium |
| LDH | Lactate dehydrogenase |
| LDL-C | Low-density lipoprotein cholesterol |
| LMT | Lipid modifying therapy |
| LPLV | Last patient last visit |
| LS | Least square |
| MACE | Major adverse cardiac event |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Myocardial infarction |
| Na | Sodium |
| non-HDL-C | Non-high-density lipoprotein cholesterol |
| OLE | Open-label extension |
| Parent study | Study 1002-040 |
| PE | Physical exam |
| PT | Preferred term |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SI | International system of units |
| SOC | System organ class |
| SP | Safety population |
| TB | Total bilirubin |
| TC | Total cholesterol |
| TEAE | Treatment-emergent adverse event |
| TESAE | Treatment-emergent serious adverse event |
| TG | Triglycerides |
| ULN | Upper limit of normal |
| WBC | White blood cell |
| WHO | World Health Organization |


DocUUID : c537653e-4d89-483e-ac62-551eb4dabd51

#### 2 Introduction

The purpose of this document is to describe the statistical methods, data derivations and data summaries to be employed in ETC-1002-050. The preparation of this statistical analysis plan (SAP) has been based on International Conference on Harmonisation (ICH) E3 and E9 Guidelines and in reference to Protocol ETC-1002-050 (Protocol Amendment 2, 15Jan2018).

The SAP will supersede the protocol in the event of any differences between the two documents in the plans for data analysis, and the protocol will be amended if appropriate. The SAP will be included as an appendix in the clinical study report for this protocol.

## 3 Study Objectives and Endpoints

## 3.1 Objectives

- The primary objective for this study is to characterize the safety and tolerability of long-term administration of bempedoic acid (ETC-1002) 180 mg
- The secondary objective is to characterize the efficacy of long-term administration of bempedoic acid 180 mg/day as assessed by changes in low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-high-density lipoprotein cholesterol (non-HDL-C), apolipoprotein B (ApoB), total cholesterol (TC), triglycerides TG, and high-sensitivity C-reactive protein (hs-CRP) in patients with hyperlipidemia

# 3.2 Endpoint

## **Primary Endpoint (Safety)**

• The primary endpoint for this study is patient incidence of treatment-emergent adverse events (TEAEs)

## **Secondary Endpoints (Efficacy)**

- Percent change from baseline in LDL-C at Weeks 52 and 78
- Change from baseline in LDL-C at Weeks 52 and 78
- Percent change from baseline in non-HDL-C at Weeks 52 and 78
- Percent change from baseline in TC at Weeks 52 and 78
- Percent change from baseline in ApoB at Weeks 52 and 78


- Percent change from baseline in hs-CRP at Weeks 52 and 78
- Percent change from baseline in TG at Weeks 52 and 78
- Percent change from baseline in HDL-C at Weeks 52 and 78

## **Other Safety Endpoints**

- Laboratory Results
- Physical Measurements
- Vital Signs
- Hepatic Safety
- Musculoskeletal Safety
- Diabetes and Hyperglycemia
- Renal Safety
- Neurocognitive Events
- Clinical Endpoints

#### 3.2.1 Adverse Events

The evaluation of adverse events (AEs) will include only incidence of TEAEs, defined as AEs that begin or worsen on or after the date of first dose of study drug administration in open-label extension (OLE) period and until 30 days after last dose of study drug. AESI will be examined further (See Section 5.4.2 for more information).

Clinical endpoints (details see section 4.2) will be collected and adjudicated by an independent Clinical Events Committee (CEC). Clinical endpoints will also be reported as AEs.

## 3.2.2 Clinical Safety Laboratories

The evaluation of clinical safety laboratories, including blood hematology, chemistry, coagulation, and urinalysis will be based on the observed values. Observed values, change from baseline, and percent change from baseline of both the parent study and OLE study will be summarized for all the scheduled post-baseline visits.

#### 3.2.3 Vital Signs

The evaluation of vital signs (including heart rate, systolic blood pressure, and diastolic blood pressure, and weight and BMI) will be based on the observed values. The summary of the observed values and change from baseline will be performed for all the scheduled visits based on the baseline of the parent study and OLE study. Baseline height will be summarized and will be used in the BMI calculations over time.


## 3.2.4 Physical Exam

Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant.'

## **3.2.5** Lipids

After enrollment, patients will return to clinic at Weeks 12, 52, 78/EOT, and 82/EOS. Clinical laboratory samples will be collected and analyzed for calculated LDL-C and lipid and cardiometabolic biomarkers including non-HDL-C, HDL-C, TC, ApoB, and TG at baseline and all clinic visits for evaluation of bempedoic acid effects on lipids and cardiometabolic parameters.

# 4 Study Design

# 4.1 Study Design

This is a multicenter OLE study designed to assess the long-term safety and efficacy of bempedoic acid (ETC-1002) 180 mg. All patients will receive open-label bempedoic acid 180 mg for up to 1.5 years after rolling over from the parent study (Study 1002-040) followed by a follow-up period off study drug for 4 weeks. Investigators, site staff, patients, and the study team will be masked to study lipid levels until the Week 12 study visit, after which time lipid values will be made available.

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other ongoing studies of bempedoic acid. A blinded independent expert Clinical Events Committee (CEC) will adjudicate designated clinical endpoints across the program, including all major adverse cardiac events (MACE) and non-MACE endpoints defined as: cardiovascular (CV) death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction [MI] (MACE), nonfatal stroke (MACE), hospitalization for unstable angina (MACE), coronary revascularization (MACE), noncoronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE) using standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs as well as a clinical endpoint.

The study will be conducted at approximately 125 clinical sites in the United States, Canada, Germany, Netherlands, Poland, and United Kingdom. The study will end when the last randomized patient completes their last study visit (last patient last visit [LPLV] for last randomized patient). The estimated overall duration of the study (first patient first visit [FPFV] to LPLV) is approximately 2.5 years.

Figure 1. Study 1002-050 Study Design



# 4.2 Study Treatments and Assessments

Day 1 for this study should occur on the same day as the end of study visit for the parent study (1002-040). Patients who provide informed consent will be eligible to enroll in the study.

The schedule of study events is provided in Appendix 1. However, a patient can be seen at any time for reasons of safety.

The investigational products were listed in Table 1 below:

**Table 1: Investigational Medicinal Products** 

| | Investigational Medicinal Product |
|---|---|
| Product Name: | Bempedoic acid |
| Dosage Form: | Film-coated tablets |
| Unit Dose: | 180 mg |
| Container/Closure <sup>a</sup> | 100-count bottle with screw on, child proof cap |
| Route of Administration: | Oral, daily with or without food |
| Physical Description: | |
| Manufacturer<br>(Fill/Finish): | |

Study drug should be taken once a day (once every 24 hours) at approximately the same time every day and may be taken with or without food. Patients will fast (no food or drink, other than water) for a minimum of 10 hours prior to collection of all laboratory samples.

Please see Pharmacy Manual for detailed storage requirements and instructions.

Patients who withdraw from investigational medicinal product (IMP) treatment will be asked to continue to be followed for safety using the protocol-specified visit schedule and procedures. For details of study assessments, see Appendix 1: Schedule of Events (Subject Visit Schedule).

An independent expert Data Monitoring Committee (DMC) will formally review accumulating unblinded safety and efficacy data from this and other any ongoing studies of ETC-1002. All clinical endpoints, including all major cardiac events (MACE) and non-MACE endpoints defined as: CV death (MACE), non-CV death (non-MACE), nonfatal myocardial infarction (MI) (MACE), nonfatal stroke (MACE), hospitalization for unstable angina (MACE), coronary revascularization (MACE), non-coronary arterial revascularization (non-MACE), and hospitalization for heart failure (non-MACE), will be adjudicated by an independent blinded expert Clinical Events Committee (CEC), using standardized definitions. Any clinical endpoints that meet serious adverse event (SAE) criteria will be reported as SAEs.

# 4.3 Randomization and Blinding

Randomization is not applicable for this OLE study.

Laboratory results for lipid panel and hs-CRP will be masked to investigators, patients, and the study team until the Week 12 visit is completed. All site staff involved with this trial should refrain from obtaining lipid panels between date of last study medication (bempedoic acid or placebo) dose at end of parent study Week 52 (Visit T7) and Week 12 in this OLE trial.

4.4 Sample Size Justification

The number of patients entering this study will depend on the number of patients completing Study 1002-040 and their willingness to enroll.

# 4.5 Interim Analyses, Final Analyses, and Unblinding

An interim analysis will be conducted in 2H 2018 in order to provide safety assessment to support NDA submission. Another interim analysis for Day120 safety update will be approximately 120 days after the NDA cutoff. The endpoints and analyses are the same as those defined in final analysis if applicable.

The final analysis will be performed after the database is locked. Confidential


# 4.6 Change from Planned Analyses in Protocol

There is no change from planned analyses for this study.

# 5 Statistical and Analytical Plans

## 5.1 General Statistical Considerations

The treatment groups will be displayed as previous treatment in parent study as well as overall treatment group in OLE study.

In general, all safety and efficacy data will be reported as observed. No imputation will be performed for missing data. Descriptive statistics (n, mean, standard deviation, median, Q1, Q3, minimum, and maximum) will be calculated for continuous data. Minimum and maximum will be presented same number of decimal places as reported/collected, one additional decimal place for mean and median, and two additional decimal places for standard deviation. Ninety-five percent (95%) confidence intervals (CIs) will be calculated for select continuous endpoint estimates.

Categorical data will be summarized using n and percentage based on number of nonmissing values. Percentage will be presented with one decimal place. The number of missing values will be presented as a separate category with no percentage, but only if 1 or more patients are missing data for the summary. Otherwise, all categories will be presented (even if no patients are counted in the category). Counts of zero in any category will be presented without percentage.

Data will be presented on listings by prior treatment group in the parent study, subject ID, assessment (in order collected on CRF, unless specified otherwise), and assessment date. Dates will be presented in format DDMMMYYYY.

Relative day calculations will be [date of interest – relative date + (date of interest >= relative date)]. This calculation will result in dates prior to the relative date being presented as negative days, and those occurring on or after the relative date as Day 1 or later, i.e., there will be no Day 0.

Two sets of baseline are defined for applicable endpoints: baseline in parent study (1002-040) and baseline in OLE study (1002-050). The parent baseline values will be directly extracted from parent study database. The baseline for the OLE study is defined as the last non-missing value on or prior to the date of first dose in the OLE.

If last dose of study treatment is missing, then the end of study date or death date, whichever occurs earlier, will be used in its place.

The visit schedules and windows are shown below:

| | | | | | | | | Week | Week |
|---|---|---|---|---|---|---|---|---|---|
| V | isit | Day 1/Week 0 | Week 12 | Week 24 | Week 36 | Week 52 | Week 64 | 78/EOT | 82/EOS |


| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOT | 19/EOS |
|---|---|---|---|---|---|---|---|---|
| Slotted Study<br>Week | EOS Parent | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 | Wk 82 |
| Target Study<br>Day | 1 | 84 | 168 | 252 | 364 | 448 | 546 | 574 |
| Analysis<br>Window | 1 | [2,126] | [127,210] | [211,308] | [309,406] | [407,497] | [498,562] | [563,∞] |
| Protocol<br>defined visit<br>Windows | [30 Days, Pre<br>M0] | 84±7 | 168±7 | 252±7 | 364±7 | 448±7 | 546±7 | 574±14 |

## 5.2 Statistical Analysis Plans

## 5.2.1 Analysis Sets

## **5.2.1.1 Safety Population (SP)**

The SP is defined as all enrolled patients who received at least 1 dose of bempedoic acid during the OLE period and will be used for demographics and baseline characteristics, treatment exposure, concomitant medications, safety and efficacy summaries. If all subjects receive at least one dose of bempedoic acid in this study, the SP will be used for all efficacy analyses as well.

## 5.2.1.2 Completer Analysis Set (CAS)

The CAS is defined as the patients who completed the full 78 weeks treatment as per End of Treatment CRF page.

#### **5.2.2** Protocol Violations and Deviations

A full list of protocol violations and deviations will be compiled and reviewed by the clinical team to identify key versus non-key violations/deviations before final database lock. For violations at study entry, patients will be assessed against the inclusion and exclusion criteria of the protocol. For on-study deviations, compliance with the protocol will be examined with regard to prohibited therapies, and timing and availability of planned assessments. The final list of protocol deviation will be approved by the study team prior to interim analysis cut of or final database lock, and will be used to generate the protocol deviation summary and listing.

#### **5.2.3** Subject Disposition

The number of patients enrolled, and included in each analysis population, along with IMP and study completion status, will be summarized by the treatment group in parent ETC-1002-040 study and overall. In addition, the number of patients who withdraw from the study and withdraw from study drug will be summarized by discontinuation reason.


## **5.2.4** Demographic and Baseline Characteristics

Two sets of baseline values will be defined: baseline of parent study and OLE study. The parent study baseline will be taken directly from the parent study, and the OLE baseline is defined as last non-missing value prior to the first dose of IMP in the OLE study. The following demographic and both baseline characteristics will be summarized using descriptive statistics by previous treatment group in parent study, as well as overall, for safety population:

- Age group (18-40, 41-64, 65-74, and >=75 years), gender, race, ethnicity, region (North America, and Europe), height (cm), weight (kg), body mass index (BMI) (kg/m²) (< 25, 25 < 30, ≥ 30 kg/ m²), , systolic and diastolic blood pressure, fasting lipid parameters (TC, LDL-C, HDL-C, non-HDL-C, and TG), apoB, and hs-CRP.
- Cardiovascular risk factors from the parent study: ASCVD (Yes/No), HeFH (Yes/No), baseline statin intensity (derived) (low or moderate, high), eGFR category, tobacco history, alcohol history, history of diabetics, and history of hypertension.
- The baseline estimated glomerular filtration rate (eGFR) categories are: normal: ≥90 mL/min/1.73m²; mild Renal Impairment: 60-89 mL/min/1.73m²; moderate Renal Impairment: 30-59 mL/min/1.73m², and severe Renal Impairment (15-29 mL/min/1.73m²).

## 5.2.5 Subgroup Variables

Subgroups defined by below variables will be evaluated for safety and the LDL-C efficacy endpoint.

- 1) Gender (male vs. female)
- 2) Age (< 65 yrs. vs.  $\ge 65$  yrs. and < 75 yrs. vs.  $\ge 75$  yrs.)
- 3) Baseline CVD risk category (HeFH (with/without ASCVD) vs. ASCVD only)
- 4) Baseline statin intensity (low vs. moderate vs. high)
- 5) Race (White vs. other)
- 6) Baseline LDL category (< 100 mg/dL vs. ≥100 mg/dL) (efficacy only)
- 7) History of diabetes (yes vs. no)
- 8) Body Mass Index (BMI) ( $< 25, 25 < 30, \ge 30 \text{ kg/m}^2$ )
- 9) Region (North America, Europe)

In case the number of patients within a subgroup is too small, e.g. less than 5% of the overall population, the analyses may not be performed or the subgroup levels may be combined.


## **5.2.6** Medical History

General medical history, cardiovascular history/risk factors, previous statin use and statin tolerance history will be summarized by previous treatment group in parent study, as well as overall in OLE study for safety population and presented in a by-patient listing. Where appropriate, terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 or later.

If a patient is entering the study beyond the 30-day rollover window, new medical history that occur between more than 30 days after the end of the parent study and treatment start in OLE study (exclusive) that period will be collected and presented in a by-patient listing.

#### **5.2.7** Concomitant Medications

Concomitant medications are defined as medications that were ongoing at the time of study drug initiation in this OLE study or new medications that started post study drug initiation and within 30 days following the date of the last dose of study drug.

Medications, including lipid modifying therapy (LMT) medications, will be coded using WHO Drug (March, 2017, or later if appropriate). The frequency of use of concomitant medications will be summarized by previous treatment group in parent study, as well as overall in OLE study, for the safety population according to Anatomical Therapeutic Chemical (ATC) class and preferred term. Concomitant medications will be listed for each patient. Concomitant LMT medications will be summarized by ATC class and medication name and listed separately in a similar fashion.

#### 5.2.8 Study Drug Exposure and Compliance

For each patient, the length of exposure to study drug will be calculated as the number of days from the first dose of study drug to the last dose of study drug, regardless if the patient missed one or more doses of study drug. Length of exposure will be summarized by previous treatment group in parent study and overall in OLE study using descriptive statistics for the safety population.

For each patient, overall compliance (%) will be calculated as: (Total Number of Tablets Dispensed – Total Number of Tablets Returned)\*100/ (Treatment Duration in Days). The number and percentage of patients who were compliant with taking study drug will be summarized by previous treatment group in parent study and overall in OLE study for the safety population for the following categories 0 - <80%; >= 80%.

The study drug administration and compliance data will be listed for each patient.

## 5.3 Efficacy Endpoints and Analyses

Given the primary objective of the study being long term safety, efficacy analyses will be using the safety population (SP). The efficacy data will be summarized by previous treatment group in parent study as well as an overall group.

For each efficacy parameter, descriptive summary statistics at each visit will be provided for the observed value, change from baseline, and percent change from baseline in both conventional and International System of Units (SI). Two sets of summaries will be provided using the baseline from the parent study and from the OLE study. The visits to be included in the overtime summary are baseline of parent study (1002-040), baseline of OLE study, week 12, week 52, week 78, and Week 82. There will be no imputation for missing data, all summaries will use the observed data. Ninety-five percent (95%) CI will be provided for the estimates at post-baseline visits.

In addition, efficacy parameters will also be summarized using the Completer Analysis Set (CAS).

For LDL-C, the same descriptive summary statistics at each scheduled visit will be provided within each subgroup for the observed value, change from baseline, and percent change from baseline.

Efficacy data (observed value, change from baseline, and percent change from baseline) from all visits will be summarized using descriptive statistics in both conventional and standard units.

Figures (mean  $\pm$  standard deviation or median/interquartile range) supporting the summary tables will be provided for each efficacy parameter.

Efficacy data from all visits will be provided in listings as well.

By-visit summary for efficacy endpoints (LDL-C, non-HDL-C, TC, HDL-C, TG, ApoB, and hs-CRP,) using the CAS will be provided in conventional and standard units.

# 5.4 Safety Data Endpoints and Analyses

The safety and tolerability of ETC-1002 will be assessed by examination of TEAEs, PEs, vital signs, clinical laboratory values (serum chemistry, hematology, coagulation, and urinalysis), and weight. SP will be used for all safety analyses.

Unless otherwise stated, descriptive summaries will be performed by previous treatment group actually received in parent study and overall group.

#### 5.4.1 Adverse Events (AEs)

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 or later and will be categorized by system organ class (SOC) and preferred


term (PT). Summary tables will focus on TEAEs; however, listings will include all AEs (with non-TEAEs flagged). An additional AE listing will be provided for AEs occurred during rollover period.

In summary tables, TEAEs will be counted as "Not Related" if relationship to study drug was recorded as 'Not Related' or "Unlikely". Events will be counted as "Related" if relationship to study drug was recorded as 'Possible', 'Probable', 'Definite' or if relationship to study drug is missing.

The severity of the AE will be characterized as mild, moderate, or severe, to the following definitions:

- Mild: Events are usually transient and do not interfere with the patient's daily activities
- Moderate: Events introduce a low level of inconvenience or concern to the patient and may interfere with daily activities
- Severe: Events interrupt the patient's usual daily activity, are incapacitating with inability to do usual activities, or significantly affect clinical status and warrant intervention and/or close follow-up

Overviews of TEAEs will include total number of TEAEs, and patient incidence of TEAEs, TESAEs, treatment-related TEAEs, treatment-related TESAEs, IMP withdrawal due to TEAEs, TEAEs with fatal outcome. Individual TEAE summary will be presented by previous treatment group in parent study and overall containing the following counts and percentages for:

- patients with TEAEs by SOC and PT
- patients with TEAEs by PT
- patients with TEAEs by SOC, PT, and maximum severity
- patients with treatment-related TEAEs
- patients with treatment-related TEAEs by PT
- patients with treatment-related TEAEs by SOC and PT
- patients with treatment-emergent serious adverse events (TESAEs) by SOC and PT
- patients with TESAEs by PT
- patients with TESAEs by SOC, PT, and maximum severity
- patients with treatment-related TESAEs
- patients with treatment-related TESAEs by SOC and PT
- TEAEs leading to withdrawal of IMP by SOC and PT
- fatal TEAEs by SOC and PT

Preferred terms for TEAEs that occurred in more than 1% of subjects overall will be plotted using the overall group. This plot will be repeated for TESAEs in the overall group.


In addition, summary tables will be provided, by prior treatment group and overall, for the number and percent of patients experiencing:

- adjudicated major adverse cardiovascular events and mortality (MACE) by event type
- non-CV deaths (non-MACE),
- nonfatal myocardial infarction [MI] (MACE),
- nonfatal stroke (MACE),
- hospitalization for unstable angina (MACE),
- coronary revascularization (MACE),
- noncoronary arterial revascularization (non-MACE),
- hospitalization for heart failure (non-MACE) using standardized definitions.

The TEAE, treatment-related TEAE, TESAE, and AESI summaries by SOC, PT and maximum severity will be provided for relevant subgroups described in 5.2.5 with the exception of baseline LDL category.

The AE overview summaries will count a patient at most once in each AE category (at the "highest/most extreme" designation of each category regardless of preferred term) and percentages will be based on the total number of patients in the safety population.

In addition to a comprehensive listing of all AEs (with non-TEAEs flagged), separate listings will be generated for serious adverse events, TEAEs resulting in withdrawal of study drug, and TEAEs with a fatal outcome, investigator reported major adverse cardiovascular events and mortality, and adjudicated major adverse cardiovascular events and mortality.

## 5.4.2 Adverse Events of Special Interest

Adverse events of special interest (AESI) will be identified based on a pre-defined list of preferred terms provided by the sponsor (Appendix 2).

AESI will be presented in a listing and summarized by SOC, PT, and previous treatment group in parent study and overall in OLE study. A separate table for treatment-emergent AESI resulting in the discontinuation of study drug will be summarized by SOC, PT, and previous treatment group in the parent study and overall in OLE study.

In addition to adverse events, AESI is also being evaluated based on safety lab parameters. The details are provided in 5.4.5.

#### **5.4.2.1** Neurocognitive Events

Neurocognitive events will be identified and evaluated by routine safety monitoring of PE findings and AEs. Summarization of neurocognitive events will occur using pre-specified MedDRA terms and will be performed by SOC, severity, and relationship to study drug by previous treatment group in parent study and overall in OLE study.


## 5.4.3 Clinical Cardiovascular Endpoints

Clinical cardiovascular endpoints will be monitored and adjudicated by an independent blinded expert CEC for this study and other ongoing studies the ETC-1002 program. Adjudicated clinical endpoints that are treatment-emergent will be summarized by event type and previous treatment group in parent study and overall in OLE study. All events will be provided in a listing. Additional details regarding clinical endpoints and clinical endpoint definitions will be included in CEC charter.

## 5.4.4 Laboratory Evaluations

Continuous laboratory parameters (serum chemistry, hematology, coagulation (only for those patients receiving anti-coagulation), urinalysis, urinalysis [microscopic]) listed in Table 4 will be summarized in conventional unit and SI unit using descriptive statistics at each scheduled visit starting from the baseline of the parent study. The similar completer analysis set approach for efficacy analysis described in section 5.3 will be used for selected parameters. Missing values for any of the laboratory evaluations will not be imputed; that is, only observed case data will be used.

Fasting serum glucose and HbA1c will be summarized using descriptive statistics for the observed value, change from baseline, and percent change from baseline at each scheduled visit by history of diabetics.

Categorical urinalysis data will be listed, but will not be summarized.

As part of the AESI evaluation, below safety lab abnormality will be summarized by treatment group. All post-baseline lab values during the on-treatment period are being considered. Further details are provided in Section 5.4.6.1 through 5.4.6.4.

- ALT or AST ( $> 3 \times \text{Upper limit of normal (ULN)}$  and  $> 5 \times \text{ULN}$ )
- Total bilirubin (TB) ( $> 2 \times ULN$ )
- Potential Hy's Law case: (ALT and/or AST  $> 3 \times ULN$  with concurrent TB  $> 2 \times ULN$ )
- CK ( $> 5 \times ULN$ ) and ( $> 10 \times ULN$ )
- Fasting Serum Glucose (mg/dL) ( $\leq$  50, and  $\geq$  126) by history of diabetics
- HbA1<sub>C</sub> ( $\geq$  6.5%) by history of diabetics
- Creatinine (change from baseline for >1 mg/dL)
- eGFR (< 15 mL/min/1.73m<sup>2</sup>, 15 –29 mL/min/1.73m<sup>2</sup>)
- Hgb (g/dL) (decrease from baseline for  $\geq 2$  g/dL)
- Hgb (< 8 g/dL)

The number and percentage of patients with the following laboratory abnormalities will be summarized by the parent study baseline statin intensity, previous treatment group in the parent study, and overall in the OLE study:


- ALT or AST ( $> 3 \times ULN$  and  $> 5 \times ULN$ )
- TB (>  $2 \times ULN$ )
- Potential Hy's Law case: (ALT and/or AST  $> 3 \times$  ULN with concurrent TB  $> 2 \times$  ULN)
- CK (>  $5 \times ULN$ ) and (> $10 \times ULN$ )
- Creatinine (change from baseline for > 1 mg/dL)
- eGFR (< 15 mL/min/1.73m<sup>2</sup>, 15 –29 mL/min/1.73m<sup>2</sup>)
- Hgb (g/dL) (decrease from baseline for  $\geq 2$  g/dL)
- Hgb (< 8 g/dL)

For labs of interest (such as uric acid, hemoglobin, creatinine, BUN, and Fasting glucose by diabetes history), a line plot will be generated to visualize the mean values over time.

A matrix display of liver dysfunction shift from baseline to maximum value will be used to visualize the abnormal values of labs including AST, ALK-P ALT, and TB.


**Table 2:** Clinical Laboratory Parameters (Safety)

| Clinical Laboratory Test | Clinical Laboratory Test |
|---|---|
| Hematology | Blood Chemistry (serum, fasting) |
| Hematocrit (Hct) | Albumin (Alb) |
| Hemoglobin (Hgb) | Alkaline phosphatase (ALK-P) |
| Mean corpuscular hemoglobin (MCH) | Alanine aminotransferase (ALT; SGPT) |
| Mean corpuscular hemoglobin | <ul> <li>Aspartate aminotransferase (AST;</li> </ul> |
| concentration (MCHC) | SGOT) |
| Mean corpuscular volume (MCV) | Blood urea nitrogen (BUN) |
| Platelet count | Calcium (Ca) |
| Red blood (RBC) cell count | Carbon dioxide (CO2) |
| White blood (WBC) cell count with | Chloride (Cl) |
| differential (absolute and %) | Creatinine |
| <u>Urinalysis (Dipstick)</u> | • Creatine kinase (CK) |
| • Clarity | Glucose |
| Bilirubin | Lactate dehydrogenase (LDH) |
| • Color | <ul> <li>Phosphorus</li> </ul> |
| • Glucose | • Potassium (K) |
| • Ketones | Sodium (Na) |
| Leukocyte esterase | <ul> <li>Total and direct bilirubin (TB)a</li> </ul> |
| Nitrate | Total protein |
| Occult blood | Uric acid |
| • pH | Coagulation—only in patients receiving |
| • Protein | anticoagulant therapy that in the investigator's |
| Specific gravity | judgment require monitoring at Month 0 and |
| <ul> <li>Urobilinogen</li> </ul> | 3 to 5 days post-Month 0 |
| | Prothrombin time |
| | International normalized ration (INR) |
| <u>Urinalysis (Microscopic)-only if urine dipstick</u> | Other Labs: |
| abnormal | Urine pregnancy test |
| Bacteria | Hemoglobin A <sub>1C</sub> (HbA <sub>1C</sub> ) |
| • Casts | |
| • Crystals | |
| Epithelial cells | |
| • RBC | |
| • WBC | |

 $<sup>^{\</sup>rm a}$  If TB  ${\ge}1.2\times$  ULN, a reflex indirect (unconjugated) bilirubin will be obtained.


The number and percentage of patients with laboratory abnormalities (i.e., laboratory values outside the stated laboratory normal range) will be summarized at each time point (i.e., including baseline and post-baseline time points) for each laboratory parameter. The determination of laboratory abnormalities will take into account any unscheduled laboratory assessments. Additional lab-related summaries will be provided as follows for hepatic safety, musculoskeletal safety, diabetes and glycemia, and renal safety.

## **5.4.4.1 Hepatic Safety**

For liver-associated enzymes and total bilirubin (TB), the number and percent of patients with abnormal values for ALT ( $>3 \times ULN$ ,  $>5 \times ULN$ ), AST ( $>3 \times ULN$ ,  $>5 \times ULN$ ), and TB ( $>2 \times ULN$ ) will be summarized by overall, normal baseline ALT/AST/TB and abnormal baseline ALT/AST/TB.

Hy's law criteria (>  $3 \times \text{upper limit}$  of normal [ULN] for either ALT or AST, with accompanying TB >  $2 \times \text{ULN}$ ) will also be applied to the data; any potential Hy's law cases will be listed separately. In the case of patients with Gilbert's disease, TB will be fractionated and the determination of  $2 \times \text{ULN}$  will be based upon direct (conjugated) bilirubin.

The number and percentage of patients experiencing a single incident or confirmed and repeated incidence of abnormal liver function test values for ALT (>3 × ULN, >5 × ULN), AST (>3 × ULN, >5 x ULN), CK (>5 × ULN, >10 × ULN) and either ALT and/or AST (>3 × ULN, >5 × ULN) will be summarized by the previous treatment group in the parent study and overall in the OLE study. A single incident is defined as the patient experiencing only one abnormal incident of the liver function test value. Repeated and confirmed incidence is defined as the patient experiencing at least one of the following: the last onstudy liver function test value is abnormal, the last on-treatment liver function test value is abnormal liver function test value for the same test.

A separate listing for direct bilirubin will be provided for those who have Gilbert's syndrome.

#### **5.4.4.2 Musculoskeletal Safety**

CK levels will be summarized by the value and change from baseline in the value, by treatment group and visit as well as baseline eGFR category. In addition, the number and percent of patients with abnormal CK values (>5 X ULN, >10 × ULN) will be summarized. These summaries of patients with abnormal CK will be performed overall, normal baseline CK, and abnormal baseline CK.

#### 5.4.4.3 Diabetes and Glycemia

For fasting glucose and HbA1<sub>C</sub> (%), a shift table from baseline with the number and percent of patients will be categorized as below:

Fasting glucose: >= 126 mg/dL; 100-125 mg/dL, and < 100 mg/dL; Confidential


 $HbA1_C$  (%): >=6.5%; >5.5 to <=6.4% and <=5.5%.

These tables will be summarized by history of Diabetes.

Descriptive summary for fasting serum glucose and HbA1<sub>C</sub> will be provided by history of diabetics, previous treatment group in parent study and overall at each scheduled visit.

### 5.4.4.4 Renal Safety

Shift tables of eGFR category from baseline over the study, will be provided by previous treatment group in parent study and overall.

In addition, renal function abnormality will be identified as: (1) A creatinine change from baseline of > 1 mg/dL (2) eGFR value <30 mL/min/1.73m<sup>2</sup>. A shift table from baseline with the number and percent of patients using the two categories will be presented.

## 5.4.5 Physical Examination (PE)

Listings of PE data will include only those records where the body system at the baseline PE was normal, but the body system at a post-baseline PE was marked as 'Change from previous exam, clinically significant'. Baseline is defined as the last value prior to the first dose of study medication in OLE study. Only changes from baseline PE findings that meet the definition of an AE will be recorded on the AE page of the eCRF and will be summarized with other AE outcomes.

#### 5.4.6 Vital Signs and Weight

The observed values and changes from baseline of both parent study and OLE study in vital signs (heart rate, systolic blood pressure, diastolic blood pressure) and weight will be summarized using descriptive statistics by previous treatment group in parent study, overall and post-baseline time point.

Vital sign data will be listed for each patient, with increases from baseline of > 15 mmHg in systolic or diastolic blood pressure flagged.

# 6 DMC Analyses

Refer to DMC charter.

## 7 Reference

- 1. Sharrett AR, Ballantyne CM, Coady SA, Heiss G, Sorlie PD, Catellier D, et al. Atherosclerosis Risk in Communities Study Group. Coronary Heart Disease Prediction from Lipoprotein Cholesterol Levels, Triglycerides, Lipoprotein(A), Apolipoproteins A-I and B, and HDL Density Subfractions. The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2001;104:1108-13.
- 2. World Health Organization (WHO) Fact Sheet No 317 Updated January 2015.
- 3. Robinson JG. Management of Familial Hypercholesterolemia: A Review of the recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Managed Care Pharm. 2013;19(2):139-49.
- 4. Pharmacokinetics in Patients with Impaired Renal Function Study Design, Data Analysis, and Impact on Dosing and Labeling. FDA Draft Guidance. March 2010
- 5. Haase A, Goldberg AC. Identification of people with heterozygous familial hypercholesterolemia. Curr Opin Lipidol. 2012;23:282-9.
- 6. Glynn RJ, Laird NM, and Rubin DB. (1986). Selection modelling versus mixture modelling with nonignorable nonresponse. In H. Wainer (ed.), Drawing Inferences from Self-Selected Samples, pp. 115–142. New York: Springer.


# 8 Appendices

# 8.1 Appendix 1: Schedule of Events (Subject Visit Schedule)

| Month | 0 | 3 | 6 | 9 | 12 | 15 | 18/EOT <sup>1</sup> | 19/EOS <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|
| Week | EOS | Wk 12 | Wk 24 | Wk 36 | Wk 52 | Wk 64 | Wk 78 | Wk 82 |
| | Parent | | | | | | | |
| Visit Window | 30 Days | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days | ±7 days | +14 days |
| | pre-M0 | | | | | | | |
| In-clinic Visit | X | X | | | X | | X | X |
| Phone Visit | | | X | X | | X | | |
| Procedure | | | | | | | | |
| Informed Consent | X | | | | | | | |
| Enrollment Criteria | X | | | | | | | |
| Medical History | X | | | | | | | |
| Concomitant | X | X | X | X | X | X | X | X |
| Medications | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X |
| Recording | | | | | | | | |
| Physical Exam | X | | | | X | | X | |
| Weight <sup>3</sup> | X | X | | | X | | X | X |
| Vital Signs <sup>4</sup> | X | X | | | X | | X | X |
| Urine Pregnancy Test <sup>5</sup> | X | | | | | | | |
| Clinical Safety Labs <sup>6</sup> | X | X | | | X | | X | X |
| Basic Fasting Lipids <sup>7</sup> | X | X | | | X | | X | X |
| Coagulation <sup>8</sup> | X | | | | | | | |
| ApoB and hsCRP | X | X | | | X | | X | X |
| HbA <sub>1C</sub> | X | | | | X | | X | X |
| IWRS Contact <sup>9</sup> | X | X | | | X | | X | |
| Drug Dispensing | X | X | | | X | | | |
| Drug Return/ | | X | | | X | | X | |
| Compliance | | | | | | | | |

NOTE: For patients who withdraw from study drug treatment, but consent to be followed for safety assessments and return to clinic for these visit, the visits will occur according to the protocol schedule. Safety assessments should include clinical safety and basic lipid laboratories, adverse events (AEs), physical examination (PE), and vital signs. For patients who withdraw from study drug treatment, but consent to be followed for safety assessments by phone, the telephone contacts will occur according the protocol schedule with information regarding current health status and to collect information on AEs (eg, recent procedures, hospitalizations, and if the patient has died, the cause of death). If a patient does not provide consent to be followed for safety assessments per the protocol (either by returning to clinic or by phone), Visit Week 78/End of Treatment (EOT) will be scheduled as soon as possible and the patient will be asked to come back 4 weeks after last investigational medicinal product (IMP) dose for Visit Week 82/End of Study (EOS). No further visits will be scheduled.


<sup>&</sup>lt;sup>1</sup> All procedures will be completed for all patients at either EOT or early withdrawal.

<sup>&</sup>lt;sup>2</sup> All procedures will be completed for all patients 4 weeks after last IMP dose if completing the study or early withdrawal.

<sup>&</sup>lt;sup>3</sup> Body weight will be measured in the morning while fasting, using consistent scales, after voiding, and without shoes and outerwear (eg, coats).

<sup>&</sup>lt;sup>4</sup> Vital signs will include diastolic blood pressure (DBP), systolic blood pressure (SBP), heart rate (HR) and will be collected prior to any blood sample collection. Patient will rest for 5 minutes prior to assessments

- <sup>6</sup> Clinical safety labs include hematology, blood chemistry, and urinalysis at all visits. Please refer to laboratory manual for detailed schedule of tests.
- <sup>7</sup> Basic fasting lipids include total cholesterol (TC), calculated low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-HDL-C,), and triglycerides (TG).
- <sup>8</sup> Only in patients receiving anticoagulant therapy that in the investigator's judgment require monitoring at Month 0 and 3 to 5 days post-Month 0
- <sup>9</sup> Interactive web response system (IWRS) contact at either an early withdrawal or an EOS visit to register study discontinuation visit date

<sup>&</sup>lt;sup>5</sup> Urine pregnancy test in women of childbearing potential only

# 8.2 Appendix 2: Adverse Event of Special Interest (AESI)

| Adverse Event Terms per Protocol | Associated MedDRA Preferred Terms |
|---|---|
| Creatine kinase elevations | Blood creatine phosphokinase abnormal |
| Creatine kinase elevations Creatine kinase elevations | Blood creatine phosphokinase achierman |
| Creatine kinase elevations Creatine kinase elevations | Blood creatine phosphokinase MM abnormal |
| Creatine kinase elevations Creatine kinase elevations | Blood creatine phosphokinase MM increased |
| | Blood glucose abnormal |
| New onset or worsening diabetes mellitus | C |
| New onset or worsening diabetes mellitus | Blood glucose increased |
| New onset or worsening diabetes mellitus | Diabetes mellitus |
| New onset or worsening diabetes mellitus | Diabetes mellitus inadequate control |
| New onset or worsening diabetes mellitus | Diabetic ketoacidosis |
| New onset or worsening diabetes mellitus | Glucose tolerance impaired |
| New onset or worsening diabetes mellitus | Glucose urine present |
| New onset or worsening diabetes mellitus | Glycosuria |
| New onset or worsening diabetes mellitus | Glycosylated haemoglobin increased |
| New onset or worsening diabetes mellitus | Hyperglycaemia |
| New onset or worsening diabetes mellitus | Impaired fasting glucose |
| New onset or worsening diabetes mellitus | Ketoacidosis |
| New onset or worsening diabetes mellitus | Ketosuria |
| New onset or worsening diabetes mellitus | Ketosis |
| New onset or worsening diabetes mellitus | Type 2 diabetes mellitus |
| New onset or worsening diabetes mellitus | Urine ketone body present |
| Hepatic disorders | Alanine aminotransferase abnormal |
| Hepatic disorders | Alanine aminotransferase increased |
| Hepatic disorders | Aspartate aminotransferase abnormal |
| Hepatic disorders | Aspartate aminotransferase increased |
| Hepatic disorders | Blood bilirubin abnormal |
| Hepatic disorders | Blood bilirubin increased |
| Hepatic disorders | Hepatic enzyme abnormal |
| Hepatic disorders | Hepatic enzyme increased |
| Hepatic disorders | Hypertransaminaseaemia |
| Hepatic disorders | Liver function test abnormal |
| Hepatic disorders | Liver function test increased |
| Hepatic disorders | Transaminases abnormal |
| Hepatic disorders | Transaminases increased |
| Hypoglycemia | Blood glucose abnormal |
| Hypoglycemia | Blood glucose decreased |
| Hypoglycemia | Hypoglycaemia |
| Hypoglycemia Hypoglycemia | Hypoglycaemic coma |
| Hypoglycemia Hypoglycemia | Hypoglycaemic encephalopathy |
| Hypoglycemia | Hypoglycaemic seizure |
| Hypoglycemia Hypoglycemia | Shock hypoglycaemic |
| Metabolic acidosis | Metabolic acidosis |
| Muscular disorders | Muscular weakness |
| Muscular disorders Muscular disorders | Muscle necrosis |
| Muscular disorders | iviuscie necrosis |


| Muscular disorders | Muscle spasms |
|---|---|
| Muscular disorders | Myalgia |
| Muscular disorders | Myoglobin blood increased |
| Muscular disorders | Myoglobin blood present |
| Muscular disorders | Myoglobin urine present |
| Muscular disorders | Myoglobinaemia |
| Muscular disorders | Myoglininuria |
| Muscular disorders | Myopathy |
| Muscular disorders | Myopathy toxic |
| Muscular disorders | Necrotizing myositis |
| Muscular disorders | Pain in extremity |
| Muscular disorders | Rhabdomyolysis |
| Neurocognitive/Neurologic disorders | Amnesia |
| Neurocognitive/Neurologic disorders | Cognitive disorder |
| Neurocognitive/Neurologic disorders | Confusional state |
| Neurocognitive/Neurologic disorders | Disorientation |
| Neurocognitive/Neurologic disorders | Memory impairment |
| Neurocognitive/Neurologic disorders | Mental status changes |
| Renal disorders | Acute kidney injury |
| Renal disorders | Acute prerenal failure |
| Renal disorders | Blood creatinine abnormal |
| Renal disorders | Blood creatinine increased |
| Renal disorders | Blood urea abnormal |
| Renal disorders | Blood urea increased |
| Renal disorders | Blood urea nitrogen/Creatinine ratio increased |
| Renal disorders | Creatinine renal clearance abnormal |
| Renal disorders | Creatinine renal clearance decreased |
| Renal disorders | Glomerular filtration rate abnormal |
| Renal disorders | Glomerular filtration rate decreased |
| Renal disorders | Gout |
| Renal disorders | Oliguria |
| Renal disorders | Prerenal failure |
| Renal disorders | Renal failure |
| Renal disorders | Renal function test abnormal |
| Renal disorders | Renal impairment |